CLINICAL TRIAL: NCT03192176
Title: A Randomized, Placebo-Controlled, Double-Blind, Dose-Ranging, Phase 2b Study to Investigate the Efficacy of ESN364 in Postmenopausal Women Suffering From Vasomotor Symptoms (Hot Flashes)
Brief Title: A Dose-ranging Study of the Efficacy of ESN364 in Postmenopausal Women Suffering Vasomotor Symptoms (Hot Flashes)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESN364_HF_205
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Results first posted 2021-09-29 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Menopause; Hot Flashes
Keywords: Vasomotor symptoms; Menopause; Hot flashes; Perimenopause
MeSH Terms: conditions — Hot Flashes | interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Placebo (Placebo Comparator): Participants received fezolinetant matching placebo capsules orally, BID for a period of 12 weeks.
  Interventions: Drug: Fezolinetant
- Fezolinetant 15 mg (Experimental): Participants received fezolinetant 15 mg capsules orally, BID for a period of 12 weeks.
  Interventions: Drug: Placebo
- Fezolinetant 30 mg (Experimental): Participants received fezolinetant 30 mg capsules orally, BID for a period of 12 weeks.
  Interventions: Drug: Fezolinetant
- Fezolinetant 60 mg (Experimental): Participants received fezolinetant 60 mg capsules orally, BID for a period of 12 weeks.
  Interventions: Drug: Fezolinetant
- Fezolinetant 90 mg (Experimental): Participants received fezolinetant 90 mg capsules orally, BID for a period of 12 weeks.
  Interventions: Drug: Fezolinetant
- Fezolinetant 30 mg + Placebo (Experimental): Participants received fezolinetant 30 mg capsules orally, QD and matching placebo QD for a period of 12 weeks.
  Interventions: Drug: Fezolinetant
- Fezolinetant 60 mg + Placebo (Experimental): Participants received fezolinetant 60 mg capsules orally, QD and matching placebo QD for a period of 12 weeks.
  Interventions: Drug: Fezolinetant
- Fezolinetant 120 mg + Placebo (Experimental): Participants received fezolinetant 120 mg capsules orally, QD and matching placebo QD for a period of 12 weeks.
  Interventions: Drug: Fezolinetant

INTERVENTIONS:
Drug: Fezolinetant — Oral Capsule
  Other Names: ESN364
  Arms: Fezolinetant 120 mg + Placebo; Fezolinetant 30 mg; Fezolinetant 30 mg + Placebo; Fezolinetant 60 mg; Fezolinetant 60 mg + Placebo; Fezolinetant 90 mg; Placebo
Drug: Placebo — Oral Capsule
  Arms: Fezolinetant 15 mg

SUMMARY:
This study determined the effects of different doses and dosing regimens of ESN364 on the frequency and severity of hot flashes. The treatment was administered for 12 weeks to postmenopausal women, aged 40 to 65, suffering at least 50 moderate to severe hot flashes per week.

DETAILED DESCRIPTION:
This was a 12-week randomized, double-blind, placebo-controlled, dose-ranging, parallel-group, multi-center study to assess the efficacy of ESN364 in postmenopausal women suffering from vasomotor symptoms (hot flashes).

This study consisted of a screening period (Days -35 to -1, including the screening visit [Visit 1] and a minimum 7-day collection of baseline vasomotor symptom frequency and severity assessments), a 12 week treatment period (Day 1 [Visit 2] to Week 12 [Visit 5]), and a follow up visit (Week 15 [Visit 6]) 3 weeks after the last dose of study drug.

The study was performed on an ambulatory basis. The screening visit (Visit 1) occurred up to 35 days prior to randomization. Eligibility was assessed via physical examination, clinical laboratory testing, vital signs, ECG, Pap smear, mammography, and endometrial biopsy. Subjects received an electronic diary to record daily vasomotor symptoms during the duration of the screening period. Subjects who had ≥7 consecutive days of vasomotor symptom recordings participated in the study. Subjects are encouraged to continue recording for the duration of the whole screening period. The electronic diary was reviewed by study site staff on Day 1 (Visit 2) to confirm study eligibility. Subjects were rescreened 1 time upon approval of the medical monitor.

During the treatment period, subjects returned to the study site every 4 weeks for assessments.

The follow-up visit occurred approximately 3 weeks following the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Women >40 years and ≤65 years of age at the screening visit;
* A body mass index between 18 kg/sqm to 38 kg/sqm (extremes included);
* Spontaneous amenorrhea for ≥12 consecutive months; or spontaneous amenorrhea for ≥6 months with biochemical criteria of menopause (follicle-stimulating hormone [FSH] >40 IU/L); or having had bilateral oophorectomy ≥6 weeks prior to the screening visit (with or without hysterectomy);
* At least 50 moderate to severe vasomotor symptoms per week (ie, 7 consecutive days), as recorded in the daily diary during the screening period;
* In good general health as determined on the basis of medical history and general physical examination, including a bimanual clinical pelvic examination and clinical breast examination devoid of relevant clinical findings, performed at the screening visit; hematology and biochemistry parameters, pulse rate and/or blood pressure, and ECG within the reference range for the population studied, or showing no clinically relevant deviations, as judged by the Investigator;
* Women >40 years of age who have documentation of a normal/negative or no clinically significant findings mammogram (obtained at Screening or within the prior 9 months of trial enrollment.) Appropriate documentation includes a written report or an electronic report indicating normal/negative or no clinically significant mammographic findings;
* Willing to undergo a transvaginal ultrasound to assess endometrial thickness at Screening and at Week 12 (end-of-treatment, - and subjects) who are withdrawn from the study prior to completion, at the Early Termination (ET) Visit. This is not required for subjects who have had a partial (supracervical) or full hysterectomy;
* Willing to undergo an endometrial biopsy at Screening (in the event that the subject's transvaginal ultrasound shows endometrial thickness ≥4 mm) and at Week 12 (end--of--treatment) - all subjects), for subjects with uterine bleeding, and for subjects who are withdrawn from the study prior to completion, at the ET Visit if study drug exposure is ≥10 weeks. This is not required for subjects who have had a partial (supracervical) or full hysterectomy;
* Negative alcohol breath test and negative urine test for selected drugs of abuse (amphetamines, tricyclic antidepressants, cocaine, or opiates) at the screening visit;
* Negative urine pregnancy test;
* Negative serology panel (including hepatitis B surface antigen, hepatitis C virus antibody, and human immunodeficiency virus antibody screens);
* Informed Consent Form signed voluntarily before any study-related procedure is performed, indicating that the subject understands the purpose of and procedures required for the study and is willing to participate in the study; and
* Documentation of a normal Pap smear (or equivalent cervical cytology) or of no clinical significance in the opinion of the Investigator within the previous 9 months or at Screening.

Exclusion Criteria:

* Use of a prohibited therapy (hormone therapy, hormonal contraceptive, or vasomotor symptom medication [prescription, over the counter, or herbal]) or not willing to wash out drugs
* History (in the past year) or presence of drug or alcohol abuse;
* Previous or current history of a malignant tumor, except for basal cell carcinoma;
* Uncontrolled hypertension and a systolic blood pressure ≥140 mmHg and/or a diastolic blood pressure ≥90 mmHg;
* Judged by the Investigator to be unsuited to participate in the study based on findings observed during physical examination, vital sign assessment, or 12-lead electrocardiogram (ECG);
* History of severe allergy, hypersensitivity, or intolerance to drugs in general, including the study drug and any of its excipients;
* Exclusion criterion 7 has been removed in Amendment 1;
* An unacceptable result from endometrial biopsy (performed when endometrial thickness is ≥ 4mm measured by transvaginal ultrasound) of endometrial hyperplasia, endometrial cancer, or inadequate specimen at Screening (1 repeat biopsy permitted if technically possible);
* History of endometrial hyperplasia or uterine/endometrial cancer;
* History of unexplained uterine bleeding;
* History of seizures or other convulsive disorders;
* Medical condition or chronic disease (including history of neurological [including cognitive], hepatic, renal, cardiovascular, gastrointestinal, pulmonary [eg, moderate asthma], endocrine, or gynecological disease) or malignancy that could confound interpretation of the study outcome;
* Presence or sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion (ADME) mechanisms of drugs as judged by the Investigator;
* Active liver disease or jaundice, or values of alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >1.5 x the upper limit of normal (ULN); or total bilirubin >1.5 x ULN; or creatinine >1.5 x ULN; or estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease formula ≤59 mL/min/1.73 sqm at the screening visit;
* Concurrent participation in another interventional study (or participation within 3 months prior to screening in this study);
* Suicide attempt in the past 3 years;
* Unable or unwilling to complete the study procedures; or
* Subject is the Investigator or any sub-Investigator, research assistant, pharmacist, study coordinator, or other staff or relative thereof, who is directly involved in the conduct of the study.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (50):
- United States (50):
  - Research Site, Anniston, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Oceanside, California
  - Research Site, Panorama City, California
  - Research Site 052, Sacramento, California
  - Research Site 058, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Thousand Oaks, California
  - Research Site, Valley Village, California
  - Research Site, Denver, Colorado
  - Research Site, Milford, Connecticut
  - Research Site, Crystal River, Florida
  - Research Site, DeLand, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Miami, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Port Saint Lucie, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Norcross, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Champaign, Illinois
  - Research Site, Marrero, Louisiana
  - Research Site, Elkridge, Maryland
  - Research Site, Watertown, Massachusetts
  - Research Site, Lincoln, Nebraska
  - Research Site, Norfolk, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, New York, New York
  - Research Site, Williamsville, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Clarksville, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Hurst, Texas
  - Research Site, Lampasas, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Riverton, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Vienna, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Fraser GL, Lederman S, Waldbaum A, Kroll R, Santoro N, Lee M, Skillern L, Ramael S. A phase 2b, randomized, placebo-controlled, double-blind, dose-ranging study of the neurokinin 3 receptor antagonist fezolinetant for vasomotor symptoms associated with menopause. Menopause. 2020 Apr;27(4):382-392. doi: 10.1097/GME.0000000000001510. PMID 32102086
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — http://www.trialsummaries.com/Study/StudyDetails?id=14565&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women participants 40 to 65 years of age who had at least 50 moderate to severe vasomotor symptoms (VMS) per week and who met the inclusion criteria and none of the exclusion criteria were enrolled in this study.
Pre-assignment Details: Prior to randomization, participants had a screening period during which a minimum 7-day collection of baseline VMS frequency and severity assessments were performed.
Groups:
- Placebo BID: Participants received fezolinetant matching placebo capsules orally, twice daily (BID) for a period of 12 weeks.
- Fezolinetant 15 mg BID: Participants received fezolinetant 15 mg capsules orally, BID for a period of 12 weeks.
- Fezolinetant 30 mg BID: Participants received fezolinetant 30 mg capsules orally, BID for a period of 12 weeks.
- Fezolinetant 60 mg BID: Participants received fezolinetant 60 mg capsules orally, BID for a period of 12 weeks.
- Fezolinetant 90 mg BID: Participants received fezolinetant 90 mg capsules orally, BID for a period of 12 weeks.
- Fezolinetant 30 mg QD: Participants received fezolinetant 30 mg capsules orally, once daily (QD) and matching placebo QD for a period of 12 weeks.
- Fezolinetant 60 mg QD: Participants received fezolinetant 60 mg capsules orally, QD and matching placebo QD for a period of 12 weeks.
- Fezolinetant 120 mg QD: Participants received fezolinetant 120 mg capsules orally, QD and matching placebo QD for a period of 12 weeks.
Period: Overall Study
Arm/Group | Placebo BID | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Started | 44 | 45 | 44 | 45 | 44 | 45 | 45 | 44
Treated | 43 | 45 | 43 | 45 | 44 | 43 | 45 | 44
Completed | 37 | 40 | 38 | 33 | 32 | 34 | 36 | 37
Not Completed | 7 | 5 | 6 | 12 | 12 | 11 | 9 | 7
Not completed — Adverse Event | 1 | 0 | 4 | 5 | 3 | 2 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 3 | 1 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Protocol Deviation | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 0 | 4 | 3 | 4 | 4 | 2
Not completed — Miscellaneous | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAF) consisted of all randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo BID: Participants received fezolinetant matching placebo capsules orally, BID for a period of 12 weeks.
- Fezolinetant 30 mg QD: Participants received fezolinetant 30 mg capsules orally, QD and matching placebo QD for a period of 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo BID | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD | Total
Number analyzed (Participants) | 43 | 45 | 43 | 45 | 44 | 43 | 45 | 44 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (5.5) | 53.7 (5.0) | 53.9 (3.8) | 54.6 (5.0) | 54.9 (4.0) | 52.7 (3.8) | 55.0 (4.9) | 56.8 (4.4) | 54.6 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 45 | 43 | 45 | 44 | 43 | 45 | 44 | 352
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 9 | 13 | 10 | 17 | 12 | 9 | 101
  Not Hispanic or Latino | 28 | 29 | 34 | 32 | 34 | 26 | 33 | 35 | 251
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Asian | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 8 | 12 | 15 | 8 | 11 | 10 | 13 | 87
  White | 30 | 37 | 31 | 28 | 36 | 31 | 34 | 30 | 257
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3
Frequency of Moderate and Severe Vasomotor Symptoms per 24h [Mean (Standard Deviation); unit: VMS per day] — The frequency of moderate to severe VMS was the number of moderate to severe VMS per 24 hours. Baseline was the average frequency of 24 h vasomotor symptom from 7 non-missing days prior to day 1. Population: The full analysis set (FAS) consisted of all randomized participants who received at least 1 dose of study drug and had baseline and at least one postbaseline efficacy evaluation.
  VMS per day
    number analyzed (Participants) | 43 | 45 | 43 | 45 | 42 | 43 | 44 | 44 | 349
    (all) | 9.71 (3.53) | 11.12 (7.13) | 9.85 (4.62) | 9.48 (3.97) | 9.32 (3.59) | 11.18 (6.44) | 9.42 (2.70) | 9.65 (3.73) | 9.97 (4.71)
Severity of Moderate and Severe Vasomotor Symptoms per 24h [Mean (Standard Deviation); unit: Score on a scale] — Severity of moderate to severe VMS per day was calculated as follows:
  [(number of moderate VMS × 2) + (number of severe VMS × 3)]/number of daily moderate/severe VMS. Higher score indicates greater severity. Baseline was the average severity of 24h vasomotor symptom from 7 non-missing days prior to Day 1. Population: FAS Population
  Score on a scale
    number analyzed (Participants) | 43 | 45 | 43 | 45 | 42 | 43 | 44 | 44 | 349
    (all) | 2.46 (0.31) | 2.45 (0.27) | 2.43 (0.31) | 2.45 (0.31) | 2.38 (0.30) | 2.43 (0.30) | 2.40 (0.26) | 2.49 (0.32) | 2.44 (0.30)
Frequency of Mild, Moderate, and Severe Vasomotor Symptoms per 24h [Mean (Standard Deviation); unit: VMS per day] — The frequency of mild, moderate and severe VMS was the number of mild, moderate and severe VMS per 24 hours. Baseline was the average frequency of 24 h vasomotor symptom from 7 non-missing days prior to day 1. Population: FAS Population
  VMS per day
    number analyzed (Participants) | 43 | 45 | 43 | 45 | 42 | 43 | 44 | 44 | 349
    (all) | 9.96 (3.49) | 11.63 (7.10) | 10.33 (4.88) | 10.14 (4.22) | 9.85 (4.31) | 11.72 (6.66) | 10.15 (2.86) | 10.15 (3.78) | 10.5 (4.88)
Severity of Mild, Moderate, and Severe Vasomotor Symptoms per 24h [Mean (Standard Deviation); unit: Score on a scale] — Severity of mild, moderate and severe VMS per day was calculated as follows:
  [(number of mild VMS × 1) + (number of moderate VMS × 2) + (number of severe VMS × 3)]/ number of daily mild/moderate/severe VMS. Higher score indicates greater severity. Baseline was the average severity of 24h vasomotor symptom from 7 non-missing days prior to Day 1. Population: FAS Population
  Score on a scale
    number analyzed (Participants) | 43 | 45 | 43 | 45 | 42 | 43 | 44 | 44 | 349
    (all) | 2.43 (0.32) | 2.38 (0.29) | 2.37 (0.33) | 2.38 (0.36) | 2.33 (0.33) | 2.38 (0.34) | 2.31 (0.31) | 2.43 (0.37) | 2.38 (0.33)

OUTCOME MEASURES:

1. Primary Outcome: Co-Primary Efficacy Endpoint: Change From Baseline (CFB) in The Mean Frequency of Moderate to Severe Vasomotor Symptoms (VMS) at Week 4
Description: The frequency of moderate to severe VMS was the number of moderate to severe VMS per 24 hours. A daily frequency and severity per week was derived by taking the mean of the data over 7 days. Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed).
Time Frame: Baseline and week 4
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: VMS per day
Arm/Group | Placebo BID | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
VMS per day | -4.2 (0.65) | -6.1 (0.65) | -7.2 (0.64) | -7.0 (0.62) | -7.7 (0.65) | -6.5 (0.65) | -7.2 (0.61) | -6.6 (0.63)
Statistical Analysis 1: Comparison: Placebo BID vs Fezolinetant 15 mg BID; Test type: Superiority; p = 0.0240, ANCOVA — LS Means(LSM), standard errors(SE), confidence intervals(CI), & p-values come from an ANCOVA model with CFB as the dependent variable & treatment group, pooled center, smoking status as factors & baseline measurement, baseline weight as covariates; LSMean difference = -1.9, 95% CI 2-sided [-3.56 to -0.25], Standard Error of Mean 0.84
Statistical Analysis 2: Comparison: Placebo BID vs Fezolinetant 30 mg BID; Test type: Superiority; p = 0.0004, ANCOVA — LS Means, SE, CI, and p-values come from an ANCOVA model with change from baseline as the dependent variable and treatment group, pooled center, smoking status as factors and baseline measurement, baseline weight as covariates; LSMean difference = -3.0, 95% CI 2-sided [-4.68 to -1.38], Standard Error of Mean 0.84
Statistical Analysis 3: Comparison: Placebo BID vs Fezolinetant 60 mg BID; Test type: Superiority; p = 0.0010, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -2.8, 95% CI 2-sided [-4.44 to -1.14], Standard Error of Mean 0.84
Statistical Analysis 4: Comparison: Placebo BID vs Fezolinetant 90 mg BID; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -3.5, 95% CI 2-sided [-5.20 to -1.89], Standard Error of Mean 0.84
Statistical Analysis 5: Comparison: Placebo BID vs Fezolinetant 30 mg QD; Test type: Superiority; p = 0.0058, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -2.3, 95% CI [-4.00 to -0.68], Standard Error of Mean 0.84
Statistical Analysis 6: Comparison: Placebo BID vs Fezolinetant 60 mg QD; Test type: Superiority; p = 0.0003, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -3.0, 95% CI 2-sided [-4.65 to -1.41], Standard Error of Mean 0.82
Statistical Analysis 7: Comparison: Placebo BID vs Fezolinetant 120 mg QD; Test type: Superiority; p = 0.0042, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -2.4, 95% CI 2-sided [-4.06 to 0.76], Standard Error of Mean 0.84

2. Primary Outcome: Co-Primary Efficacy Endpoint: Change From Baseline in The Mean Frequency of Moderate to Severe VMS at Week 12
Description: as for outcome 1
Time Frame: Baseline and week 12
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: VMS per day
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
VMS per day | -5.3 (0.58) | -7.2 (0.54) | -7.5 (0.56) | -7.6 (0.55) | -8.0 (0.58) | -7.4 (0.58) | -7.9 (0.54) | -7.4 (0.57)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Test type: Superiority; p = 0.0154, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -1.8, 95% CI 2-sided [-3.30 to -0.35], Standard Error of Mean 0.75
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Test type: Superiority; p = 0.0043, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -2.1, 95% CI 2-sided [-3.60 to -0.67], Standard Error of Mean 0.74
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Test type: Superiority; p = 0.0023, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -2.3, 95% CI 2-sided [-3.76 to -0.83], Standard Error of Mean 0.75
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Test type: Superiority; p = 0.0005, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -2.6, 95% CI 2-sided [-4.09 to -1.16], Standard Error of Mean 0.75
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Test type: Superiority; p = 0.0064, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -2.1, 95% CI 2-sided [-3.52 to -0.58], Standard Error of Mean 0.75
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Test type: Superiority; p = 0.0005, ANCOVA — [p-value comment as in outcome 1, analysis 2]; -2.6 = -2.6, 95% CI 2-sided [-4.04 to -1.15], Standard Error of Mean 0.74
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Test type: Superiority; p = 0.0063, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -2.1, 95% CI 2-sided [-3.52 to -0.59], Standard Error of Mean 0.75

3. Primary Outcome: Co-Primary Efficacy Endpoint: Change From Baseline in The Mean Severity of Moderate to Severe VMS at Week 4
Description: Severity of moderate to severe VMS per day was calculated as follows:
  [(number of moderate VMS × 2) + (number of severe VMS × 3)]/number of daily moderate/severe VMS.
  Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed).
  Severity was zero for participants that had no moderate or severe VMS. Higher score indicates greater severity.
Time Frame: Baseline and week 4
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
Score on a scale | -0.3 (0.15) | -0.8 (0.14) | -0.9 (0.15) | -1.2 (0.14) | -1.3 (0.15) | -0.7 (0.15) | -0.9 (0.14) | -1.0 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Test type: Superiority; p = 0.0215, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -0.5, 95% CI 2-sided [-0.84 to -0.07], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Test type: Superiority; p = 0.0017, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -0.6, 95% CI 2-sided [-1.01 to -0.24], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -0.8, 95% CI 2-sided [-1.21 to -0.44], Standard Error of Mean 0.20
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -1.0, 95% CI 2-sided [-1.37 to -0.59], Standard Error of Mean 0.20
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Test type: Superiority; p = 0.0322, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -0.4, 95% CI 2-sided [-0.81 to -0.04], Standard Error of Mean 0.20
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Test type: Superiority; p = 0.0017, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -0.6, 95% CI 2-sided [-0.99 to -0.23], Standard Error of Mean 0.19
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Test type: Superiority; p = 0.0004, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean differencce = -0.7, 95% CI 2-sided [-1.08 to -0.31], Standard Error of Mean 0.20

4. Primary Outcome: Co-Primary Efficacy Endpoint: Change From Baseline in The Mean Severity of Moderate to Severe VMS at Week 12
Description: Severity of moderate to severe VMS per day was calculated as follows:
  [(number of moderate VMS × 2) + (number of severe VMS × 3)]/number of daily moderate/severe VMS.
  Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed).
  Severity was zero for participants that had no moderate or severe VMS. Higher scores indicates greater severity.
Time Frame: Baseline and week 12
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
Score on a scale | -0.8 (0.16) | -1.0 (0.15) | -1.1 (0.16) | -1.3 (0.16) | -1.4 (0.17) | -0.9 (0.16) | -1.3 (0.15) | -1.1 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Test type: Superiority; p = 0.2324, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -0.3, 95% CI 2-sided [-0.67 to -0.16], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Test type: Superiority; p = 0.0736, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -0.4, 95% CI 2-sided [-0.80 to 0.04], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Test type: Superiority; p = 0.0080, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -0.6, 95% CI 2-sided [-0.98 to -0.15], Standard Error of Mean 0.21
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Test type: Superiority; p = 0.0028, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -0.6, 95% CI 2-sided [-1.07 to -0.22], Standard Error of Mean 0.21
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Test type: Superiority; p = 0.4647, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean differnce = -0.2, 95% CI 2-sided [-0.58 to 0.26], Standard Error of Mean 0.21
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Test type: Superiority; p = 0.0160, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -0.5, 95% CI 2-sided [-0.92 to -0.10], Standard Error of Mean 0.21
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Test type: Superiority; p = 0.0901, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LSMean difference = -0.4, 95% CI 2-sided [-0.78 to 0.06], Standard Error of Mean 0.21

5. Secondary Outcome: Change From Baseline in The Mean Frequency of Mild, Moderate, and Severe VMS to Each Study Week
Description: The frequency of mild, moderate and severe VMS was the number of mild, moderate and severe VMS per 24 hours. A daily frequency and severity per week was derived by taking the mean of the data over 7 days. Mild VMS was defined as sensation of heat without sweating/dampness. If at night, subject does not wake up but later notices damp sheets or clothing. Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed).
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: VMS per day
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
VMS per day
  Week 1 | -2.0 (0.60) | -3.4 (0.56) | -4.7 (0.59) | -5.5 (0.58) | -6.1 (0.61) | -3.0 (0.61) | -4.4 (0.56) | -4.8 (0.59)
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | -3.6 (0.62) | -4.9 (0.58) | -6.3 (0.61) | -6.8 (0.60) | -7.3 (0.63) | -5.1 (0.63) | -5.4 (0.59) | -6.0 (0.61)
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | -3.8 (0.63) | -5.6 (0.60) | -6.8 (0.62) | -7.3 (0.61) | 7.7 (0.64) | -5.8 (0.64) | -6.1 (0.60) | -6.6 (0.62)
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | -4.0 (0.63) | -5.7 (0.60) | -7.0 (0.62) | -7.2 (0.61) | -8.1 (0.64) | -6.0 (0.64) | -6.8 (0.60) | -7.1 (0.62)
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | -4.6 (0.60) | -5.8 (0.57) | -7.2 (0.59) | -7.6 (0.58) | -8.5 (0.61) | -6.6 (0.61) | -6.8 (0.56) | -7.1 (0.59)
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | -4.9 (0.60) | -6.2 (0.57) | -7.2 (0.59) | -8.0 (0.58) | -8.6 (0.62) | -6.6 (0.61) | -7.1 (0.57) | -7.6 (0.59)
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | -4.9 (0.61) | -6.2 (0.58) | -7.4 (0.60) | -7.8 (0.59) | -8.7 (0.63) | -6.8 (0.62) | -7.2 (0.58) | -7.7 (0.60)
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | -5.5 (0.61) | -6.2 (0.58) | -7.5 (0.60) | -8.1 (0.60) | -8.5 (0.63) | -6.8 (0.63) | -7.4 (0.58) | -7.8 (0.61)
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | -5.8 (0.59) | -6.8 (0.55) | -7.5 (0.57) | -8.3 (0.57) | -8.7 (0.60) | -6.8 (0.60) | -7.7 (0.56) | -7.9 (0.58)
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | -5.6 (0.60) | -7.0 (0.57) | -7.1 (0.59) | -8.3 (0.59) | -8.7 (0.62) | -7.2 (0.62) | -7.8 (0.58) | -8.0 (0.60)
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | -5.7 (0.59) | -7.0 (0.56) | -7.5 (0.58) | -8.7 (0.58) | -8.6 (0.61) | -7.3 (0.60) | -8.0 (0.56) | -8.0 (0.59)
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | -5.7 (0.58) | -7.1 (0.54) | -7.6 (0.57) | -8.5 (0.57) | -8.8 (0.59) | -7.4 (0.59) | -8.0 (0.55) | -8.1 (0.57)
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | -4.7 (0.65) | -5.9 (0.58) | -5.1 (0.60) | -4.9 (0.63) | -5.7 (0.64) | -6.1 (0.65) | -5.9 (0.62) | -5.5 (0.61)
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | -4.4 (0.65) | -5.2 (0.58) | -4.5 (0.60) | -4.5 (0.63) | -5.0 (0.64) | -5.6 (0.65) | -5.7 (0.63) | -5.1 (0.61)
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | -4.9 (0.62) | -4.5 (0.56) | -4.7 (0.58) | -4.2 (0.62) | -4.5 (0.62) | -4.6 (0.64) | -5.6 (0.61) | -4.7 (0.59)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0865, MMRM — LSM, SE, CI, & p-values come from an MMRM model with CFB as dependent variable & TG, visit and smoking status as factors & baseline measurement as a covariate, as well as interaction of treatment by week & interaction of baseline measurement by week; MMRM: Mixed Model Repeated Measures; LSMean difference = -1.4, 95% CI 2-sided [-2.92 to 0.20], Standard Error of Mean 0.79
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0009, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.7, 95% CI 2-sided [-4.22 to -1.10], Standard Error of Mean 0.79
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.00001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.5, 95% CI 2-sided [-5.06 to -1.94], Standard Error of Mean 0.79
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.00001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.0, 95% CI 2-sided [-5.63 to -2.47], Standard Error of Mean 0.80
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.2360, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-2.55 to 0.63], Standard Error of Mean 0.81
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0032, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.4, 95% CI 2-sided [-3.92 to -0.80], Standard Error of Mean -2.4
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.7, 95% CI 2-sided [-4.29 to -1.19], Standard Error of Mean 0.79
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.1318, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.2, 95% CI 2-sided [-2.86 to 0.38], Standard Error of Mean 0.82
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0014, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.7, 95% CI 2-sided [-4.30 to -1.04], Standard Error of Mean 0.83
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -3.2, 95% CI 2-sided [-4.82 to -1.58], Standard Error of Mean 0.82
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.6, 95% CI 2-sided [-5.30 to -2.00], Standard Error of Mean 0.84
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0752, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-3.15 to 0.15], Standard Error of Mean 0.84
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0343, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-3.38 to -0.13], Standard Error of Mean 0.83
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0049, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-3.95 to -0.71], Standard Error of Mean 0.82
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0285, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-3.50 to -0.20], Standard Error of Mean 0.84
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.0, 95% CI 2-sided [-4.69 to -1.37], Standard Error of Mean 0.85
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.5, 95% CI 2-sided [-5.14 to -1.84], Standard Error of Mean 0.85
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRm — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.0, 95% CI 2-sided [-5.65 to -2.28], Standard Error of Mean 0.86
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0169, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.1, 95% CI 2-sided [-3.74 to -0.37], Standard Error of Mean 0.86
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0049, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.4, 95% CI 2-sided [-4.04 to -0.73], Standard Error of Mean 0.84
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.8, 95% CI 2-sided [-4.48 to -1.18], Standard Error of Mean 0.84
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0428, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.7, 95% CI 2-sided [-3.36 to -0.06], Standard Error of Mean 0.84
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.0, 95% CI 2-sided [-4.65 to -1.34], Standard Error of Mean 0.84
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.00001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.2, 95% CI 2-sided [-4.88 to -1.58], Standard Error of Mean -0.84
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.1, 95% CI 2-sided [-5.73 to -2.37], Standard Error of Mean 0.85
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0225, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-3.64 to -0.28], Standard Error of Mean 0.85
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.8, 95% CI 2-sided [-4.49 to -1.19], Standard Error of Mean 0.84
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.1, 95% CI 2-sided [-4.70 to -1.42], Standard Error of Mean 0.84
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.1168, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.2, 95% CI 2-sided [-2.80 to 0.31], Standard Error of Mean 0.79
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0012, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-4.15 to -1.03], Standard Error of Mean 0.79
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.0, 95% CI 2-sided [-4.54 to -1.42], Standard Error of Mean 0.79
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.9, 95% CI 2-sided [-5.44 to -2.28], Standard Error of Mean 0.80
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0134, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-3.58 to -0.42], Standard Error of Mean 0.80
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0057, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-3.76 to -0.65], Standard Error of Mean 0.79
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0016, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.5, 95% CI 2-sided [-4.06 to -0.96], Standard Error of Mean 0.79
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.0843, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-2.94 to 0.19], Standard Error of Mean 0.79
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0035, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-3.90 to -0.77], Standard Error of Mean 0.80
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.1, 95% CI 2-sided [-4.66 to -1.52], Standard Error of Mean 0.80
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.7, 95% CI 2-sided [-5.28 to -2.10], Standard Error of Mean 0.81
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.0315, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.7, 95% CI 2-sided [-3.33 to -0.16], Standard Error of Mean 0.81
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0063, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-3.75 to -0.62], Standard Error of Mean 0.80
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.7, 95% CI 2-sided [-4.25 to -1.14], Standard Error of Mean 0.79
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.1090, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.3, 95% CI 2-sided [-2.89 to 0.29], Standard Error of Mean 0.81
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0018, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.5, 95% CI 2-sided [-4.14 to -0.95], Standard Error of Mean 0.81
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.9, 95% CI 2-sided [-4.54 to -1.34], Standard Error of Mean 0.81
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.8, 95% CI 2-sided [-5.40 to -2.15], Standard Error of Mean 0.83
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0231, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.9, 95% CI 2-sided [-3.50 to -0.26], Standard Error of Mean 0.82
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0056, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-3.86 to -0.67], Standard Error of Mean 0.81
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.8, 95% CI 2-sided [-4.35 to -1.17], Standard Error of Mean 0.81
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.3568, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-2.35 to 0.85], Standard Error of Mean 0.81
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0129, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-3.65 to -0.43], Standard Error of Mean 0.82
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0018, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-4.19 to -0.97], Standard Error of Mean 0.82
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.1, 95% CI 2-sided [-4.70 to -1.42], Standard Error of Mean 0.83
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.1004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-3.00 to 0.27], Standard Error of Mean 0.83
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0173, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-3.57 to -0.35], Standard Error of Mean 0.82
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0038, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.4, 95% CI 2-sided [-3.97 to -0.77], Standard Error of Mean 0.81
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.1767, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-2.57 to 0.48], Standard Error of Mean 0.78
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.0308, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.7, 95% CI 2-sided [-3.20 to -0.16], Standard Error of Mean 0.77
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0013, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.5, 95% CI 2-sided [-4.07 to -1.00], Standard Error of Mean 0.78
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.9, 95% CI 2-sided [-4.47 to -1.36], Standard Error of Mean 0.79
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.2109, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-2.55 to 0.56], Standard Error of Mean 0.79
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0152, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.9, 95% CI 2-sided [-3.44 to -0.37], Standard Error of Mean 0.78
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0075, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.1, 95% CI 2-sided [-3.61 to -0.56], Standard Error of Mean 0.77
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.0869, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-2.96 to 0.20], Standard Error of Mean 0.80
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.0520, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-3.14 to 0.01], Standard Error of Mean 0.80
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0009, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.7, 95% CI 2-sided [-4.30 to -1.12], Standard Error of Mean 0.81
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.1, 95% CI 2-sided [-4.68 to -1.46], Standard Error of Mean 0.82
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Wek 10; Test type: Superiority; p = 0.0456, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-3.25 to -0.03], Standard Error of Mean 0.82
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0073, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-3.76 to -0.59], Standard Error of Mean 0.81
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0026, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.4, 95% CI 2-sided [-4.01 to -0.86], Standard Error of Mean 0.80
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.0878, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.3, 95% CI 2-sided [-2.87 to 0.20], Standard Error of Mean 0.78
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0182, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.9, 95% CI 2-sided [-3.39 to -0.32], Standard Error of Mean 0.78
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.0, 95% CI 2-sided [-4.55 to -1.44], Standard Error of Mean 0.79
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.0, 95% CI 2-sided [-4.53 to -1.40], Standard Error of Mean 0.80
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0387, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.7, 95% CI 2-sided [-3.22 to -0.09], Standard Error of Mean 0.80
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0031, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-3.89 to -0.80], Standard Error of Mean 0.79
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0029, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-3.88 to -0.81], Standard Error of Mean 0.78
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.0653, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-2.90 to 0.09], Standard Error of Mean 0.76
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.0102, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-3.46 to -0.47], Standard Error of Mean 0.76
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.9, 95% CI 2-sided [-4.38 to -1.36], Standard Error of Mean 0.77
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.2, 95% CI 2-sided [-4.72 to -1.67], Standard Error of Mean 0.78
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.0231, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-3.30 to -0.25], Standard Error of Mean 0.78
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0021, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.4, 95% CI 2-sided [-3.88 to -0.87], Standard Error of Mean 0.78
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0021, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.4, 95% CI 2-sided [-3.88 to -0.87], Standard Error of Mean 0.76
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0013, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.5, 95% CI 2-sided [-3.96 to -0.97], Standard Error of Mean 0.76
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.1460, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.2, 95% CI 2-sided [-2.89 to 0.43], Standard Error of Mean 0.84
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.6066, MMMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-2.10 to 1.23], Standard Error of Mean 0.84
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.8422, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-1.88 to 1.54], Standard Error of Mean 0.87
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.2346, LSMean difference — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-2.74 to 0.67], Standard Error of Mean 0.87
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.1128, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-3.11 to 0.33], Standard Error of Mean 0.87
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.1811, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.2, 95% CI 2-sided [-2.89 to 0.55], Standard Error of Mean 0.87
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.3521, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-2.45 to 0.87], Standard Error of Mean 0.84
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.3570, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-2.44 to 0.88], Standard Error of Mean 0.84
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.9227, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -0.1, 95% CI 2-sided [-1.73 to 1.57], Standard Error of Mean 0.84
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.8894, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-1.84 to 1.60], Standard Error of Mean 0.87
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.5074, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-2.29 to 1.13], Standard Error of Mean 0.87
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.1753, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -1.2, 95% CI 2-sided [-2.91 to 0.53], Standard Error of Mean 0.87
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.1212, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-3.09 to 0.36], Standard Error of Mean 0.88
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.3702, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-2.41 to 0.90], Standard Error of Mean 0.84
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.6459, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.4, 95% CI 2-sided [-1.22 to 1.96], Standard Error of Mean 0.81
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.8248, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-1.40 to 1.75], Standard Error of Mean 0.80
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.4226, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.7, 95% CI 2-sided [-0.98 to 2.33], Standard Error of Mean 0.84
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.6469, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.4, 95% CI 2-sided [-1.25 to 2.01], Standard Error of Mean 0.83
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.7642, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.3, 95% CI 2-sided [-1.41 to 1.91], Standard Error of Mean 0.84
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.4068, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-2.36 to 0.966], Standard Error of Mean 0.84
Statistical Analysis 106: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.7974, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-1.37 to 1.78], Standard Error of Mean 0.80

6. Secondary Outcome: Change From Baseline in The Mean Frequency of Moderate and Severe VMS to Each Study Week
Description: as for outcome 1
Time Frame: Baseline and weeks 1, 2, 3, 5, 6, 7, 8, 9, 10, 11, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: VMS per day
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
VMS per day
  Week 1 | -2.1 (0.59) | -3.8 (0.56) | -5.3 (0.58) | -5.7 (0.57) | -6.4 (0.60) | -3.3 (0.60) | -4.7 (0.56) | -4.7 (0.58)
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | -3.7 (0.60) | -5.3 (0.57) | -6.8 (0.59) | -6.8 (0.58) | -7.3 (0.61) | -5.4 (0.61) | -6.0 (0.57) | -5.7 (0.59)
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | -3.7 (0.61) | -5.8 (0.58) | -7.3 (0.60) | -7.0 (0.59) | -7.7 (0.62) | -6.3 (0.62) | -6.9 (0.58) | -6.3 (0.60)
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | -4.5 (0.58) | -6.3 (0.55) | -7.6 (0.57) | -7.3 (0.56) | -8.3 (0.59) | -6.9 (0.59) | -7.3 (0.55) | -6.7 (0.57)
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | -4.8 (0.58) | -6.6 (0.55) | -7.5 (0.57) | -7.6 (0.57) | -8.3 (0.60) | -7.0 (0.60) | -7.5 (0.55) | -7.1 (0.58)
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | -4.9 (0.59) | -6.5 (0.56) | -7.7 (0.58) | -7.5 (0.58) | -8.4 (0.61) | -7.1 (0.60) | -7.4 (0.56) | -7.2 (0.59)
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | -5.5 (0.59) | -6.6 (0.56) | -7.6 (0.58) | -7.7 (0.58) | -8.3 (0.61) | -7.1 (0.61) | -7.7 (0.56) | -7.3 (0.59)
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | -5.7 (0.57) | -7.1 (0.54) | -7.7 (0.56) | -8.0 (0.56) | -8.4 (0.59) | -7.1 (0.59) | -7.9 (0.54) | -7.3 (0.57)
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | -5.4 (0.59) | -7.2 (0.56) | -7.5 (0.58) | -7.9 (0.58) | -8.3 (0.61) | -7.4 (0.60) | -7.8 (0.56) | -7.6 (0.59)
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | -5.5 (0.57) | -7.3 (0.54) | -7.8 (0.56) | -8.3 (0.56) | -8.3 (0.59) | -7.6 (0.58) | -8.0 (0.54) | -7.6 (0.57)
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | -4.4 (0.65) | -6.4 (0.58) | -5.4 (0.60) | -5.3 (0.63) | -5.7 (0.64) | -6.8 (0.65) | -6.0 (0.62) | -5.2 (0.61)
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | -4.1 (0.66) | -5.7 (0.60) | -4.5 (0.61) | -4.8 (0.65) | -5.0 (0.66) | -6.2 (0.67) | -5.8 (0.65) | -4.8 (0.63)
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | -4.6 (0.65) | -5.1 (0.59) | -4.5 (0.60) | -4.5 (0.65) | -4.4 (0.65) | -5.6 (0.67) | -5.5 (0.65) | -4.4 (0.61)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0297, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.7, 95% CI 2-sided [-3.23 to -0.17], Standard Error of Mean 0.78
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.1, 95% CI 2-sided [-4.66 to -1.58], Standard Error of Mean 0.78
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.00001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.6, 95% CI 2-sided [-5.10 to -2.02], Standard Error of Mean 0.78
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.2, 95% CI 2-sided [-5.78 to -2.66], Standard Error of Mean 0.79
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.1318, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.2, 95% CI 2-sided [-2.76 to 0.36], Standard Error of Mean 0.79
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0010, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-4.13 to -1.05], Standard Error of Mean 0.78
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0011, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-4.10 to -1.04], Standard Error of Mean 0.78
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0405, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-3.20 to -0.07], Standard Error of Mean 0.79
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.1, 95% CI 2-sided [-4.70 to -1.55], Standard Error of Mean 0.80
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -3.1, 95% CI 2-sided [-4.66 to -1.52], Standard Error of Mean 0.80
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.7, 95% CI 2-sided [-5.26 to -2.07], Standard Error of Mean 0.81
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0325, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.7, 95% CI 2-sided [-3.34 to -0.15], Standard Error of Mean 0.81
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0035, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.4, 95% CI 2-sided [-3.92 to -0.78], Standard Error of Mean 0.80
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0102, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.1, 95% CI 2-sided [-3.61 to -0.49], Standard Error of Mean 0.79
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0098, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.1, 95% CI 2-sided [-3.69 to -0.51], Standard Error of Mean 0.81
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.6, 95% CI 2-sided [-5.18 to -1.98], Standard Error of Mean 0.81
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.3, 95% CI 2-sided [-4.89 to -1.70], Standard Error of Mean 0.81
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.0, 95% CI 2-sided [-5.61 to -2.37], Standard Error of Mean 0.82
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0021, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-4.17 to -0.93], Standard Error of Mean 0.82
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.1, 95% CI 2-sided [-4.71 to -1.52], Standard Error of Mean 0.81
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0020, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.5, 95% CI 2-sided [-4.11 to -0.93], Standard Error of Mean 0.81
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.0210, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-3.27 to -0.27], Standard Error of Mean 0.76
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.1, 95% CI 2-sided [-4.59 to -1.58], Standard Error of Mean 0.77
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.88, 95% CI 2-sided [-4.34 to -1.33], Standard Error of Mean 0.77
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.8, 95% CI 2-sided [-5.29 to -2.23], Standard Error of Mean 0.73
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0023, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.4, 95% CI 2-sided [-3.91 to -0.86], Standard Error of Mean 0.77
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.7, 95% CI 2-sided [-4.25 to -1.24], Standard Error of Mean 0.76
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0036, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-3.73 to -0.74], Standard Error of Mean 0.76
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.0195, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-3.33 to -0.29], Standard Error of Mean 0.77
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.7, 95% CI 2-sided [-4.21 to -1.17], Standard Error of Mean 0.77
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.8, 95% CI 2-sided [-4.32 to -1.27], Standard Error of Mean 0.77
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.5, 95% CI 2-sided [-5.01 to -1.92], Standard Error of Mean 0.79
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.0061, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-3.71 to -0.62], Standard Error of Mean 0.78
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.7, 95% CI 2-sided [-4.19 to -1.14], Standard Error of Mean 0.77
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0030, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-3.81 to -0.78], Standard Error of Mean 0.77
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.0383, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-3.17 to -0.09], Standard Error of Mean 0.78
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.8, 95% CI 2-sided [-4.33 to -1.24], Standard Error of Mean 0.79
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0011, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-4.14 to -1.04], Standard Error of Mean 0.79
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.5, 95% CI 2-sided [-5.07 to -1.93], Standard Error of Mean 0.80
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0055, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-3.80 to -0.66], Standard Error of Mean 0.80
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0014, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.5, 95% CI 2-sided [-4.09 to -0.99], Standard Error of Mean 0.79
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0040, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-3.80 to -0.73], Standard Error of Mean 0.78
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.1502, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-2.68 to 0.41], Standard Error of Mean 0.78
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0057, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-3.74 to -0.64], Standard Error of Mean 0.79
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0054, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-3.76 to -0.66], Standard Error of Mean 0.79
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.8, 95% CI 2-sided [-4.38 to -1.22], Standard Error of Mean 0.80
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.0412, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-3.21 to -0.07], Standard Error of Mean 0.80
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0054, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-3.76 to -0.66], Standard Error of Mean 0.79
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0167, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.9, 95% CI 2-sided [-3.43 to -0.34], Standard Error of Mean 0.78
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.0533, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-2.94 to 0.02], Standard Error of Mean 0.75
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.0065, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.1, 95% CI 2-sided [-3.54 to -0.58], Standard Error of Mean 0.75
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0025, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-3.80 to -0.82], Standard Error of Mean 0.76
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0005, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.7, 95% CI 2-sided [-4.22 to -1.20], Standard Error of Mean 0.77
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.0541, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-2.99 to 0.03], Standard Error of Mean 0.77
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0039, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-3.69 to -0.71], Standard Error of Mean 0.76
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0245, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.7, 95% CI 2-sided [-3.18 to -0.22], Standard Error of Mean 0.75
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.0187, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-3.36 to -0.31], Standard Error of Mean 0.78
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.0060, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.1, 95% CI 2-sided [-3.68 to -0.62], Standard Error of Mean 0.78
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0014, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.5, 95% CI 2-sided [-4.06 to -0.98], Standard Error of Mean 0.78
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.9, 95% CI 2-sided [-4.49 to -1.37], Standard Error of Mean 0.79
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.0100, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.1, 95% CI 2-sided [-3.61 to -0.49], Standard Error of Mean 0.79
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0019, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.4, 95% CI 2-sided [-3.98 to -0.91], Standard Error of Mean 0.78
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0049, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-3.73 to -0.67], Standard Error of Mean 0.78
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.0186, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-3.25 to -0.30], Standard Error of Mean 0.75
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0024, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-3.77 to -0.82], Standard Error of Mean 0.75
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.8, 95% CI 2-sided [-4.28 to -1.30], Standard Error of Mean 0.76
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.8, 95% CI 2-sided [-4.30 to -1.29], Standard Error of Mean 0.77
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0058, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.1, 95% CI 2-sided [-3.63 to -0.62], Standard Error of Mean 0.76
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-4.04 to -1.7], Standard Error of Mean 0.75
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0050, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.1, 95% CI 2-sided [-3.59 to -0.64], Standard Error of Mean 0.75
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.0205, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-3.63 to -0.31], Standard Error of Mean 0.85
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.2818, MMMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-2.58 to 0.75], Standard Error of Mean 0.85
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.3102, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-2.60 to 0.83], Standard Error of Mean 0.87
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.1422, LSMean difference — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.3, 95% CI 2-sided [-2.99 to 0.43], Standard Error of Mean 0.87
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.0064, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.4, 95% CI 2-sided [-4.12 to -0.68], Standard Error of Mean 0.87
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.0752, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-3.28 to 0.16], Standard Error of Mean 0.87
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.3632, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-2.43 to 0.89], Standard Error of Mean 0.85
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.0625, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -1.6, 95% CI 2-sided [-3.32 to 0.09], Standard Error of Mean 0.87
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.6613, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-2.07 to 1.32], Standard Error of Mean 0.86
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.4209, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-2.48 to 1.04], Standard Error of Mean 0.90
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.3288, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -0.9, 95% CI 2-sided [-2.63 to 0.88], Standard Error of Mean 0.89
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.0202, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.1, 95% CI 2-sided [-3.86 to -0.33], Standard Error of Mean 0.90
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.0682, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-3.42 to 0.12], Standard Error of Mean 0.90
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.3912, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-2.44 to 0.96], Standard Error of Mean 0.86
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.4964, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-2.25 to 1.09], Standard Error of Mean 0.85
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.9830, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-1.64 to 1.68], Standard Error of Mean 0.84
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.9715, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-1.71 to 1.78], Standard Error of Mean 0.89
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.8715, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.1, 95% CI 2-sided [-1.58 to 1.86], Standard Error of Mean 0.87
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.2233, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-2.83 to 0.66], Standard Error of Mean 0.89
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.2882, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-2.69 to 0.80], Standard Error of Mean 0.89
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.8643, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.1, 95% CI [-1.52 to 1.80], Standard Error of Mean 0.84

7. Secondary Outcome: Change From Baseline in The Mean Severity of Mild, Moderate, and Severe VMS to Each Study Week
Description: Severity of mild, moderate & severe VMS per day was calculated as follows
  [(number of mild VMS × 1) + (number of moderate VMS × 2) + (number of severe VMS × 3)]/number of daily mild/moderate/severe VMS
  Mild VMS was defined as sensation of heat without sweating/dampness. If at night, participant did not wake up but later noticed damp sheets or clothing. Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot & was sweating & needed to take action Severity was zero for participants that had no moderate or severe VMS. Higher score indicates greater severity.
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
Score on a scale
  Week 1 | -0.2 (0.09) | -0.5 (0.08) | -0.5 (0.09) | -0.6 (0.09) | -0.8 (0.09) | -0.2 (0.09) | -0.5 (0.08) | -0.5 (0.09)
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | -0.2 (0.11) | -0.6 (0.11) | -0.7 (0.11) | -1.0 (0.11) | -1.1 (0.11) | -0.4 (0.11) | -0.7 (0.11) | -0.8 (0.11)
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | -0.3 (0.13) | -0.8 (0.12) | -0.9 (0.13) | -1.1 (0.12) | -1.2 (0.13) | -0.6 (0.13) | -0.9 (0.12) | -1.0 (0.13)
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | -0.3 (0.13) | -0.8 (0.12) | -1.0 (0.13) | -1.1 (0.13) | -1.4 (0.13) | -0.8 (0.13) | -0.9 (0.12) | -1.1 (0.13)
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | -0.5 (0.13) | -0.8 (0.13) | -1.0 (0.13) | -1.3 (0.13) | -1.5 (0.14) | -0.8 (0.14) | -0.9 (0.13) | -1.0 (0.13)
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | -0.5 (0.14) | -0.9 (0.13) | -1.0 (0.14) | -1.4 (0.14) | -1.6 (0.14) | -0.8 (0.14) | -1.0 (0.13) | -1.2 (0.14)
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | -0.5 (0.14) | -0.9 (0.14) | -1.1 (0.14) | -1.4 (0.14) | -1.6 (0.15) | -1.0 (0.14) | -1.0 (0.14) | -1.2 (0.14)
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | -0.7 (0.15) | -1.0 (0.14) | -1.2 (0.15) | -1.5 (0.15) | -1.6 (0.15) | -0.9 (0.15) | -1.1 (0.15) | -1.3 (0.15)
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | -0.8 (0.15) | -1.1 (0.14) | -1.1 (0.15) | -1.6 (0.15) | -1.6 (0.15) | -0.9 (0.15) | -1.2 (0.15) | -1.3 (0.15)
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | -0.7 (0.15) | -1.2 (0.14) | -1.1 (0.15) | -1.5 (0.15) | -1.7 (0.15) | -1.0 (0.15) | -1.2 (0.14) | -1.4 (0.15)
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | -0.7 (0.15) | -1.1 (0.14) | -1.1 (0.15) | -1.6 (0.15) | -1.8 (0.15) | -1.0 (0.15) | -1.2 (0.15) | -1.4 (0.15)
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | -0.8 (0.15) | -1.2 (0.15) | -1.3 (0.15) | -1.6 (0.15) | -1.6 (0.16) | -1.0 (0.15) | -1.3 (0.15) | -1.3 (0.15)
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | -0.1 (0.10) | -0.5 (0.09) | -0.3 (0.09) | -0.4 (0.09) | -0.3 (0.09) | -0.5 (0.10) | -0.4 (0.09) | -0.2 (0.09)
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | -0.1 (0.10) | -0.3 (0.08) | -0.2 (0.09) | -0.3 (0.09) | -0.1 (0.09) | -0.4 (0.09) | -0.3 (0.09) | -0.2 (0.09)
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 0.0 (0.10) | -0.2 (0.09) | -0.2 (0.09) | -0.4 (0.10) | -0.1 (0.09) | -0.5 (0.10) | -0.3 (0.10) | -0.1 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0104, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.53 to -0.07], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0060, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.56 to -0.09], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.71 to -0.24], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.85 to -0.38], Standard Error of Mean 0.12
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.6977, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.28 to 0.19], Standard Error of Mean 0.12
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0121, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.53 to -0.07], Standard Error of Mean 0.12
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0086, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.54 to -0.08], Standard Error of Mean 0.12
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0138, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.66 to -0.08], Standard Error of Mean 0.15
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0014, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.78 to -0.19], Standard Error of Mean 0.15
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -0.7, 95% CI 2-sided [-1.02 to -0.43], Standard Error of Mean 0.12
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.19 to -0.59], Standard Error of Mean 0.15
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.2831, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.46 to 0.14], Standard Error of Mean 0.15
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0051, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.72 to -0.13], Standard Error of Mean 0.15
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.81 to -0.22], Standard Error of Mean 0.15
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0058, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.83 to -0.14], Standard Error of Mean 0.17
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.97 to -0.28], Standard Error of Mean 0.18
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.14 to -0.46], Standard Error of Mean 0.17
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.27 to -0.57], Standard Error of Mean 0.18
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0807, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.66 to 0.04], Standard Error of Mean 0.18
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0014, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.91 to -0.22], Standard Error of Mean 0.18
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.02 to -0.34], Standard Error of Mean 0.17
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0046, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.85 to -0.16], Standard Error of Mean 0.18
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.99 to -0.29], Standard Error of Mean 0.18
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.14 to -0.45], Standard Error of Mean 0.18
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.14 to -0.70], Standard Error of Mean 0.18
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0209, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.77 to -0.06], Standard Error of Mean 0.18
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0011, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.93 to -0.24], Standard Deviation 0.18
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.07 to -0.38], Standard Error of Mean 0.18
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.0956, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.67 to 0.05], Standard Error of Mean 0.18
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0050, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.89 to -0.16], Standard Error of Mean 0.19
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.18 to -0.45], Standard Error of Mean 0.19
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.40 to -0.65], Standard Error of Mean 0.19
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0915, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.69 to 0.05], Standard Error of Mean 0.19
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0378, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.75 to -0.02], Standard Error of Mean 0.19
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0053, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.89 to -0.16], Standard Error of Mean 0.19
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.0614, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.83 to -0.08], Standard Error of Mean 0.19
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0040, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.92 to -0.18], Standard Error of Mean 0.19
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.33 to -0.58], Standard Error of Mean 0.19
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.47 to -0.71], Standard Error of Mean 0.19
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.0967, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.70 to 0.06], Standard Error of Mean 0.19
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0063, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.90 to -0.15], Standard Error of Mean 0.19
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.13 to -0.38], Standard Error of Mean 0.19
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.0632, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.75 to 0.02], Standard Error of Mean 0.20
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0020, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.00 to -0.23], Standard Error of Mean 0.20
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.29 to -0.51], Standard Error of Mean 0.20
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.48 to -0.69], Standard Error of Mean 0.20
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0308, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.82 to -0.04], Standard Error of Mean 0.20
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0105, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.89 to -0.12], Standard Error of Mean 0.20
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0010, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.03 to -0.26], Standard Error of Mean 0.20
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.1469, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.69 to 0.11], Standard Error of Mean 0.20
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0315, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.84 to -0.04], Standard Error of Mean 0.20
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.18 to -0.38], Standard Error of Mean 0.21
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.26 to -0.43], Standard Error of Mean 0.21
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.4494, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.56 to 0.25], Standard Error of Mean 0.21
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0595, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.79 to 0.02], Standard Error of Mean 0.20
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0065, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.96 to -0.16], Standard Error of Mean 0.20
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.0745, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.77 to 0.04], Standard Error of Mean 0.20
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.0540, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.80 to 0.01], Standard Error of Mean 0.21
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.22 to -0.41], Standard Error of Mean 0.21
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.26 to -0.43], Standard Error of Mean 0.21
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.5317, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.54 to 0.28], Standard Error of Mean 0.21
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0424, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.83 to -0.01], Standard Error of Mean 0.21
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0134, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.91 to -0.11], Standard Error of Mean 0.21
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.0300, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.84 to -0.04], Standard Error of Mean 0.20
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.0605, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.78 to 0.02], Standard Error of Mean 0.20
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.20 to -0.40], Standard Error of Mean 0.20
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.38 to -0.56], Standard Error of Mean 0.21
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Wek 10; Test type: Superiority; p = 0.1848, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.68 to 0.13], Standard Error of Mean 0.21
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0321, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.84 to -0.04], Standard Error of Mean 0.20
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0025, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.01 to -0.22], Standard Error of Mean 0.20
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.0441, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.81 to -0.01], Standard Error of Mean 0.20
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0422, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.82 to -0.01], Standard Error of Mean 0.20
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.27 to -0.45], Standard Error of Mean 0.21
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.44 to -0.62], Standard Error of Mean 0.21
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.1464, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.71 to 0.11], Standard Error of Mean 0.21
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0144, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.91 to -0.10], Standard Error of Mean 0.21
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0013, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.06 to -0.26], Standard Error of Mean 0.20
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.0596, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.80 to 0.02], Standard Error of Mean 0.21
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.0360, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.85 to -0.03], Standard Error of Mean 0.21
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.15 to -0.32], Standard Error of Mean 0.21
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.23 to -0.39], Standard Error of Mean 0.21
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.3227, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.62 to 0.21], Standard Error of Mean 0.21
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0220, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.89 to -0.07], Standard Error of Mean 0.21
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0380, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.84 to -0.02], Standard Error of Mean 0.21
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.0067, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.60 to -0.10], Standard Error of Mean 0.13
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.1227, MMMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.45 to 0.05], Standard Error of Mean 0.13
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.0208, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.57 to -0.05], Standard Error of Mean 0.13
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.2396, LSMean difference — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.41 to 0.10], Standard Error of Mean 0.13
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.0022, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.67 to -0.15], Standard Error of Mean 0.13
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.0479, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.53 to -0.00], Standard Error of Mean 0.13
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.4152, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.35 to 0.15], Standard Error of Mean 0.13
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.0262, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -0.3, 95% CI 2-sided [-0.52 to -0.03], Standard Error of Mean 0.12
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.1210, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.43 to 0.05], Standard Error of Mean 0.12
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.0369, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.52 to -0.02], Standard Error of Mean 0.13
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.5855, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -0.1, 95% CI 2-sided [-0.32 to 0.18], Standard Error of Mean 0.13
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.0041, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.62 to -0.12], Standard Error of Mean 0.13
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.0614, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.50 to 0.01], Standard Error of Mean 0.13
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.3391, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.36 to 0.12], Standard Error of Mean 0.12
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.0515, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.49 to 0.00], Standard Error of Mean 0.12
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.0667, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.47 to 0.02], Standard Error of Mean 0.12
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.0047, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.63 to -0.12], Standard Error of Mean 0.13
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.5130, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.34 to 0.17], Standard Error of Mean 0.13
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.75 to -0.23], Standard Error of Mean 0.13
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.0126, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.60 to -0.07], Standard Error of Mean 0.13
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.3507, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.36 to 0.13], Standard Error of Mean 0.12

8. Secondary Outcome: Change From Baseline in The Mean Severity of Moderate and Severe VMS to Each Study Week
Description: Severity of moderate to severe VMS per day was calculated as follows:
  [(number of moderate VMS × 2) + (number of severe VMS × 3)]/number of daily moderate/severe VMS.
  Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed). Severity was zero for patients that had no moderate or severe VMS. Higher score indicates greater severity.
Time Frame: Baseline and weeks 1, 2, 3, 5, 6, 7, 8, 9, 10, 11, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
Score on a scale
  Week 1 | -0.1 (0.10) | -0.4 (0.09) | -0.5 (0.10) | -0.6 (0.10) | -0.8 (0.10) | -0.1 (0.10) | -0.4 (0.09) | -0.4 (0.10)
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | -0.2 (0.12) | -0.5 (0.12) | -0.7 (0.12) | -1.0 (0.12) | -1.2 (0.13) | -0.3 (0.13) | -0.6 (0.12) | -0.8 (0.12)
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | -0.2 (0.14) | -0.7 (0.14) | -1.0 (0.14) | -1.2 (0.14) | -1.3 (0.15) | -0.6 (0.14) | -0.8 (0.14) | -1.0 (0.14)
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | -0.5 (0.15) | -0.8 (0.14) | -1.1 (0.15) | -1.4 (0.15) | -1.6 (0.15) | -0.9 (0.15) | -0.8 (0.14) | -1.1 (0.15)
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | -0.5 (0.15) | -0.9 (0.15) | -1.1 (0.15) | -1.5 (0.15) | -1.6 (0.16) | -0.9 (0.15) | -1.0 (0.15) | -1.3 (0.15)
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | -0.5 (0.15) | -0.9 (0.15) | -1.2 (0.15) | -1.5 (0.15) | -1.7 (0.16) | -1.0 (0.16) | -1.0 (0.15) | -1.2 (0.15)
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | -0.7 (0.16) | -1.0 (0.15) | -1.2 (0.16) | -1.6 (0.16) | -1.6 (0.17) | -0.9 (0.16) | -1.2 (0.16) | -1.3 (0.16)
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | -0.8 (0.16) | -1.1 (0.15) | -1.2 (0.16) | -1.6 (0.16) | -1.7 (0.16) | -0.9 (0.16) | -1.2 (0.15) | -1.3 (0.16)
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | -0.8 (0.16) | -1.2 (0.15) | -1.2 (0.16) | -1.7 (0.16) | -1.8 (0.16) | -1.1 (0.16) | -1.2 (0.15) | -1.4 (0.16)
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | -0.8 (0.16) | -1.1 (0.15) | -1.2 (0.16) | -1.7 (0.16) | -1.8 (0.16) | -1.1 (0.16) | -1.3 (0.15) | -1.5 (0.16)
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | -0.1 (0.13) | -0.5 (0.12) | -0.3 (0.12) | -0.6 (0.13) | -0.3 (0.13) | -0.6 (0.13) | -0.4 (0.13) | -0.2 (0.12)
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | -0.1 (0.13) | -0.3 (0.11) | -0.3 (0.11) | -0.5 (0.12) | -0.1 (0.12) | -0.5 (0.13) | -0.3 (0.13) | -0.2 (0.12)
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 0.0 (0.13) | -0.2 (0.12) | -0.3 (0.12) | -0.6 (0.13) | -0.1 (0.13) | -0.5 (0.13) | -0.4 (0.13) | -0.1 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0098, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.60 to -0.08], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0048, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.63 to -0.11], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.80 to -0.28], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.00 to -0.47], Standard Error of Mean 0.13
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.6761, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.32 to 0.21], Standard Error of Mean 0.12
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0188, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.57 to -0.05], Standard Error of Mean 0.13
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0067, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.61 to -0.10], Standard Error of Mean 0.13
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0335, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.68 to -0.03], Standard Error of Mean 0.17
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.91 to -0.25], Standard Error of Mean 0.17
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -0.8, 95% CI 2-sided [-1.14 to -0.48], Standard Error of Mean 0.17
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.41 to -0.74], Standard Error of Mean 0.17
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.3227, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.50 to 0.17], Standard Error of Mean 0.17
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0085, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.77 to -0.11], Standard Error of Mean 0.17
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.95 to -0.30], Standard Error of Mean 0.17
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0102, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.87 to -0.12], Standard Error of Mean 0.19
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.15 to -0.39], Standard Error of Mean 0.19
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.29 to -0.54], Standard Error of Mean 0.19
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.46 to -0.68], Standard Error of Mean 0.20
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0740, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.73 to 0.03], Standard Error of Mean 0.20
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0024, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.97 to -0.21], Standard Error of Mean 0.19
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.17 to -0.41], Standard Error of Mean 0.19
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.1197, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.72 to 0.08], Standard Error of Mean 0.20
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0046, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.98 to -0.18], Standard Error of Mean 0.20
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.28 to -0.47], Standard Error of Mean 0.20
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.51 to -0.69], Standard Error of Mean 0.21
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0553, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.80 to 0.01], Standard Error of Mean 0.21
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0823, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.76 to 0.05], Standard Error of Mean 0.20
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0060, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.96 to -0.16], Standard Error of Mean 0.20
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.0374, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.83 to -0.03], Standard Error of Mean 0.21
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0042, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.00 to -0.19], Standard Error of Mean 0.21
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.38 to -0.56], Standard Error of Mean 0.21
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.54 to -0.71], Standard Error of Mean 0.21
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.0710, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.79 to 0.03], Standard Error of Mean 0.21
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0160, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.91 to -0.09], Standard Error of Mean 0.21
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.15 to -0.34], Standard Error of Mean 0.21
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.1013, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.76 to 0.07], Standard Error of Mean 0.21
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0011, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.11 to -0.28], Standard Error of Mean 0.21
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.36 to -0.53], Standard Error of Mean 0.21
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.57 to -0.72], Standard Error of Mean 0.22
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0476, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.85 to -0.00], Standard Error of Mean 0.21
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0220, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.90 to -0.07], Standard Error of Mean 0.21
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0019, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.07 to -0.24], Standard Error of Mean 0.21
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.1457, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.74 to 0.11], Standard Error of Mean 0.22
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0284, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.91 to -0.05], Standard Error of Mean 0.22
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.26 to -0.39], Standard Error of Mean 0.22
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.36 to -0.48], Standard Error of Mean 0.22
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.4223, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.61 to 0.26], Standard Error of Mean 0.22
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0442, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.87 to -0.01], Standard Error of Mean 0.22
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0071, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.02 to -0.16], Standard Error of Mean 0.22
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.0823, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.80 to 0.05], Standard Error of Mean 0.22
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.0336, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.89 to -0.04], Standard Error of Mean 0.22
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.32 to -0.46], Standard Error of Mean 0.22
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.34 to -0.47], Standard Error of Mean 0.22
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.4819, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.59 to 0.28], Standard Error of Mean 0.22
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0371, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.88 to -0.03], Standard Error of Mean 0.22
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0121, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.97 to -0.12], Standard Error of Mean 0.22
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.0281, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.89 to -0.05], Standard Error of Mean 0.21
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.0436, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.86 to -0.01], Standard Error of Mean 0.22
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.34 to -0.49], Standard Error of Mean 0.22
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.47 to -0.60], Standard Error of Mean 0.22
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Wek 10; Test type: Superiority; p = 0.1488, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.75 to 0.11], Standard Error of Mean 0.22
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0251, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.91 to -0.06], Standard Error of Mean 0.22
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0027, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.08 to -0.23], Standard Error of Mean 0.22
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.1053, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.77 to 0.07], Standard Error of Mean 0.22
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0304, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.90 to -0.04], Standard Error of Mean 0.22
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.33 to -0.43], Standard Error of Mean 0.22
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.49 to -0.61], Standard Error of Mean 0.22
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0873, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.81 to 0.06], Standard Error of Mean 0.22
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0124, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.97 to -0.12], Standard Error of Mean 0.22
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0014, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.12 to -0.27], Standard Error of Mean 0.22
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.0479, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.68 to -0.00], Standard Error of Mean 0.17
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.2342, MMMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.54 to 0.13], Standard Error of Mean 0.17
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.0070, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.84 to -0.13], Standard Error of Mean 0.18
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.4291, LSMean difference — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.49 to 0.21], Standard Error of Mean 0.18
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.0076, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.83 to -0.13], Standard Error of Mean 0.18
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.1506, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.62 to 0.10], Standard Error of Mean 0.18
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.5479, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.44 to 0.24], Standard Error of Mean 0.17
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.1427, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -0.2, 95% CI 2-sided [-0.57 to 0.08], Standard Error of Mean 0.17
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.1498, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.56 to 0.09], Standard Error of Mean 0.16
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.0103, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.79 to -0.11], Standard Error of Mean 0.17
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.8984, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -0.0, 95% CI 2-sided [-0.36 to 0.32], Standard Error of Mean 0.17
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.0095, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.79 to -0.11], Standard Error of Mean 0.17
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.1370, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.60 to 0.08], Standard Error of Mean 0.17
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.4223, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.46 to 0.19], Standard Error of Mean 0.17
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.3265, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.50 to 0.17], Standard Error of Mean 0.17
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.0852, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.62 to 0.04], Standard Error of Mean 0.17
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.0021, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.91 to -0.21], Standard Error of Mean 0.18
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.5717, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.45 to 0.25], Standard Error of Mean 0.18
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.0084, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.82 to -0.12], Standard Error of Mean 0.18
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.0277, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.75 to -0.04], Standard Error of Mean 0.18
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.4627, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.46 to 0.21], Standard Error of Mean 0.17

9. Secondary Outcome: Change From Baseline in The Hot Flash Score of Mild, Moderate, and Severe VMS to Each Study Week
Description: The hot flash score per 24h (or 12 h day time or 12 h night time) of VMS (mild, moderate, and severe) is calculated as follows:
  (number of mild VMS x 1) + (number of moderate VMS x 2) + (number of severe VMS x 3).
  Mild VMS was defined as sensation of heat without sweating/dampness. If at night, participant did not wake up but later noticed damp sheets or clothing.
  Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed). Higher score indicates greater severity.
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
Score on a scale
  Week 1 | -5.0 (1.48) | -9.8 (1.39) | -12.9 (1.45) | -14.1 (1.42) | -15.5 (1.50) | -8.4 (1.50) | -11.9 (1.39) | -11.9 (1.45)
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | -8.9 (1.50) | -13.0 (1.41) | -16.5 (1.47) | -17.0 (1.44) | -18.1 (1.52) | -13.5 (1.52) | -14.8 (1.41) | -14.5 (1.47)
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | -8.9 (1.54) | -14.5 (1.45) | -17.6 (1.51) | -17.7 (1.48) | -19.1 (1.57) | -15.4 (1.56) | -16.6 (1.45) | -15.9 (1.51)
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | -9.5 (1.53) | -14.9 (1.45) | -17.9 (1.51) | -17.6 (1.47) | -19.7 (1.57) | -15.9 (1.56) | -17.7 (1.45) | -17.1 (1.51)
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | -10.6 (1.45) | -15.4 (1.37) | -18.4 (1.43) | -18.6 (1.40) | -20.5 (1.49) | -16.9 (1.48) | -17.8 (1.37) | -17.2 (1.44)
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | -11.6 (1.44) | -16.4 (1.36) | -18.4 (1.42) | -19.4 (1.39) | -20.6 (1.48) | -16.9 (1.47) | -18.2 (1.36) | -18.1 (1.43)
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | -11.8 (1.46) | -16.2 (1.38) | -18.9 (1.44) | -19.1 (1.41) | -20.9 (1.50) | -17.4 (1.49) | -18.2 (1.39) | -18.3 (1.45)
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | -13.0 (1.46) | -16.3 (1.38) | -18.9 (1.44) | -19.5 (1.42) | -20.5 (1.51) | -17.4 (1.50) | -18.8 (1.39) | -18.7 (1.45)
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | -13.6 (1.40) | -17.6 (1.32) | -19.0 (1.37) | -20.2 (1.36) | -20.9 (1.44) | -17.3 (1.43) | -19.3 (1.33) | -18.7 (1.39)
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | -13.1 (1.44) | -17.9 (1.37) | -18.5 (1.42) | -20.1 (1.41) | -20.8 (1.49) | -18.2 (1.48) | -19.4 (1.38) | -19.1 (1.44)
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | -13.2 (1.41) | -17.9 (1.33) | -19.2 (1.39) | -20.9 (1.38) | -20.8 (1.46) | -18.6 (1.45) | -19.9 (1.35) | -19.2 (1.41)
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | -13.1 (1.38) | -18.2 (1.31) | -19.2 (1.36) | -20.7 (1.35) | -21.3 (1.43) | -18.7 (1.42) | -19.8 (1.32) | -19.4 (1.38)
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | -10.7 (1.63) | -16.0 (1.46) | -13.6 (1.51) | -12.7 (1.57) | -14.4 (1.61) | -16.3 (1.62) | -15.3 (1.56) | -13.3 (1.54)
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | -10.0 (1.66) | -14.1 (1.50) | -11.5 (1.53) | -11.5 (1.63) | -12.5 (1.66) | -15.3 (1.67) | -14.7 (1.62) | -12.3 (1.57)
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | -11.0 (1.59) | -12.3 (1.46) | -11.7 (1.48) | -10.8 (1.61) | -11.0 (1.60) | -13.6 (1.65) | -14.2 (1.59) | -10.9 (1.51)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0142, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.8, 95% CI 2-sided [-8.62 to -0.97], Standard Error of Mean 1.94
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.9, 95% CI 2-sided [-11.73 to -4.05], Standard Error of Mean 1.95
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -9.1, 95% CI 2-sided [-12.98 to -5.31], Standard Error of Mean 1.95
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -10.5, 95% CI 2-sided [-14.39 to -6.61], Standard Error of Mean 1.98
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.0819, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.5, 95% CI 2-sided [-7.36 to 0.44], Standard Error of Mean 1.98
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.9, 95% CI 2-sided [-10.78 to -3.09], Standard Error of Mean 1.95
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0005, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.9, 95% CI 2-sided [-10.69 to -3.05], Standard Error of Mean 1.94
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0380, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.1, 95% CI 2-sided [-8.01 to -0.23], Standard Error of Mean 1.98
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.6, 95% CI 2-sided [-11.46 to -3.64], Standard Error of Mean 1.99
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -8.1, 95% CI 2-sided [-11.96 to -4.17], Standard Error of Mean 1.98
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -9.2, 95% CI 2-sided [-13.17 to -5.25], Standard Error of Mean 2.01
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0245, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.6, 95% CI 2-sided [-8.52 to -0.59], Standard Error of Mean 2.02
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0031, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.9, 95% CI 2-sided [-9.83 to -2.01], Standard Error of Mean 1.99
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0046, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.6, 95% CI 2-sided [-9.53 to -1.75], Standard Error of Mean 1.98
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0064, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.6, 95% CI 2-sided [-9.61 to -1.59], Standard Error of Mean 2.04
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.7, 95% CI 2-sided [-12.72 to -4.65], Standard Error of Mean 2.05
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.8, 95% CI 2-sided [-12.78 to -4.75], Standard Error of Mean 2.04
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -10.2, 95% CI 2-sided [-14.27 to -6.09], Standard Error of Mean 2.08
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0021, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.4, 95% CI 2-sided [-10.54 to -2.36], Standard Error of Mean 2.08
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.7, 95% CI 2-sided [-11.71 to -3.66], Standard Error of Mean 2.05
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.0, 95% CI 2-sided [-10.96 to -2.95], Standard Error of Mean 2.04
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0075, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.5, 95% CI 2-sided [-9.46 to -1.47], Standard Error of Mean 2.03
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.4, 95% CI 2-sided [-12.44 to -4.42], Standard Error of Mean 2.04
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.2, 95% CI 2-sided [-12.15 to -4.16], Standard Error of Mean 2.03
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -10.2, 95% CI 2-sided [-14.30 to -6.16], Standard Error of Mean 2.07
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0021, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.4, 95% CI 2-sided [-10.46 to -2.34], Standard Error of Mean 2.06
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.3, 95% CI 2-sided [-12.25 to -4.25], Standard Error of Mean 0.18
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.6, 95% CI 2-sided [-11.58 to -3.62], Standard Error of Mean 2.02
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.0123, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.8, 95% CI 2-sided [-8.60 to -1.05], Standard Error of Mean 1.92
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.8, 95% CI 2-sided [-11.63 to -4.07], Standard Error of Mean 1.92
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.0, 95% CI 2-sided [-11.80 to -4.23], Standard Error of Mean 1.92
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -9.9, 95% CI 2-sided [-13.73 to -6.03], Standard Error of Mean 1.95
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0013, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.3, 95% CI 2-sided [-10.13 to -2.47], Standard Error of Mean 1.95
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.2, 95% CI 2-sided [-10.97 to -3.41], Standard Error of Mean 1.92
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.7, 95% CI 2-sided [-10.41 to -2.89], Standard Error of Mean 1.91
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.0119, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.8, 95% CI 2-sided [-8.54 to -1.07], Standard Error of Mean 1.90
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.8, 95% CI 2-sided [-10.58 to -3.09], Standard Error of Mean 1.90
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.8, 95% CI 2-sided [-11.57 to -4.06], Standard Error of Mean 1.91
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -9.1, 95% CI 2-sided [-12.89 to -5.27], Standard Error of Mean 1.94
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.0057, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.4, 95% CI 2-sided [-9.18 to -1.58], Standard Error of Mean 1.93
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.7, 95% CI 2-sided [-10.40 to -2.90], Standard Error of Mean 1.91
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.5, 95% CI 2-sided [-10.27 to -2.81], Standard Error of Mean 1.89
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.0210, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.5, 95% CI 2-sided [-8.27 to -0.68], Standard Error of Mean 1.93
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.2, 95% CI 2-sided [-10.98 to -3.38], Standard Error of Mean 1.93
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.3, 95% CI 2-sided [-11.12 to -3.49], Standard Error of Mean 1.94
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -9.1, 95% CI 2-sided [-12.99 to -5.25], Standard Error of Mean 1.97
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0047, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.6, 95% CI 2-sided [-9.45 to -1.73], Standard Error of Mean 1.96
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0009, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.5, 95% CI 2-sided [-10.29 to -2.67], Standard Error of Mean 1.94
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.5, 95% CI 2-sided [-10.28 to -2.71], Standard Error of Mean 1.92
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.0889, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.3, 95% CI 2-sided [-7.10 to 0.51], Standard Error of Mean 1.93
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0023, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.9, 95% CI 2-sided [-9.76 to -2.13], Standard Error of Mean 1.94
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0009, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.5, 95% CI 2-sided [-10.36 to -2.71], Standard Error of Mean 1.94
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.5, 95% CI 2-sided [-11.36 to -3.58], Standard Error of Mean 1.98
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.0255, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.4, 95% CI 2-sided [-8.30 to -0.55], Standard Error of Mean 1.97
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0031, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.8, 95% CI 2-sided [-9.63 to -1.98], Standard Error of Mean 1.94
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0037, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.7, 95% CI 2-sided [-9.45 to -1.85], Standard Error of Mean 1.93
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.0316, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.0, 95% CI 2-sided [-7.59 to -0.35], Standard Error of Mean 1.84
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.0036, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.4, 95% CI 2-sided [-9.02 to -1.78], Standard Error of Mean 1.84
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.6, 95% CI 2-sided [-10.23 to -2.94], Standard Error of Mean 1.85
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.2, 95% CI 2-sided [-10.93 to -3.54], Standard Error of Mean 1.88
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.0502, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.7, 95% CI 2-sided [-7.37 to 0.00], Standard Error of Mean 1.87
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0025, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.6, 95% CI 2-sided [-9.28 to -1.99], Standard Error of Mean 1.85
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0063, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.1, 95% CI 2-sided [-8.67 to -1.44], Standard Error of Mean 1.84
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.0117, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.8, 95% CI 2-sided [-8.58 to -1.08], Standard Error of Mean 1.90
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.0047, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.4, 95% CI 2-sided [-9.17 to -1.67], Standard Error of Mean 1.91
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.0, 95% CI 2-sided [-10.80 to -3.23], Standard Error of Mean 1.92
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.7, 95% CI 2-sided [-11.51 to -3.86], Standard Error of Mean 1.94
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Wek 10; Test type: Superiority; p = 0.0083, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.2, 95% CI 2-sided [-8.97 to -1.34], Standard Error of Mean 1.94
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0011, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.3, 95% CI 2-sided [-10.10 to -2.56], Standard Error of Mean 1.92
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0017, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.0, 95% CI 2-sided [-9.77 to -2.29], Standard Error of Mean 1.90
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.0119, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.7, 95% CI 2-sided [-8.37 to -1.05], Standard Error of Mean 1.86
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0015, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.0, 95% CI 2-sided [-9.61 to -2.29], Standard Error of Mean 1.86
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.7, 95% CI 2-sided [-11.38 to -3.99], Standard Error of Mean 1.88
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.6, 95% CI 2-sided [-11.33 to -3.87], Standard Error of Mean 1.90
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0051, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.3, 95% CI 2-sided [-9.07 to -1.62], Standard Error of Mean 1.89
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.6, 95% CI 2-sided [-10.33 to -2.96], Standard Error of Mean 1.87
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0014, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.0, 95% CI 2-sided [-9.64 to -2.34], Standard Error of Mean 1.86
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.0054, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.1, 95% CI 2-sided [-8.67 to -1.51], Standard Error of Mean 1.82
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.1, 95% CI 2-sided [-9.71 to -2.55], Standard Error of Mean 1.82
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.6, 95% CI 2-sided [-11.20 to -3.97], Standard Error of Mean 1.84
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.2, 95% CI 2-sided [-11.88 to -4.59], Standard Error of Mean 1.85
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.0026, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.6, 95% CI 2-sided [-9.27 to -1.99], Standard Error of Mean 1.85
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.8, 95% CI 2-sided [-10.35 to -3.16], Standard Error of Mean 1.83
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.3, 95% CI 2-sided [-9.88 to -2.75], Standard Error of Mean 1.81
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.0126, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.3, 95% CI 2-sided [-9.48 to -1.15], Standard Error of Mean 2.12
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.1724, MMMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.9, 95% CI 2-sided [-7.06 to 1.27], Standard Error of Mean 2.12
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.3548, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-6.31 to 2.27], Standard Error of Mean 2.18
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.0860, LSMean difference — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.8, 95% CI 2-sided [-8.04 to 0.53], Standard Error of Mean 2.18
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.0111, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.6, 95% CI 2-sided [-9.89 to -1.28], Standard Error of Mean 2.19
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.0349, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.6, 95% CI 2-sided [-8.94 to -0.33], Standard Error of Mean 2.19
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.2205, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-6.77 to 1.57], Standard Error of Mean 2.12
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.0645, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -4.0, 95% CI 2-sided [-8.29 to 0.24], Standard Error of Mean 2.17
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.5031, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-5.69 to 2.80], Standard Error of Mean 2.16
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.5263, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-5.84 to 2.99], Standard Error of Mean 2.24
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.2782, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -2.4, 95% CI 2-sided [-6.83 to 1.97], Standard Error of Mean 2.24
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.0198, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.3, 95% CI 2-sided [-9.67 to -0.84], Standard Error of Mean 2.24
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.0417, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.6, 95% CI 2-sided [-9.05 to -0.18], Standard Error of Mean 2.25
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.2963, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-6.52 to 2.00], Standard Error of Mean 2.16
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.5408, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.3, 95% CI 2-sided [-5.39 to 2.83], Standard Error of Mean 2.09
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.7473, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-4.74 to 3.41], Standard Error of Mean 2.07
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.9214, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-4.07 to 4.50], Standard Error of Mean 2.18
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.9876, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-4.19 to 4.26], Standard Error of Mean 2.14
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.2379, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-6.86 to 1.71], Standard Error of Mean 2.18
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.1491, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.2, 95% CI 2-sided [-7.45 to 1.14], Standard Error of Mean 2.18
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.9560, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.1, 95% CI 2-sided [-3.96 to 4.19], Standard Error of Mean 2.07

10. Secondary Outcome: Change From Baseline in The Hot Flash Score of Moderate and Severe VMS to Each Study Week
Description: The hot flash score per 24h of moderate and severe VMS is calculated as follows:
  (number of moderate VMS x 2) + (number of severe VMS x 3).
  Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed). VMS. Baseline is the average frequency of 24h vasomotor symptom from 7 non-missing days prior to Day 1. Higher score indicates greater severity.
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
Score on a scale
  Week 1 | -5.1 (1.49) | -10.2 (1.40) | -13.4 (1.46) | -14.3 (1.43) | -15.7 (1.51) | -8.8 (1.51) | -12.2 (1.40) | -11.8 (1.46)
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | -8.9 (1.51) | -13.5 (1.41) | -17.0 (1.48) | -16.9 (1.44) | -18.2 (1.53) | -13.8 (1.53) | -15.5 (1.42) | -14.3 (1.48)
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | -8.9 (1.54) | -14.8 (1.45) | -18.2 (1.52) | -17.5 (1.48) | -19.1 (1.57) | -15.9 (1.57) | -17.3 (1.46) | -15.6 (1.52)
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | -9.5 (1.54) | -15.2 (1.46) | -18.3 (1.51) | -17.4 (1.48) | -19.6 (1.57) | -16.4 (1.56) | -18.0 (1.45) | -16.7 (1.51)
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | -10.5 (1.46) | -15.8 (1.38) | -18.8 (1.44) | -18.3 (1.41) | -20.3 (1.50) | -17.2 (1.49) | -18.2 (1.38) | -16.8 (1.45)
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | -11.5 (1.45) | -16.7 (1.37) | -18.7 (1.43) | -19.0 (1.40) | -20.3 (1.49) | -17.3 (1.48) | -18.6 (1.37) | -17.6 (1.44)
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | -11.8 (1.47) | -16.6 (1.39) | -19.2 (1.45) | -18.7 (1.42) | -20.6 (1.51) | -17.7 (1.50) | -18.5 (1.39) | -17.8 (1.46)
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | -13.0 (1.47) | -16.6 (1.38) | -19.1 (1.44) | -19.1 (1.42) | -20.2 (1.51) | -17.7 (1.50) | -19.0 (1.39) | -18.2 (1.46)
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | -13.5 (1.41) | -17.9 (1.33) | -19.3 (1.38) | -19.8 (1.37) | -20.5 (1.45) | -17.7 (1.44) | -19.4 (1.34) | -18.2 (1.40)
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | -12.9 (1.45) | -18.2 (1.37) | -18.9 (1.42) | -19.7 (1.41) | -20.4 (1.49) | -18.4 (1.48) | -19.5 (1.38) | -18.7 (1.44)
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | -13.0 (1.42) | -18.2 (1.34) | -19.4 (1.39) | -20.5 (1.38) | -20.5 (1.46) | -18.9 (1.45) | -19.9 (1.35) | -18.8 (1.41)
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | -12.8 (1.39) | -18.4 (1.31) | -19.3 (1.36) | -20.3 (1.36) | -21.0 (1.43) | -19.0 (1.42) | -19.8 (1.32) | -19.0 (1.38)
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | -10.4 (1.65) | -16.4 (1.49) | -13.8 (1.54) | -13.1 (1.60) | -14.4 (1.64) | -17.0 (1.65) | -15.4 (1.59) | -13.0 (1.56)
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | -9.7 (1.70) | -14.5 (1.53) | -11.5 (1.57) | -11.7 (1.66) | -12.5 (1.69) | -15.9 (1.70) | -14.6 (1.66) | -12.0 (1.60)
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | -10.7 (1.65) | -12.9 (1.51) | -11.6 (1.53) | -11.1 (1.67) | -10.9 (1.66) | -14.7 (1.71) | -14.1 (1.65) | -10.6 (1.56)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0089, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.2, 95% CI 2-sided [-9.01 to -1.30], Standard Error of Mean 1.96
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.4, 95% CI 2-sided [-12.22 to -4.48], Standard Error of Mean 1.97
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -9.2, 95% CI 2-sided [-13.06 to -5.34], Standard Error of Mean 1.96
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -10.7, 95% CI 2-sided [-14.58 to -6.75], Standard Error of Mean 1.99
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.0630, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.7, 95% CI 2-sided [-7.65 to 0.20], Standard Error of Mean 2.00
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.2, 95% CI 2-sided [-11.04 to -3.30], Standard Error of Mean 1.97
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.7, 95% CI 2-sided [-10.53 to -2.84], Standard Error of Mean 1.96
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0231, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.5, 95% CI 2-sided [-8.43 to -0.63], Standard Error of Mean 1.98
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.0, 95% CI 2-sided [-11.94 to -4.09], Standard Error of Mean 1.99
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -8.0, 95% CI 2-sided [-11.87 to -4.05], Standard Error of Mean 1.99
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -9.2, 95% CI 2-sided [-13.21 to -5.26], Standard Error of Mean 2.02
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0177, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.8, 95% CI 2-sided [-8.80 to -0.84], Standard Error of Mean 2.02
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0012, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.5, 95% CI 2-sided [-10.45 to -2.60], Standard Error of Mean 1.99
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0072, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.6, 95% CI 2-sided [-9.26 to -2.64], Standard Error of Mean 2.04
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0044, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.9, 95% CI 2-sided [-9.86 to -1.84], Standard Error of Mean 2.04
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -9.2, 95% CI 2-sided [-13.27 to -5.21], Standard Error of Mean 2.05
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.6, 95% CI 2-sided [-12.57 to -4.55], Standard Error of Mean 2.04
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -10.2, 95% CI 2-sided [-14.29 to -6.11], Standard Error of Mean 2.08
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0009, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.0, 95% CI 2-sided [-11.04 to -2.87], Standard Error of Mean 2.08
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.4, 95% CI 2-sided [-12.44 to -4.39], Standard Error of Mean 2.05
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0012, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.6, 95% CI 2-sided [-10.65 to -2.64], Standard Error of Mean 2.04
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0053, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.7, 95% CI 2-sided [-9.72 to -1.71], Standard Error of Mean 2.04
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.8, 95% CI 2-sided [-12.77 to -4.73], Standard Error of Mean 2.04
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.8, 95% CI 2-sided [-11.84 to -3.84], Standard Error of Mean 2.04
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -10.0, 95% CI 2-sided [-14.12 to -5.96], Standard Error of Mean 2.07
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0010, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.9, 95% CI 2-sided [-10.92 to -2.78], Standard Error of Mean 2.07
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.5, 95% CI 2-sided [-12.49 to -4.46], Standard Error of Mean 2.04
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0005, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.1, 95% CI 2-sided [-11.12 to -3.13], Standard Error of Mean 2.03
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.0057, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.4, 95% CI 2-sided [-9.15 to -1.58], Standard Error of Mean 1.93
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.4, 95% CI 2-sided [-12.15 to -4.56], Standard Error of Mean 1.93
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.9, 95% CI 2-sided [-11.68 to -4.08], Standard Error of Mean 1.93
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -9.8, 95% CI 2-sided [-13.66 to -5.93], Standard Error of Mean 1.96
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.7, 95% CI 2-sided [-10.54 to -2.85], Standard Error of Mean 1.95
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.7, 95% CI 2-sided [-11.55 to -3.95], Standard Error of Mean 1.93
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0010, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.4, 95% CI 2-sided [-10.16 to -2.60], Standard Error of Mean 1.92
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.0064, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.2, 95% CI 2-sided [-8.99 to -1.48], Standard Error of Mean 1.91
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.2, 95% CI 2-sided [-10.94 to -3.42], Standard Error of Mean 1.91
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.5, 95% CI 2-sided [-11.29 to -3.75], Standard Error of Mean 1.92
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.9, 95% CI 2-sided [-12.69 to -5.03], Standard Error of Mean 1.95
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.0030, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.8, 95% CI 2-sided [-9.62 to -1.99], Standard Error of Mean 1.94
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.1, 95% CI 2-sided [-10.92 to -3.37], Standard Error of Mean 1.92
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0013, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.2, 95% CI 2-sided [-9.91 to -2.42], Standard Error of Mean 1.90
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.0137, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.8, 95% CI 2-sided [-8.61 to -0.99], Standard Error of Mean 1.94
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.4, 95% CI 2-sided [-11.24 to -3.60], Standard Error of Mean 1.94
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.0, 95% CI 2-sided [-10.79 to -3.13], Standard Error of Mean 1.95
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.9, 95% CI 2-sided [-12.74 to -4.97], Standard Error of Mean 1.98
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0028, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.9, 95% CI 2-sided [-9.82 to -2.07], Standard Error of Mean 1.97
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.8, 95% CI 2-sided [-10.60 to -2.94], Standard Error of Mean 1.95
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0020, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.0, 95% CI 2-sided [-9.82 to -2.21], Standard Error of Mean 1.93
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.0588, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.7, 95% CI 2-sided [-7.46 to 0.14], Standard Error of Mean 1.93
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0018, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.7, 95% CI 2-sided [-9.90 to 0.14], Standard Error of Mean 1.93
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0017, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.2, 95% CI 2-sided [-9.98 to -2.34], Standard Error of Mean 1.94
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.2, 95% CI 2-sided [-11.09 to -3.32], Standard Error of Mean 1.97
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.0810, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.7, 95% CI 2-sided [-8.55 to -0.81], Standard Error of Mean 1.97
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0020, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.1, 95% CI 2-sided [-9.88 to -2.23], Standard Error of Mean 1.94
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0076, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.2, 95% CI 2-sided [-8.98 to -1.39], Standard Error of Mean 1.93
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.0182, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.4, 95% CI 2-sided [-8.01 to -0.75], Standard Error of Mean 1.85
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.0019, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.8, 95% CI 2-sided [-9.42 to -2.16], Standard Error of Mean 1.84
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.4, 95% CI 2-sided [-10.02 to -2.71], Standard Error of Mean 1.86
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.1, 95% CI 2-sided [-10.76 to -3.35], Standard Error of Mean 1.88
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.0263, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.2, 95% CI 2-sided [-7.89 to -0.50], Standard Error of Mean 1.88
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0015, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.0, 95% CI 2-sided [-9.61 to -2.29], Standard Error of Mean 1.86
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0113, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.7, 95% CI 2-sided [-8.32 to -1.07], Standard Error of Mean 1.84
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.0059, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.3, 95% CI 2-sided [-9.04 to -1.54], Standard Error of Mean 1.91
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.0018, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.0, 95% CI 2-sided [-9.76 to -2.25], Standard Error of Mean 1.91
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.8, 95% CI 2-sided [-10.62 to -3.05], Standard Error of Mean 1.93
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.6, 95% CI 2-sided [-11.39 to -3.73], Standard Error of Mean 1.95
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Wek 10; Test type: Superiority; p = 0.0044, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.6, 95% CI 2-sided [-9.40 to -1.75], Standard Error of Mean 1.94
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.6, 95% CI 2-sided [-10.40 to -2.84], Standard Error of Mean 1.92
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0025, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.8, 95% CI 2-sided [-9.57 to -2.07], Standard Error of Mean 1.91
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.0059, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.2, 95% CI 2-sided [-8.81 to -1.49], Standard Error of Mean 1.86
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.4, 95% CI 2-sided [-10.06 to -2.74], Standard Error of Mean 1.86
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.5, 95% CI 2-sided [-11.18 to -3.79], Standard Error of Mean 1.88
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.5, 95% CI 2-sided [-11.18 to -3.72], Standard Error of Mean 1.90
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0022, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.8, 95% CI 2-sided [-9.56 to -2.11], Standard Error of Mean 1.89
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.9, 95% CI 2-sided [-10.56 to -3.19], Standard Error of Mean 1.87
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0020, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.8, 95% CI 2-sided [-9.44 to -2.13], Standard Error of Mean 1.86
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.0023, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.6, 95% CI 2-sided [-9.18 to -2.01], Standard Error of Mean 1.82
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.5, 95% CI 2-sided [-10.06 to -2.89], Standard Error of Mean 1.82
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -7.4, 95% CI 2-sided [-11.05 to -3.81], Standard Error of Mean 1.84
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -8.1, 95% CI 2-sided [-11.80 to -4.49], Standard Error of Mean 1.86
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.0011, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.1, 95% CI 2-sided [-9.77 to -2.47], Standard Error of Mean 1.85
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.9, 95% CI 2-sided [-10.54 to -3.32], Standard Error of Mean 1.83
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.1, 95% CI 2-sided [-9.71 to -2.56], Standard Error of Mean 1.82
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.0054, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.0, 95% CI 2-sided [-10.26 to -1.80], Standard Error of Mean 2.15
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.1145, MMMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.4, 95% CI 2-sided [-7.63 to 0.83], Standard Error of Mean 2.15
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.2106, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.8, 95% CI 2-sided [-7.13 to 1.58], Standard Error of Mean 2.21
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.0685, LSMean difference — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.0, 95% CI 2-sided [-8.39 to 0.31], Standard Error of Mean 2.21
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.0029, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.7, 95% CI 2-sided [-11.02 to -2.29], Standard Error of Mean 2.22
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.0239, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -5.0, 95% CI 2-sided [-9.42 to -0.67], Standard Error of Mean 2.22
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.2224, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-6.86 to 1.60], Standard Error of Mean 2.15
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.0308, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -4.8, 95% CI 2-sided [-9.17 to -0.45], Standard Error of Mean 2.22
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.4194, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-6.13 to 2.56], Standard Error of Mean 2.21
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.3759, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-6.55 to 2.48], Standard Error of Mean 2.29
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.2285, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean differencce = -2.8, 95% CI 2-sided [-7.26 to 1.74], Standard Error of Mean 2.29
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.0072, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -6.2, 95% CI 2-sided [-10.71 to -1.70], Standard Error of Mean 2.29
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.0338, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.9, 95% CI 2-sided [-9.46 to -0.38], Standard Error of Mean 2.31
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.3026, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-6.64 to 2.07], Standard Error of Mean 2.21
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.3120, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-6.45 to 2.07], Standard Error of Mean 2.16
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.6816, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-5.11 to 3.34], Standard Error of Mean 2.15
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.8599, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-4.85 to 4.05], Standard Error of Mean 2.26
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.9093, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-4.64 to 4.13], Standard Error of Mean 2.23
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.0788, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -4.0, 95% CI 2-sided [-8.43 to 0.46], Standard Error of Mean 2.26
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.1278, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = -3.5, 95% CI 2-sided [-7.92 to 1.00], Standard Error of Mean 2.26
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.9848, MMRM — [p-value comment as in outcome 5, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-4.19 to 4.27], Standard Error of Mean 2.15

11. Secondary Outcome: Mean Percent Reduction of Mild, Moderate, And Severe Vasomotor Symptoms From Baseline to Each Study Week
Description: as for outcome 5
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Percent Reduction
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
Percent Reduction
  Week 1 | 14.5 (5.33) | 29.1 (5.01) | 37.6 (5.21) | 51.8 (5.12) | 55.5 (5.39) | 22.7 (5.40) | 40.1 (5.02) | 44.7 (5.22)
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 30.3 (5.30) | 46.2 (4.99) | 54.8 (5.20) | 64.0 (5.09) | 68.3 (5.39) | 44.8 (5.38) | 49.8 (5.01) | 56.1 (5.21)
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 32.0 (5.66) | 52.2 (5.37) | 60.3 (5.58) | 68.9 (5.44) | 72.5 (5.77) | 51.7 (5.75) | 56.9 (5.37) | 62.8 (5.56)
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 34.7 (5.58) | 55.3 (5.33) | 63.5 (5.52) | 68.1 (5.39) | 76.2 (5.72) | 54.5 (5.69) | 64.7 (5.30) | 67.9 (5.50)
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 41.3 (5.32) | 56.7 (5.08) | 66.1 (5.26) | 72.1 (5.17) | 80.1 (5.49) | 60.4 (5.42) | 63.6 (5.06) | 66.4 (5.28)
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 45.4 (5.01) | 60.0 (4.74) | 65.3 (4.93) | 75.1 (4.86) | 81.1 (5.16) | 60.1 (5.12) | 65.9 (4.75) | 72.0 (4.97)
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 45.1 (5.17) | 59.6 (4.92) | 68.1 (5.10) | 74.0 (5.05) | 81.9 (5.34) | 60.7 (5.29) | 66.3 (4.93) | 72.2 (5.14)
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 50.9 (5.13) | 60.5 (4.87) | 69.0 (5.05) | 76.1 (5.01) | 81.5 (5.32) | 62.1 (5.26) | 69.2 (4.90) | 74.5 (5.11)
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 53.8 (4.90) | 65.7 (4.64) | 68.4 (4.81) | 78.2 (4.78) | 83.4 (5.06) | 62.2 (5.03) | 72.3 (4.67) | 74.5 (4.88)
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 51.8 (5.03) | 67.6 (4.78) | 64.6 (4.95) | 77.6 (4.95) | 83.4 (5.20) | 66.1 (5.17) | 73.0 (4.82) | 76.2 (5.02)
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 53.5 (4.88) | 68.0 (4.63) | 68.8 (4.81) | 80.0 (4.81) | 83.4 (5.05) | 67.4 (5.02) | 75.4 (4.66) | 76.9 (4.87)
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 53.2 (4.87) | 68.0 (4.62) | 70.2 (4.80) | 79.6 (4.80) | 84.2 (5.04) | 68.0 (5.01) | 75.1 (4.65) | 76.4 (4.86)
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 43.6 (5.69) | 53.3 (5.07) | 45.9 (5.24) | 45.1 (5.47) | 50.7 (5.59) | 49.3 (5.66) | 54.0 (5.44) | 48.0 (5.32)
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 39.9 (6.12) | 42.0 (5.50) | 41.2 (5.60) | 39.6 (5.99) | 43.8 (6.08) | 41.5 (6.14) | 52.9 (6.01) | 47.0 (5.72)
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 45.0 (5.97) | 37.1 (5.49) | 42.9 (5.56) | 37.8 (6.06) | 39.4 (6.01) | 32.4 (6.21) | 51.4 (6.00) | 43.0 (5.64)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0388, MMRM — LSM, SE, CI, & p-values come from an MMRM model with PR from baseline as dependent variable & TG, visit and smoking status as factors & baseline measurement (BM) as a covariate, as well as interaction of treatment by week & interaction of BM by week; MMRM: Mixed Model Repeated Measures; LSMean difference = 14.6, 95% CI 2-sided [0.76 to 28.49], Standard Error of Mean 7.05
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0012, MMRM — LSM, SE, CI, & p-values come from an MMRM model with PR from baseline as dependent variable & TG, visit and smoking status as factors & BM as a covariate, as well as interaction of treatment by week & interaction of BM by week; LSMean difference = 23.1, 95% CI 2-sided [9.17 to 37.02], Standard Error of Mean 7.08
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 37.3, 95% CI 2-sided [23.41 to 51.22], Standard Error of Mean 7.07
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 41.0, 95% CI 2-sided [26.88 to 55.05], Standard Error of Mean 7.16
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.2569, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 8.2, 95% CI 2-sided [-5.98 to 22.32], Standard Error of Mean 7.19
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.6, 95% CI 2-sided [11.65 to 39.47], Standard Error of Mean 7.07
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 30.2, 95% CI 2-sided [16.39 to 44.06], Standard Error of Mean 7.03
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0240, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 15.9, 95% CI 2-sided [2.11 to 29.71], Standard Error of Mean 7.02
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 24.5, 95% CI 2-sided [10.62 to 38.37], Standard Error of Mean 7.05
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean differencce = 33.7, 95% CI 2-sided [19.87 to 47.52], Standard Error of Mean 7.03
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 38.0, 95% CI 2-sided [23.93 to 52.04], Standard Error of Mean 7.15
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0441, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 14.5, 95% CI 2-sided [0.38 to 28.53], Standard Error of Mean 7.16
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0061, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.4, 95% CI 2-sided [5.58 to 33.28], Standard Error of Mean 7.04
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.7, 95% CI 2-sided [11.96 to 39.53], Standard Error of Mean 7.01
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0078, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.2, 95% CI 2-sided [5.36 to 35.07], Standard Error of Mean 7.55
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 28.3, 95% CI 2-sided [13.36 to 43.22], Standard Error of Mean 7.59
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 36.9, 95% CI 2-sided [22.07 to 51.77], Standard Error of Mean 7.55
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRm — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 40.5, 95% CI 2-sided [25.41 to 55.67], Standard Error of Mean 7.69
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0108, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.7, 95% CI 2-sided [4.59 to 34.88], Standard Error of Mean 7.70
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0011, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.0, 95% CI 2-sided [10.09 to 39.84], Standard Error of Mean 7.56
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 30.9, 95% CI 2-sided [16.03 to 45.67], Standard Error of Mean 7.53
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0063, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.5, 95% CI 2-sided [5.84 to 35.23], Standard Error of Mean 7.47
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 28.7, 95% CI 2-sided [13.98 to 43.46], Standard Error of Mean 7.49
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 33.3, 95% CI 2-sided [18.66 to 48.00], Standard Error of Mean 7.46
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 41.5, 95% CI 2-sided [26.52 to 56.41], Standard Error of Mean 7.60
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0098, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.7, 95% CI 2-sided [4.78 to 34.66], Standard Error of Mean 7.59
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 29.9, 95% CI 2-sided [15.26 to 44.61], Standard Error of Mean 7.46
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 33.1, 95% CI 2-sided [18.50 to 47.73], Standard Error of Mean 7.43
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.0303, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 15.4, 95% CI 2-sided [1.48 to 29.40], Standard Error of Mean 7.10
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 24.8, 95% CI 2-sided [10.77 to 38.74], Standard Error of Mean 7.11
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 30.8, 95% CI 2-sided [16.77 to 44.75], Standard Error of Mean 7.11
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 38.8, 95% CI 2-sided [24.55 to 53.00], Standard Error of Mean 7.23
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0086, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.1, 95% CI 2-sided [4.88 to 33.23], Standard Error of Mean 7.20
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0018, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 22.3, 95% CI 2-sided [8.33 to 36.24], Standard Error of Mean 7.09
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.1, 95% CI 2-sided [11.24 to 39.05], Standard Error of Mean 7.07
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.0282, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 14.6, 95% CI 2-sided [1.56 to 27.60], Standard Error of Mean 6.62
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0029, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.9, 95% CI 2-sided [6.85 to 32.92], Standard Error of Mean 6.63
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 29.7, 95% CI 2-sided [16.58 to 42.73], Standard Error of Mean 6.65
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 35.7, 95% CI 2-sided [22.42 to 48.99], Standard Error of Mean 6.75
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.0304, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 14.6, 95% CI 2-sided [1.40 to 27.90], Standard Error of Mean 6.74
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0022, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.4, 95% CI 2-sided [7.38 to 33.50], Standard Error of Mean 6.64
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 26.5, 95% CI 2-sided [13.56 to 39.50], Standard Error of Mean 6.59
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.0362, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 14.4, 95% CI 2-sided [0.93 to 27.95], Standard Error of Mean 6.87
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0009, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 22.9, 95% CI 2-sided [9.41 to 36.47], Standard Error of Mean 6.88
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 28.9, 95% CI 2-sided [15.27 to 42.46], Standard Error of Mean 6.91
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 36.8, 95% CI 2-sided [22.99 to 50.57], Standard Error of Mean 7.01
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0265, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 15.6, 95% CI 2-sided [1.83 to 29.34], Standard Error of Mean 6.99
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0023, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 21.2, 95% CI 2-sided [7.60 to 34.71], Standard Error of Mean 6.89
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 27.1, 95% CI 2-sided [13.64 to 40.59], Standard Error of Mean 6.85
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.1580, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 9.6, 95% CI 2-sided [-3.75 to 22.99], Standard Error of Mean 6.80
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0082, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 18.1, 95% CI 2-sided [4.72 to 31.50], Standard Error of Mean 6.80
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.2, 95% CI 2-sided [11.77 to 38.71], Standard Error of Mean 6.85
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 30.6, 95% CI 2-sided [16.93 to 44.31], Standard Error of Mean 6.96
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.1074, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 11.2, 95% CI 2-sided [-2.45 to 24.84], Standard Error of Mean 6.93
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0077, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 18.3, 95% CI 2-sided [4.87 to 31.76], Standard Error of Mean 6.83
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 23.6, 95% CI 2-sided [10.29 to 37.01], Standard Error of Mean 6.79
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.0689, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 11.8, 95% CI 2-sided [-0.92 to 24.53], Standard Error of Mean 6.47
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.0250, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 14.6, 95% CI 2-sided [1.84 to 27.27], Standard Error of Mean 6.46
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 24.4, 95% CI 2-sided [11.54 to 37.17], Standard Error of Mean 6.51
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 29.6, 95% CI 2-sided [16.60 to 42.57], Standard Error of Mean 6.60
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.2041, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 8.4, 95% CI 2-sided [-4.58 to 21.36], Standard Error of Mean 6.59
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0049, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 18.4, 95% CI 2-sided [5.62 to 31.20], Standard Error of Mean 6.50
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0015, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.7, 95% CI 2-sided [8.00 to 33.37], Standard Error of Mean 6.45
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.0184, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 15.8, 95% CI 2-sided [2.68 to 28.89], Standard Error of Mean 6.66
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.0551, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 12.8, 95% CI 2-sided [-0.28 to 25.93], Standard Error of Mean 6.66
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.8, 95% CI 2-sided [12.51 to 39.00], Standard Error of Mean 6.73
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 31.6, 95% CI 2-sided [18.17 to 44.93], Standard Error of Mean 6.80
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Wek 10; Test type: Superiority; p = 0.0367, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 14.3, 95% CI 2-sided [0.89 to 27.62], Standard Error of Mean 6.79
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0017, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 21.2, 95% CI 2-sided [7.99 to 34.34], Standard Error of Mean 6.70
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 24.4, 95% CI 2-sided [11.29 to 37.44], Standard Error of Mean 6.65
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.0255, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 14.5, 95% CI 2-sided [1.78 to 27.15], Standard Error of Mean 6.45
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0186, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 15.3, 95% CI 2-sided [2.57 to 27.94], Standard Error of Mean 6.45
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 26.5, 95% CI 2-sided [13.71 to 39.36], Standard Error of Mean 6.52
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 29.9, 95% CI 2-sided [16.94 to 42.81], Standard Error of Mean 6.58
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0347, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 13.9, 95% CI 2-sided [1.01 to 26.85], Standard Error of Mean 6.57
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 21.9, 95% CI 2-sided [9.16 to 34.65], Standard Error of Mean 6.48
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 23.4, 95% CI 2-sided [10.75 to 36.04], Standard Error of Mean 6.43
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.0221, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 14.8, 95% CI 2-sided [2.13 to 27.43], Standard Error of Mean 6.43
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.0087, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 17.0, 95% CI 2-sided [4.32 to 29.62], Standard Error of Mean 6.43
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 26.4, 95% CI 2-sided [13.65 to 39.23], Standard Error of Mean 6.50
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 31.0, 95% CI 2-sided [18.13 to 43.94], Standard Error of Mean 6.56
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.0244, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 14.8, 95% CI 2-sided [1.92 to 27.70], Standard Error of Mean 6.55
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 21.9, 95% CI 2-sided [9.21 to 34.62], Standard Error of Mean 6.46
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 23.2, 95% CI 2-sided [10.63 to 35.83], Standard Error of Mean 6.41
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.1871, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 9.8, 95% CI 2-sided [-4.77 to 24.30], Standard Error of Mean 7.38
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.7552, MMMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 2.3, 95% CI 2-sided [-12.23 to 16.83], Standard Error of Mean 7.38
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.8407, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 1.5, 95% CI 2-sided [-13.44 to 16.50], Standard Error of Mean 7.61
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.3450, LSMean difference — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 7.2, 95% CI 2-sided [-7.77 to 22.14], Standard Error of Mean 7.60
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.4550, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 5.7, 95% CI 2-sided [-9.34 to 20.80], Standard Error of Mean 7.66
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.1747, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 10.4, 95% CI 2-sided [-4.64 to 25.44], Standard Error of Mean 7.64
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.5476, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 4.4, 95% CI 2-sided [-10.08 to 18.97], Standard Error of Mean 7.38
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.7954, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 2.1, 95% CI 2-sided [-13.69 to 17.84], Standard Error of Mean 8.01
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.8731, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean differencce = 1.3, 95% CI 2-sided [-14.41 to 16.95], Standard Error of Mean 7.96
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.9689, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = -0.3, 95% CI 2-sided [-16.68 to 16.03], Standard Error of Mean 8.31
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.6378, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 3.9, 95% CI 2-sided [-12.40 to 20.21], Standard Error of Mean 8.28
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.8503, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean differencce = 1.6, 95% CI 2-sided [-14.82 to 17.97], Standard Error of Mean 8.33
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.1224, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 13.0, 95% CI 2-sided [-3.51 to 29.44], Standard Error of Mean 8.37
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.3743, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 7.1, 95% CI 2-sided [-8.62 to 22.85], Standard Error of Mean 7.99
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.3173, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = -7.9, 95% CI 2-sided [-23.44 to 7.63], Standard Error of Mean 7.89
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.7905, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = -2.1, 95% CI 2-sided [-17.48 to 13.32], Standard Error of Mean 7.82
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.3804, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = -7.2, 95% CI 2-sided [-23.46 to 8.98], Standard Error of Mean 8.24
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.4905, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = -5.6, 95% CI 2-sided [-21.58 to 10.38], Standard Error of Mean 8.11
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.1289, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = -12.6, 95% CI 2-sided [-28.83 to 3.68], Standard Error of Mean 8.25
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.4398, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 6.4, 95% CI 2-sided [-9.86 to 22.61], Standard Error of Mean 8.24
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.7921, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = -2.1, 95% CI 2-sided [-17.45 to 13.33], Standard Error of Mean 7.81

12. Secondary Outcome: Mean Percent Reduction of Moderate And Severe Vasomotor Symptoms From Baseline to Each Study Week
Description: as for outcome 1
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Percent Reduction
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
Percent Reduction
  Week 1 | 17.5 (5.51) | 36.6 (5.18) | 44.5 (5.39) | 57.0 (5.30) | 62.3 (5.57) | 29.6 (5.59) | 45.3 (5.20) | 47.0 (5.40)
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 33.8 (5.34) | 53.7 (5.01) | 62.4 (5.23) | 67.6 (5.12) | 73.3 (5.42) | 51.4 (5.41) | 57.9 (5.03) | 57.7 (5.25)
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 34.8 (5.61) | 58.1 (5.31) | 69.2 (5.53) | 70.5 (5.40) | 77.8 (5.73) | 60.3 (5.71) | 66.0 (5.32) | 63.7 (5.52)
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 38.6 (5.57) | 61.7 (5.31) | 70.7 (5.50) | 70.0 (5.37) | 80.5 (5.71) | 64.2 (5.68) | 70.0 (5.28) | 68.1 (5.49)
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 43.6 (5.31) | 63.8 (5.06) | 74.2 (5.25) | 72.7 (5.17) | 83.7 (5.49) | 68.0 (5.42) | 70.3 (5.04) | 67.0 (5.28)
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 48.5 (5.02) | 67.7 (4.75) | 72.4 (4.94) | 75.7 (4.87) | 84.1 (5.19) | 68.5 (5.14) | 72.6 (4.76) | 71.7 (4.99)
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 49.1 (5.16) | 66.7 (4.90) | 74.9 (5.09) | 74.9 (5.04) | 85.4 (5.34) | 69.7 (5.28) | 72.0 (4.91) | 71.9 (5.14)
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 54.5 (5.09) | 68.3 (4.81) | 74.5 (5.01) | 76.6 (4.96) | 84.5 (5.28) | 69.4 (5.23) | 74.1 (4.85) | 74.1 (5.08)
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 56.4 (4.91) | 72.4 (4.64) | 74.5 (4.82) | 79.0 (4.78) | 85.7 (5.08) | 70.1 (5.05) | 76.5 (4.68) | 73.8 (4.90)
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 53.5 (5.03) | 74.2 (4.77) | 72.3 (4.95) | 77.9 (4.95) | 85.6 (5.21) | 72.6 (5.18) | 76.6 (4.81) | 76.4 (5.03)
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 55.6 (4.82) | 74.1 (4.55) | 75.8 (4.75) | 80.6 (4.73) | 85.4 (4.99) | 75.1 (4.96) | 79.0 (4.59) | 77.3 (4.82)
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 55.0 (4.85) | 74.3 (4.58) | 75.8 (4.77) | 80.2 (4.77) | 86.9 (5.02) | 75.1 (4.99) | 77.7 (4.61) | 76.9 (4.84)
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 44.9 (6.02) | 61.9 (5.37) | 51.7 (5.55) | 52.5 (5.78) | 55.8 (5.92) | 61.3 (5.98) | 56.6 (5.76) | 48.8 (5.63)
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 41.0 (6.47) | 50.4 (5.83) | 44.9 (5.93) | 45.9 (6.34) | 47.2 (6.44) | 51.4 (6.49) | 55.3 (6.36) | 47.7 (6.06)
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 45.6 (6.49) | 44.7 (5.98) | 45.6 (6.04) | 46.0 (6.61) | 41.7 (6.54) | 45.5 (6.76) | 53.2 (6.57) | 42.9 (6.12)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0090, MMRM — [p-value comment as in outcome 11, analysis 2]; MMRM: Mixed Model Repeated Measures; LSMean difference = 19.1, 95% CI 2-sided [4.82 to 33.46], Standard Error of Mean 7.28
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 27.0, 95% CI 2-sided [12.61 to 41.39], Standard Error of Mean 7.32
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 39.5, 95% CI 2-sided [25.14 to 53.90], Standard Error of Mean 7.31
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 44.8, 95% CI 2-sided [30.27 to 59.39], Standard Error of Mean 7.40
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.1019, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 12.2, 95% CI 2-sided [-2.43 to 26.79], Standard Error of Mean 7.43
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 27.8, 95% CI 2-sided [13.45 to 42.22], Standard Error of Mean 7.31
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 29.5, 95% CI 2-sided [15.21 to 43.82], Standard Error of Mean 7.27
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0049, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.9, 95% CI 2-sided [6.10 to 33.76], Standard Error of Mean 7.03
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 28.6, 95% CI 2-sided [14.64 to 42.46], Standard Error of Mean 7.07
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean differencce = 33.8, 95% CI 2-sided [19.96 to 47.69], Standard Error of Mean 7.05
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 39.5, 95% CI 2-sided [25.40 to 53.58], Standard Error of Mean 7.16
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0146, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 17.6, 95% CI 2-sided [3.50 to 31.70], Standard Error of Mean 7.17
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 24.1, 95% CI 2-sided [10.21 to 38.00], Standard Error of Mean 7.06
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 23.9, 95% CI 2-sided [10.05 to 37.70], Standard Error of Mean 7.03
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0020, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 23.2, 95% CI 2-sided [8.56 to 37.90], Standard Error of Mean 7.46
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 34.4, 95% CI 2-sided [19.60 to 49.11], Standard Error of Mean 7.50
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 35.6, 95% CI 2-sided [20.96 to 50.32], Standard Error of Mean 7.46
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 43.0, 95% CI 2-sided [28.03 to 57.93], Standard Error of Mean 7.60
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0009, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.4, 95% CI 2-sided [10.48 to 40.37], Standard Error of Mean 7.60
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 31.2, 95% CI 2-sided [16.49 to 45.90], Standard Error of Mean 7.48
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 28.9, 95% CI 2-sided [14.24 to 43.52], Standard Error of Mean 7.44
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0021, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 23.1, 95% CI 2-sided [8.46 to 37.66], Standard Error of Mean 7.42
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 32.1, 95% CI 2-sided [17.42 to 46.71], Standard Error of Mean 7.45
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 31.3, 95% CI 2-sided [16.73 to 45.91], Standard Error of Mean 7.42
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 41.8, 95% CI 2-sided [26.95 to 56.68], Standard Error of Mean 7.56
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0008, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.6, 95% CI 2-sided [10.77 to 40.43], Standard Error of Mean 7.54
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 31.3, 95% CI 2-sided [16.75 to 45.94], Standard Error of Mean 7.42
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 29.4, 95% CI 2-sided [14.91 to 43.97], Standard Error of Mean 7.39
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.0045, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.2, 95% CI 2-sided [6.31 to 34.06], Standard Error of Mean 7.05
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 30.6, 95% CI 2-sided [16.68 to 44.49], Standard Error of Mean 7.07
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 29.1, 95% CI 2-sided [15.14 to 42.98], Standard Error of Mean 7.08
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 40.1, 95% CI 2-sided [25.96 to 54.26], Standard Error of Mean 7.19
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0007, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 24.4, 95% CI 2-sided [10.28 to 38.42], Standard Error of Mean 7.15
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 26.7, 95% CI 2-sided [1.78 to 40.55], Standard Error of Mean 7.06
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0010, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 23.4, 95% CI 2-sided [9.55 to 37.22], Standard Error of Mean 7.03
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.0040, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.1, 95% CI 2-sided [6.13 to 32.11], Standard Error of Mean 6.60
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 23.8, 95% CI 2-sided [10.80 to 36.83], Standard Error of Mean 6.62
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 27.2, 95% CI 2-sided [14.10 to 40.24], Standard Error of Mean 6.64
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 35.6, 95% CI 2-sided [22.34 to 48.88], Standard Error of Mean 6.75
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.0032, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.0, 95% CI 2-sided [6.76 to 33.19], Standard Error of Mean 6.72
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 24.1, 95% CI 2-sided [11.02 to 37.13], Standard Error of Mean 6.64
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0005, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 23.1, 95% CI 2-sided [10.17 to 36.08], Standard Error of Mean 6.59
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.0102, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 17.6, 95% CI 2-sided [4.20 to 31.04], Standard Error of Mean 6.82
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.9, 95% CI 2-sided [12.42 to 39.29], Standard Error of Mean 6.83
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.8, 95% CI 2-sided [12.29 to 39.33], Standard Error of Mean 6.87
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 36.3, 95% CI 2-sided [22.58 to 49.98], Standard Error of Mean 6.97
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0031, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.6, 95% CI 2-sided [7.00 to 34.29], Standard Error of Mean 6.94
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0009, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 22.9, 95% CI 2-sided [9.43 to 36.38], Standard Error of Mean 6.85
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0009, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 22.8, 95% CI 2-sided [9.42 to 36.19], Standard Error of Mean 6.80
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.0408, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 13.8, 95% CI 2-sided [0.58 to 26.97], Standard Error of Mean 6.71
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0031, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.0, 95% CI 2-sided [6.77 to 33.21], Standard Error of Mean 6.72
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0012, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 22.1, 95% CI 2-sided [8.80 to 35.40], Standard Error of Mean 6.76
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 29.9, 95% CI 2-sided [16.39 to 43.42], Standard Error of Mean 6.87
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.0303, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 14.9, 95% CI 2-sided [1.42 to 28.32], Standard Error of Mean 6.84
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0040, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.6, 95% CI 2-sided [6.30 to 32.87], Standard Error of Mean 6.75
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0038, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.5, 95% CI 2-sided [6.34 to 32.73], Standard Error of Mean 6.71
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.0137, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 16.0, 95% CI 2-sided [3.29 to 28.68], Standard Error of Mean 6.45
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.0052, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 18.1, 95% CI 2-sided [5.44 to 30.82], Standard Error of Mean 6.45
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 22.6, 95% CI 2-sided [9.81 to 35.39], Standard Error of Mean 6.50
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 29.4, 95% CI 2-sided [16.41 to 42.32], Standard Error of Mean 6.58
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.0378, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 13.7, 95% CI 2-sided [0.78 to 26.63], Standard Error of Mean 6.57
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.1, 95% CI 2-sided [7.31 to 32.85], Standard Error of Mean 6.49
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0071, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 17.4, 95% CI 2-sided [4.77 to 30.09], Standard Error of Mean 6.44
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.0020, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.7, 95% CI 2-sided [7.61 to 33.71], Standard Error of Mean 6.63
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.0050, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 18.7, 95% CI 2-sided [5.68 to 31.79], Standard Error of Mean 6.63
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 24.4, 95% CI 2-sided [11.20 to 37.60], Standard Error of Mean 6.71
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 32.1, 95% CI 2-sided [18.77 to 45.42], Standard Error of Mean 6.77
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Wek 10; Test type: Superiority; p = 0.0050, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.1, 95% CI 2-sided [5.79 to 32.38], Standard Error of Mean 6.76
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 23.1, 95% CI 2-sided [9.95 to 36.22], Standard Error of Mean 6.68
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 22.8, 95% CI 2-sided [9.79 to 35.85], Standard Error of Mean 6.62
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.0036, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 18.5, 95% CI 2-sided [6.11 to 30.98], Standard Error of Mean 6.32
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0015, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.2, 95% CI 2-sided [7.77 to 32.65], Standard Error of Mean 6.32
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.0, 95% CI 2-sided [12.41 to 37.57], Standard Error of Mean 6.39
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 29.8, 95% CI 2-sided [17.12 to 42.49], Standard Error of Mean 6.45
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0026, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.6, 95% CI 2-sided [6.90 to 32.21], Standard Error of Mean 6.43
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 23.4, 95% CI 2-sided [10.92 to 35.94], Standard Error of Mean 6.36
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 21.7, 95% CI 2-sided [9.34 to 34.14], Standard Error of Mean 6.30
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.0026, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 19.3, 95% CI 2-sided [6.78 to 31.83], Standard Error of Mean 6.37
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.0012, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.8, 95% CI 2-sided [8.29 to 33.33], Standard Error of Mean 6.36
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 25.1, 95% CI 2-sided [12.48 to 37.82], Standard Error of Mean 6.44
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 11, analysis 1]; LSMean difference = 31.9, 95% CI 2-sided [19.11 to 44.67], Standard Error of Mean 6.50
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.0021, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 20.1, 95% CI 2-sided [7.32 to 32.81], Standard Error of Mean 6.48
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 22.7, 95% CI 2-sided [10.10 to 35.29], Standard Error of Mean 6.40
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0006, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 21.9, 95% CI 2-sided [9.42 to 34.38], Standard Error of Mean 6.34
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.0304, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 17.0, 95% CI 2-sided [1.62 to 32.40], Standard Error of Mean 7.82
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.3857, MMMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 6.8, 95% CI 2-sided [-8.60 to 22.19], Standard Error of Mean 7.82
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.3497, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 7.5, 95% CI 2-sided [-8.31 to 23.40], Standard Error of Mean 8.06
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.1771, LSMean difference — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 10.9, 95% CI 2-sided [-4.95 to 26.75], Standard Error of Mean 8.05
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.0444, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 16.3, 95% CI 2-sided [0.41 to 32.29], Standard Error of Mean 8.10
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.1500, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 11.7, 95% CI 2-sided [-4.25 to 27.63], Standard Error of Mean 8.10
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.6196, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 3.9, 95% CI 2-sided [-11.51 to 19.29], Standard Error of Mean 7.83
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.2664, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 9.4, 95% CI 2-sided [-7.25 to 26.15], Standard Error of Mean 8.48
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.6388, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean differencce = 4.0, 95% CI 2-sided [-12.66 to 20.59], Standard Error of Mean 8.44
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.5797, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 4.9, 95% CI 2-sided [-12.43 to 22.19], Standard Error of Mean 8.79
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.4817, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 6.2, 95% CI 2-sided [-11.10 to 23.47], Standard Error of Mean 8.78
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.2358, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean differencce = 10.5, 95% CI 2-sided [-6.87 to 27.79], Standard Error of Mean 8.80
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.1070, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 14.3, 95% CI 2-sided [-3.11 to 31.77], Standard Error of Mean 8.86
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.4268, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 6.7, 95% CI 2-sided [-9.94 to 23.43], Standard Error of Mean 8.47
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.9197, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = -0.9, 95% CI 2-sided [-17.81 to 16.08], Standard Error of Mean 8.61
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.9954, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 0.0, 95% CI 2-sided [-16.77 to 16.87], Standard Error of Mean 8.54
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.9607, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 0.4, 95% CI 2-sided [-17.28 to 18.17], Standard Error of Mean 9.00
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.6625, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = -3.9, 95% CI 2-sided [-21.33 to 13.59], Standard Error of Mean 8.87
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.9952, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = -0.1, 95% CI 2-sided [-17.81 to 17.70], Standard Error of Mean 9.01
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.4001, MMRM — [p-value comment as in outcome 11, analysis 2]; LSMean difference = 7.6, 95% CI 2-sided [-10.16 to 25.36], Standard Error of Mean 9.02
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.7510, MMRM — [p-value comment as in outcome 11, analysis 1]; LSMean difference = -2.7, 95% CI 2-sided [-19.52 to 14.10], Standard Error of Mean 8.54

13. Secondary Outcome: Number of Participants With Mean Percent Reduction of 50% in The Mean Frequency of Mild, Moderate, and Severe VMS From Baseline to Each Study Week
Description: The frequency of mild, moderate and severe VMS was the number of mild, moderate and severe VMS per 24 hours. A daily frequency and severity per week was derived by taking the mean of the data over 7 days. Mild VMS was defined as sensation of heat without sweating/dampness. If at night, participant does not wake up but later notices damp sheets or clothing. Moderate VMS was defined as sensation of heat with sweating/dampness, but was able to continue activity. If at night, participant woke up because she was feeling hot and/or was sweating, but no action was necessary other than rearranging the bed sheets. Severe VMS was defined as sensation of intense heat with sweating, caused disruption of activity. If at night, participant woke up hot and was sweating and needed to take action (e.g., remove layers of clothes, open the window, or get out of bed).
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 5 | 19 | 22 | 24 | 25 | 10 | 21 | 23
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 14 | 26 | 29 | 32 | 30 | 22 | 26 | 28
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 16 | 26 | 29 | 33 | 32 | 26 | 29 | 29
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 19 | 26 | 29 | 31 | 31 | 25 | 32 | 31
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 22 | 24 | 31 | 30 | 29 | 28 | 30 | 29
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 24 | 24 | 30 | 31 | 28 | 24 | 30 | 33
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 25 | 25 | 32 | 29 | 28 | 28 | 30 | 30
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 26 | 28 | 32 | 32 | 28 | 25 | 31 | 32
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 27 | 29 | 33 | 31 | 31 | 25 | 30 | 31
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 23 | 28 | 26 | 26 | 31 | 26 | 32 | 32
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 23 | 28 | 30 | 25 | 30 | 27 | 33 | 31
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 21 | 27 | 27 | 27 | 28 | 24 | 32 | 32
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 12 | 19 | 17 | 14 | 15 | 16 | 14 | 17
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 11 | 14 | 15 | 10 | 13 | 15 | 14 | 17
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 30 | 21 | 29
  Week 15 | 14 | 10 | 12 | 6 | 9 | 9 | 12 | 13
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0018, Regression, Logistic — Odds ratio, corresponding 95% CI and p-value are based on a logistic regression with responder as the dependent variable and treatment group and smoking status as factors and baseline measurement (mean frequency of vasomotor symptoms) as a covariate; Odds Ratio (OR) = 6.02, 95% CI 2-sided [1.95 to 18.64]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.28, 95% CI 2-sided [2.70 to 25.42]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.92, 95% CI 2-sided [3.53 to 33.74]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 12.18, 95% CI 2-sided [3.91 to 37.89]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.2244, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.10, 95% CI 2-sided [0.64 to 6.92]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.58, 95% CI 2-sided [2.77 to 26.53]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.25, 95% CI 2-sided [2.71 to 25.13]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0149, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.04, 95% CI 2-sided [1.24 to 7.45]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0011, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.65, 95% CI 2-sided [1.85 to 11.73]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.36, 95% CI 2-sided [2.46 to 16.45]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.87, 95% CI 2-sided [2.56 to 18.46]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0897, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.18, 95% CI 2-sided [0.89 to 5.34]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0070, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.46, 95% CI 2-sided [1.42 to 8.53]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0041, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.75, 95% CI 2-sided [1.52 to 9.23]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0254, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.13 to 6.78]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0032, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.00, 95% CI 2-sided [1.59 to 10.04]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.25, 95% CI 2-sided [2.37 to 16.51]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.78, 95% CI 2-sided [3.00 to 25.70]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0214, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.90, 95% CI 2-sided [1.17 to 7.18]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0049, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.67, 95% CI 2-sided [1.48 to 9.09]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0078, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.36, 95% CI 2-sided [1.38 to 8.22]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0727, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.28, 95% CI 2-sided [0.93 to 5.63]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0199, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.94, 95% CI 2-sided [1.19 to 7.29]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0034, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.21, 95% CI 2-sided [1.61 to 11.01]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0007, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.26, 95% CI 2-sided [2.16 to 18.26]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.1206, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.83 to 4.92]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0070, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.58, 95% CI 2-sided [1.42 to 9.03]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0088, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.41, 95% CI 2-sided [1.36 to 8.54]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.4485, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.58 to 3.40]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0255, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.92, 95% CI 2-sided [1.14 to 7.47]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0066, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.18, 95% CI 2-sided [1.49 to 11.75]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p = 0.0061, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.46, 95% CI 2-sided [1.53 to 13.01]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0879, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.89 to 5.57]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0389, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.68, 95% CI 2-sided [1.05 to 6.83]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0446, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.02 to 6.73]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.8196, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.45 to 2.72]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.1450, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.79 to 5.10]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0114, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.08, 95% CI 2-sided [1.37 to 12.11]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0307, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.29, 95% CI 2-sided [1.12 to 9.71]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.5921, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.51 to 3.24]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0502, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.69, 95% CI 2-sided [1.00 to 7.26]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0224, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.31, 95% CI 2-sided [1.18 to 9.25]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.7225, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.47 to 2.93]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0762, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.43, 95% CI 2-sided [0.91 to 6.48]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0252, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.51, 95% CI 2-sided [1.17 to 10.53]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0490, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.98, 95% CI 2-sided [1.00 to 8.87]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.1773, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.74 to 5.30]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0609, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.62, 95% CI 2-sided [0.96 to 7.16]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.1364, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.11, 95% CI 2-sided [0.79 to 5.61]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.5268, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.53 to 3.51]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.1645, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.75 to 5.46]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0215, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.92, 95% CI 2-sided [1.22 to 12.57]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0600, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.04, 95% CI 2-sided [0.95 to 9.69]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.6503, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.47 to 3.32]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0683, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.70, 95% CI 2-sided [0.93 to 7.88]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0618, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.83, 95% CI 2-sided [0.95 to 8.44]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.5621, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.50 to 3.63]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.2182, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.92, 95% CI 2-sided [0.68 to 5.40]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0600, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.11, 95% CI 2-sided [0.95 to 10.15]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0290, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.60, 95% CI 2-sided [1.17 to 18.12]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.8485, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.40 to 3.04]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.1652, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.16, 95% CI 2-sided [0.73 to 6.42]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.2244, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.94, 95% CI 2-sided [0.67 to 5.65]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.2097, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.71 to 4.84]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.3708, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.60 to 3.92]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0704, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.66, 95% CI 2-sided [0.92 to 7.66]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0040, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.21, 95% CI 2-sided [1.88 to 27.73]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.1625, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.04, 95% CI 2-sided [0.75 to 5.55]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0093, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.59, 95% CI 2-sided [1.46 to 14.50]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0103, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.44, 95% CI 2-sided [1.42 to 13.87]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.1965, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.89, 95% CI 2-sided [0.72 to 4.95]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0549, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.69, 95% CI 2-sided [0.98 to 7.42]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.0503, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.01, 95% CI 2-sided [1.00 to 9.09]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0046, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.03, 95% CI 2-sided [1.82 to 27.10]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0866, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.46, 95% CI 2-sided [0.88 to 6.88]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0045, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.96, 95% CI 2-sided [1.74 to 20.40]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0207, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.59, 95% CI 2-sided [1.22 to 10.62]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.2127, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.86, 95% CI 2-sided [0.70 to 4.91]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.1521, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.04, 95% CI 2-sided [0.77 to 5.43]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0098, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.12, 95% CI 2-sided [1.48 to 17.70]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0047, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.08, 95% CI 2-sided [1.82 to 27.50]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.1817, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.72 to 5.51]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0042, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.09, 95% CI 2-sided [1.77 to 20.95]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0039, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.09, 95% CI 2-sided [1.78 to 20.74]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.7025, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.42 to 3.57]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.9599, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.36 to 2.97]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.9671, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.34 to 3.10]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.6810, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.42 to 3.83]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.6346, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.43 to 4.04]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.7929, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.38 to 3.57]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.8188, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.39 to 3.28]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.8226, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.30 to 2.60]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.9088, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.32 to 2.72]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.6189, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.24 to 2.35]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.6463, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.42 to 4.03]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.5060, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.47 to 4.54]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.3842, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.53 to 5.31]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.5021, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.49 to 4.23]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.1349, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.14 to 1.31]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.3191, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.19 to 1.71]
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.0623, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.09 to 1.06]
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.1958, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.15 to 1.48]
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.4353, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.19 to 2.05]
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.9729, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.31 to 3.31]
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.4211, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.22 to 1.89]

14. Secondary Outcome: Number of Participants With Mean Percent Reduction of 70% in The Mean Frequency of Mild, Moderate, and Severe VMS From Baseline to Each Study Week
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 2 | 6 | 11 | 17 | 18 | 6 | 7 | 16
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 9 | 15 | 19 | 26 | 24 | 13 | 13 | 21
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 11 | 17 | 20 | 27 | 27 | 17 | 16 | 26
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 10 | 14 | 22 | 24 | 30 | 19 | 24 | 26
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 15 | 17 | 21 | 26 | 29 | 22 | 22 | 25
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 14 | 18 | 21 | 27 | 28 | 19 | 22 | 26
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 15 | 19 | 24 | 25 | 28 | 20 | 22 | 25
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 18 | 19 | 25 | 24 | 27 | 19 | 21 | 26
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 18 | 21 | 22 | 27 | 28 | 19 | 24 | 26
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 16 | 21 | 20 | 23 | 29 | 21 | 26 | 24
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 19 | 25 | 23 | 24 | 28 | 20 | 28 | 28
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 18 | 21 | 22 | 25 | 26 | 22 | 26 | 27
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 4 | 12 | 7 | 9 | 7 | 10 | 5 | 11
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 8 | 6 | 5 | 3 | 2 | 7 | 7 | 10
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 8 | 4 | 5 | 3 | 0 | 2 | 5 | 7
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.1938, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.05, 95% CI 2-sided [0.57 to 16.35]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0162, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.97, 95% CI 2-sided [1.43 to 33.91]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p = 0.0008, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 14.37, 95% CI 2-sided [3.04 to 67.96]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p = 0.0005, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 16.02, 95% CI 2-sided [3.39 to 75.68]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.1971, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.02, 95% CI 2-sided [0.56 to 16.17]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0811, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.31, 95% CI 2-sided [0.83 to 22.27]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0021, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.44, 95% CI 2-sided [2.43 to 53.94]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.1370, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.11, 95% CI 2-sided [0.79 to 5.64]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0181, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.20, 95% CI 2-sided [1.22 to 8.40]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.43, 95% CI 2-sided [2.43 to 17.05]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.08, 95% CI 2-sided [2.26 to 16.31]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.3241, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.61 to 4.49]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.2249, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.68 to 5.03]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0096, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.53, 95% CI 2-sided [1.36 to 9.18]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0768, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.35, 95% CI 2-sided [0.91 to 6.05]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.00251, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.91, 95% CI 2-sided [1.14 to 7.39]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.99, 95% CI 2-sided [2.30 to 15.57]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.29, 95% CI 2-sided [2.70 to 19.71]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.1144, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.14, 95% CI 2-sided [0.83 to 5.50]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.1341, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.80 to 5.30]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0017, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.43, 95% CI 2-sided [1.75 to 11.22]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.1488, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.77 to 5.50]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0043, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.99, 95% CI 2-sided [1.54 to 10.30]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0005, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.53, 95% CI 2-sided [2.10 to 14.57]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 14.54, 95% CI 2-sided [4.85 to 43.58]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0262, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.96, 95% CI 2-sided [1.14 to 7.68]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0009, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.07, 95% CI 2-sided [1.95 to 13.19]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0006, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.33, 95% CI 2-sided [2.06 to 13.80]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.3673, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.61 to 3.75]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.1207, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.83 to 4.91]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0011, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.01, 95% CI 2-sided [1.90 to 13.21]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.19, 95% CI 2-sided [3.08 to 27.38]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0594, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.38, 95% CI 2-sided [0.97 to 5.86]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0500, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.47, 95% CI 2-sided [1.00 to 6.09]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0123, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.22, 95% CI 2-sided [1.29 to 8.03]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.2243, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.71 to 4.37]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0976, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.87 to 5.24]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0004, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.09, 95% CI 2-sided [2.25 to 16.44]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.13, 95% CI 2-sided [3.04 to 27.40]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.1237, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.82 to 5.17]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0226, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.94, 95% CI 2-sided [1.16 to 7.41]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0069, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.55, 95% CI 2-sided [1.42 to 8.91]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.1666, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.76 to 4.75]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0317, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.70, 95% CI 2-sided [1.09 to 6.67]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0011, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.28, 95% CI 2-sided [1.94 to 14.39]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.45, 95% CI 2-sided [2.81 to 25.46]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.1142, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.10, 95% CI 2-sided [0.84 to 5.27]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0250, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.91, 95% CI 2-sided [1.14 to 7.39]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0166, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.08, 95% CI 2-sided [1.23 to 7.75]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.6033, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.52 to 3.11]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.1170, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.05, 95% CI 2-sided [0.84 to 5.02]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0400, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.69, 95% CI 2-sided [1.05 to 6.91]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0020, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.61, 95% CI 2-sided [1.88 to 16.72]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.5177, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.54 to 3.37]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.2117, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.72 to 4.48]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0426, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.03 to 6.67]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.3508, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.62 to 3.82]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.4431, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.58 to 3.45]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0050, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.27, 95% CI 2-sided [1.55 to 11.78]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0023, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.47, 95% CI 2-sided [1.84 to 16.30]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.5663, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.52 to 3.32]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0461, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.02 to 6.83]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0552, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.50, 95% CI 2-sided [0.98 to 6.38]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.1536, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.78 to 4.88]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.2575, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.69, 95% CI 2-sided [0.68 to 4.20]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0096, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.73, 95% CI 2-sided [1.38 to 10.11]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.48, 95% CI 2-sided [2.69 to 26.76]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.1047, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.18, 95% CI 2-sided [1.48 to 10.35]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0060, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.91, 95% CI 2-sided [1.48 to 10.35]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0414, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.04 to 6.71]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.0809, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.31, 95% CI 2-sided [0.90 to 5.89]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.2377, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.69 to 4.34]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.0087, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.21, 95% CI 2-sided [1.44 to 12.34]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0022, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.00, 95% CI 2-sided [1.90 to 18.94]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.4788, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.55 to 3.55]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0074, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.98, 95% CI 2-sided [1.45 to 10.94]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0187, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.26, 95% CI 2-sided [1.22 to 8.75]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.3443, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.62 to 4.00]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.2867, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.65 to 4.22]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0044, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.12, 95% CI 2-sided [1.66 to 15.78]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0038, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.58, 95% CI 2-sided [1.74 to 17.87]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.1424, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.09, 95% CI 2-sided [0.78 to 5.60]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0191, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.32, 95% CI 2-sided [1.22 to 9.07]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0244, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.15, 95% CI 2-sided [1.16 to 8.56]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.1462, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.63, 95% CI 2-sided [0.71 to 9.67]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.7403, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.32 to 4.97]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.2144, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.35, 95% CI 2-sided [0.61 to 9.07]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.4321, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.44 to 6.96]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.1778, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.53, 95% CI 2-sided [0.66 to 9.75]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.8016, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.28 to 5.20]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.1486, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.62, 95% CI 2-sided [0.71 to 9.64]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.2881, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.15 to 1.77]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.1217, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.10 to 1.31]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.1027, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.07 to 1.28]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.0428, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.18, 95% CI 2-sided [0.03 to 0.94]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.5943, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.21 to 2.44]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.9280, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.27 to 3.28]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.9160, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.30 to 2.94]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.2262, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.11 to 1.69]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.2682, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.13 to 1.75]
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.2344, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.09 to 1.81]
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.0835, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.22, 95% CI 2-sided [0.04 to 1.22]
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.6322, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.19 to 2.72]
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.4845, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.20 to 2.17]

15. Secondary Outcome: Number of Participants With Mean Percent Reduction of 90% in The Mean Frequency of Mild, Moderate, and Severe VMS From Baseline to Each Study Week
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 1 | 1 | 1 | 6 | 6 | 0 | 3 | 2
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 2 | 5 | 6 | 15 | 16 | 2 | 5 | 12
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 4 | 9 | 9 | 19 | 16 | 6 | 9 | 17
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 6 | 10 | 12 | 19 | 17 | 7 | 12 | 18
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 6 | 7 | 11 | 18 | 20 | 9 | 10 | 18
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 9 | 9 | 16 | 21 | 23 | 9 | 9 | 21
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 6 | 8 | 15 | 20 | 24 | 10 | 12 | 20
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 13 | 11 | 17 | 22 | 23 | 10 | 14 | 22
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 13 | 11 | 15 | 21 | 25 | 10 | 14 | 20
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 13 | 12 | 14 | 20 | 26 | 11 | 15 | 20
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 14 | 13 | 13 | 19 | 25 | 12 | 18 | 20
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 13 | 15 | 15 | 17 | 22 | 10 | 16 | 20
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 1 | 0 | 1 | 2 | 1 | 3 | 1 | 2
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.9587, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.06 to 17.98]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.9895, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.06 to 16.89]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p = 0.0736, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.24, 95% CI 2-sided [0.83 to 63.32]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p = 0.0767, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.08, 95% CI 2-sided [0.81 to 61.78]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.2880, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.51, 95% CI 2-sided [0.35 to 35.49]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.5894, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.96, 95% CI 2-sided [0.17 to 22.47]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.3093, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.45, 95% CI 2-sided [0.44 to 13.78]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.1606, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.31, 95% CI 2-sided [0.62 to 17.58]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0019, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.92, 95% CI 2-sided [2.50 to 56.87]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0008, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 14.40, 95% CI 2-sided [3.02 to 68.73]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.8803, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.11 to 6.55]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.2096, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.98, 95% CI 2-sided [0.54 to 16.46]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0110, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.69, 95% CI 2-sided [1.60 to 37.11]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0845, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.09, 95% CI 2-sided [0.86 to 11.11]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.1094, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.83, 95% CI 2-sided [0.79 to 10.13]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0004, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.97, 95% CI 2-sided [2.68 to 30.07]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0016, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.11, 95% CI 2-sided [2.10 to 24.09]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.4375, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.44 to 6.64]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0898, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.02, 95% CI 2-sided [0.84 to 10.85]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0027, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.32, 95% CI 2-sided [1.90 to 21.06]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.1242, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.44, 95% CI 2-sided [0.78 to 7.64]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0815, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.66, 95% CI 2-sided [0.88 to 8.03]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0009, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.21, 95% CI 2-sided [2.11 to 18.27]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0027, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.28, 95% CI 2-sided [1.78 to 15.64]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.6267, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.41 to 4.46]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0709, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.77, 95% CI 2-sided [0.92 to 8.38]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0049, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.62, 95% CI 2-sided [1.59 to 13.59]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.5107, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.45 to 4.98]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.1297, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.78 to 7.22]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0005, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.04, 95% CI 2-sided [2.34 to 21.22]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.50, 95% CI 2-sided [2.82 to 25.63]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.2990, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.58 to 5.81]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.1355, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.38, 95% CI 2-sided [0.76 to 7.42]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0028, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.17, 95% CI 2-sided [1.76 to 15.14]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.7422, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.41 to 3.47]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0750, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.44, 95% CI 2-sided [0.91 to 6.52]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0006, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.00, 95% CI 2-sided [2.16 to 16.67]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.63, 95% CI 2-sided [2.69 to 21.65]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.8405, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.38 to 3.23]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.6257, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.45 to 3.79]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0060, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.92, 95% CI 2-sided [1.48 to 10.36]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.3556, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.54 to 5.68]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0190, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.67, 95% CI 2-sided [1.24 to 10.90]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.90, 95% CI 2-sided [3.20 to 30.68]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 14.81, 95% CI 2-sided [4.67 to 47.05]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.1936, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.68 to 6.67]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0335, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.39, 95% CI 2-sided [1.10 to 10.47]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0009, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.18, 95% CI 2-sided [2.10 to 18.17]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.8330, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.34 to 2.39]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.3410, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.62 to 3.91]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0075, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.71, 95% CI 2-sided [1.42 to 9.69]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0020, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.86, 95% CI 2-sided [1.78 to 13.26]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.6216, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.29 to 2.10]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.4615, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.55 to 3.71]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0281, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.84, 95% CI 2-sided [1.12 to 7.19]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.8028, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.33 to 2.35]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.6846, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.48 to 3.07]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0149, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.31, 95% CI 2-sided [1.26 to 8.67]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0009, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.64, 95% CI 2-sided [2.03 to 15.65]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.6434, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.29 to 2.15]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.4784, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.54 to 3.69]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0955, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.87 to 5.55]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.9082, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.40 to 2.79]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.6478, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.48 to 3.21]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0104, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.65, 95% CI 2-sided [1.35 to 9.82]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0004, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.66, 95% CI 2-sided [2.34 to 18.94]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.8560, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.34 to 2.45]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.3319, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.62 to 4.17]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0747, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.92 to 5.95]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.8986, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.41 to 2.76]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.9712, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.38 to 2.53]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.0910, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.31, 95% CI 2-sided [1.22 to 8.98]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0011, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.68, 95% CI 2-sided [2.01 to 16.06]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.8466, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.35 to 2.39]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.1409, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.79 to 5.21]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.1212, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.82 to 5.25]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.4269, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.56 to 3.88]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.5454, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.52 to 3.49]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0595, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.62, 95% CI 2-sided [0.96 to 7.15]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0041, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.58, 95% CI 2-sided [1.62 to 12.98]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.6121, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.28 to 2.13]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.2329, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.68 to 4.75]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0891, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.28, 95% CI 2-sided [0.88 to 5.90]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.6857, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.03 to 9.97]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.7291, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.12 to 19.71]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.8951, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.05 to 14.41]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.6865, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.14 to 19.74]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.9132, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.07 to 20.24]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.7982, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.12 to 16.59]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.9029, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.09 to 15.57]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.7971, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.04 to 11.94]

16. Secondary Outcome: Number of Participants With Mean Percent Reduction of 100% in The Mean Frequency of Mild, Moderate, and Severe VMS From Baseline to Each Study Week
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 1 | 2 | 0 | 5 | 7 | 0 | 3 | 4
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 1 | 3 | 3 | 9 | 8 | 2 | 4 | 9
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 1 | 2 | 4 | 6 | 11 | 3 | 6 | 8
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 3 | 2 | 3 | 10 | 10 | 3 | 6 | 6
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 1 | 6 | 3 | 11 | 13 | 3 | 5 | 12
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 1 | 5 | 5 | 13 | 11 | 6 | 6 | 14
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 2 | 7 | 7 | 15 | 12 | 5 | 6 | 14
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 3 | 7 | 11 | 12 | 15 | 3 | 7 | 12
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 4 | 7 | 6 | 9 | 16 | 3 | 8 | 15
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 3 | 7 | 7 | 13 | 17 | 7 | 8 | 13
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 8 | 7 | 10 | 11 | 14 | 5 | 12 | 10
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.7899, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.04 to 12.34]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p = 0.9186, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.05 to 14.73]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.5303, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.19, 95% CI 2-sided [0.19 to 25.46]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.1149, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.85, 95% CI 2-sided [0.65 to 52.66]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0442, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.07, 95% CI 2-sided [1.06 to 77.71]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.2851, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.53, 95% CI 2-sided [0.35 to 35.68]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.2073, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.22, 95% CI 2-sided [0.45 to 39.48]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.2700, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.68, 95% CI 2-sided [0.36 to 37.16]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.2982, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.41, 95% CI 2-sided [0.34 to 34.27]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0204, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 12.30, 95% CI 2-sided [1.47 to 102.6]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0270, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.10, 95% CI 2-sided [1.31 to 93.74]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.5224, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.19 to 25.68]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.1635, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.92, 95% CI 2-sided [0.52 to 46.35]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0266, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.97, 95% CI 2-sided [1.32 to 91.15]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.4299, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.69, 95% CI 2-sided [0.23 to 31.21]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.1667, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.87, 95% CI 2-sided [0.52 to 45.84]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0592, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.11, 95% CI 2-sided [0.92 to 71.35]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0070, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 18.28, 95% CI 2-sided [2.21 to 151.2]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.2594, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.79, 95% CI 2-sided [0.37 to 38.32]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0589, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.14, 95% CI 2-sided [0.92 to 71.67]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0338, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.08, 95% CI 2-sided [1.19 to 85.20]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.7756, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.12 to 4.88]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.9246, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.20 to 5.74]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0177, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.42, 95% CI 2-sided [1.34 to 21.93]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p = 0.0178, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.38, 95% CI 2-sided [1.34 to 21.65]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.8564, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.22 to 6.20]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.2202, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.52, 95% CI 2-sided [0.58 to 11.00]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.2498, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.55 to 10.25]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.0576, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.22, 95% CI 2-sided [0.93 to 72.29]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.3065, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.34, 95% CI 2-sided [0.33 to 33.59]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0056, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 19.90, 95% CI 2-sided [2.40 to 165.1]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0027, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 25.05, 95% CI 2-sided [3.05 to 205.5]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.2762, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.61, 95% CI 2-sided [0.36 to 36.51]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0851, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.93, 95% CI 2-sided [0.77 to 62.69]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0081, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 17.02, 95% CI 2-sided [2.09 to 138.7]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.0995, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.37, 95% CI 2-sided [0.70 to 57.62]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.1184, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.76, 95% CI 2-sided [0.64 to 51.80]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0023, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 26.54, 95% CI 2-sided [3.23 to 218.3]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0062, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 19.09, 95% CI 2-sided [2.31 to 157.9]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0695, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.49, 95% CI 2-sided [0.85 to 65.87]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0520, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.64, 95% CI 2-sided [0.98 to 75.98]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0036, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 22.30, 95% CI 2-sided [2.75 to 180.6]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.0676, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.66, 95% CI 2-sided [0.89 to 24.23]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0903, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.14, 95% CI 2-sided [0.80 to 21.38]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0007, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 15.46, 95% CI 2-sided [3.18 to 75.14]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0032, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.94, 95% CI 2-sided [2.22 to 53.77]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.2031, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.04, 95% CI 2-sided [0.55 to 16.85]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0972, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.13, 95% CI 2-sided [0.77 to 22.10]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0027, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.04, 95% CI 2-sided [2.30 to 53.06]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.1306, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.06, 95% CI 2-sided [0.72 to 13.02]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.0248, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.83, 95% CI 2-sided [1.22 to 19.10]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0054, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.14, 95% CI 2-sided [1.79 to 28.53]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0010, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.01, 95% CI 2-sided [2.55 to 39.36]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.8271, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.23 to 6.45]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.1089, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.27, 95% CI 2-sided [0.77 to 13.95]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0138, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.58, 95% CI 2-sided [1.42 to 21.93]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.1987, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.40, 95% CI 2-sided [0.63 to 9.15]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.3984, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.46 to 7.02]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0402, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.92, 95% CI 2-sided [1.06 to 14.45]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0010, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.05, 95% CI 2-sided [2.32 to 27.95]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.8287, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.17 to 4.08]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.1083, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.93, 95% CI 2-sided [0.79 to 10.92]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0043, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.03, 95% CI 2-sided [1.76 to 20.66]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.1126, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.23, 95% CI 2-sided [0.76 to 13.79]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.1479, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.90, 95% CI 2-sided [0.69 to 12.30]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.0010, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.49, 95% CI 2-sided [2.59 to 42.46]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 13.01, 95% CI 2-sided [3.31 to 51.14]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.1483, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.91, 95% CI 2-sided [0.68 to 12.41]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0557, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.03, 95% CI 2-sided [0.97 to 16.84]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0072, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.47, 95% CI 2-sided [1.66 to 25.28]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.9715, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.32 to 3.24]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.4720, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.50 to 4.39]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.1262, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.35, 95% CI 2-sided [0.79 to 7.05]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0396, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.07, 95% CI 2-sided [1.05 to 8.92]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.5137, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.19 to 2.29]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.1370, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.77 to 6.58]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.5526, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.47 to 4.07]

17. Secondary Outcome: Number of Participants With Mean Percent Reduction of 50% in The Mean Frequency of Moderate and Severe Vasomotor Symptoms From Baseline to Each Study Week
Description: as for outcome 1
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 6 | 21 | 25 | 27 | 28 | 14 | 23 | 25
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 15 | 31 | 31 | 32 | 32 | 25 | 29 | 27
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 18 | 31 | 31 | 33 | 33 | 30 | 33 | 29
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 23 | 29 | 31 | 32 | 32 | 29 | 32 | 31
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 23 | 30 | 34 | 29 | 31 | 32 | 35 | 30
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 25 | 29 | 31 | 31 | 30 | 28 | 34 | 32
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 26 | 29 | 33 | 30 | 30 | 31 | 32 | 29
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 28 | 31 | 33 | 32 | 28 | 30 | 33 | 32
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 27 | 30 | 33 | 32 | 31 | 28 | 32 | 29
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 25 | 31 | 29 | 26 | 31 | 29 | 35 | 31
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 25 | 31 | 31 | 25 | 30 | 31 | 34 | 31
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 22 | 31 | 29 | 27 | 29 | 26 | 32 | 31
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 12 | 22 | 18 | 14 | 18 | 19 | 16 | 16
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 11 | 19 | 16 | 9 | 14 | 18 | 14 | 18
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 13 | 12 | 12 | 8 | 12 | 14 | 12 | 13
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0012, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.75, 95% CI 2-sided [1.99 to 16.62]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.86, 95% CI 2-sided [3.06 to 25.68]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.55, 95% CI 2-sided [3.94 to 33.85]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 13.55, 95% CI 2-sided [4.55 to 40.38]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.0555, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.90, 95% CI 2-sided [0.98 to 8.61]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.98, 95% CI 2-sided [2.75 to 23.18]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.07, 95% CI 2-sided [2.81 to 23.19]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0012, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.55, 95% CI 2-sided [1.82 to 11.39]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0005, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.25, 95% CI 2-sided [2.06 to 13.43]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.62, 95% CI 2-sided [2.20 to 14.39]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.42, 95% CI 2-sided [2.99 to 23.74]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0277, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.74, 95% CI 2-sided [1.12 to 6.70]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0022, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.15, 95% CI 2-sided [1.66 to 10.32]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0314, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.06, 95% CI 2-sided [1.26 to 7.41]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0041, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.92, 95% CI 2-sided [1.54 to 9.97]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0028, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.19, 95% CI 2-sided [1.64 to 10.74]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0011, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.96, 95% CI 2-sided [1.90 to 12.98]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.79, 95% CI 2-sided [2.86 to 26.99]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0036, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.09, 95% CI 2-sided [1.59 to 10.57]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0018, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.52, 95% CI 2-sided [1.75 to 11.67]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0243, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.76, 95% CI 2-sided [1.14 to 6.68]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0770, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.33, 95% CI 2-sided [0.91 to 5.96]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0451, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.61, 95% CI 2-sided [1.02 to 6.69]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0165, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.36, 95% CI 2-sided [1.25 to 9.04]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0037, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.28, 95% CI 2-sided [1.72 to 16.23]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0812, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.90 to 5.82]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0577, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.46, 95% CI 2-sided [0.97 to 6.22]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0706, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.33, 95% CI 2-sided [0.93 to 5.85]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.0404, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.70, 95% CI 2-sided [1.04 to 7.00]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0054, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.30, 95% CI 2-sided [1.54 to 11.99]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0186, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.37, 95% CI 2-sided [1.22 to 9.27]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p = 0.0023, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.58, 95% CI 2-sided [1.96 to 22.14]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0118, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.63, 95% CI 2-sided [1.33 to 9.93]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0020, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.57, 95% CI 2-sided [1.88 to 16.53]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0430, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.71, 95% CI 2-sided [1.03 to 7.14]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.2197, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.70 to 4.66]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.1341, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.80 to 5.42]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0196, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.69, 95% CI 2-sided [1.23 to 11.05]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0121, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.79, 95% CI 2-sided [1.41 to 16.26]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.1511, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.77 to 5.56]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0068, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.94, 95% CI 2-sided [1.55 to 15.68]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0741, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.49, 95% CI 2-sided [0.91 to 6.79]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.2772, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.70, 95% CI 2-sided [0.65 to 4.43]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0705, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.55, 95% CI 2-sided [0.92 to 7.02]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0220, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.88, 95% CI 2-sided [1.22 to 12.39]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0196, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.33, 95% CI 2-sided [1.27 to 14.82]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0433, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.09, 95% CI 2-sided [1.03 to 9.24]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0355, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.15, 95% CI 2-sided [1.08 to 9.20]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.3238, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.62 to 4.28]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.3208, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.60 to 4.68]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.2281, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.67 to 5.40]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0566, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.18, 95% CI 2-sided [0.97 to 10.46]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.1491, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.39, 95% CI 2-sided [0.73 to 7.78]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.1477, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.32, 95% CI 2-sided [0.74 to 7.23]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0532, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.24, 95% CI 2-sided [0.98 to 10.64]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.1616, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.73 to 6.76]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.4320, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.55 to 4.11]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.2231, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.68 to 5.35]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0347, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.88, 95% CI 2-sided [1.10 to 13.64]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0291, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.59, 95% CI 2-sided [1.17 to 18.07]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.2805, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.61 to 5.38]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0602, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.10, 95% CI 2-sided [0.95 to 10.11]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.5087, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.51 to 3.88]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.1224, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.80 to 6.38]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.2280, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.68 to 5.02]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.1835, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.71 to 6.02]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0107, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.85, 95% CI 2-sided [1.51 to 22.69]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.0576, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.94, 95% CI 2-sided [0.97 to 8.96]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0047, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.68, 95% CI 2-sided [2.00 to 46.77]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0569, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.89, 95% CI 2-sided [0.97 to 8.64]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.1078, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.35, 95% CI 2-sided [0.83 to 6.68]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0772, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.60, 95% CI 2-sided [0.90 to 7.47]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.1311, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.36, 95% CI 2-sided [0.77 to 7.22]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.01255, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.64, 95% CI 2-sided [1.45 to 21.96]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0128, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.97, 95% CI 2-sided [1.41 to 17.54]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0079, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.32, 95% CI 2-sided [1.62 to 24.63]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0572, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.90, 95% CI 2-sided [0.97 to 8.67]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.0284, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.33, 95% CI 2-sided [1.14 to 9.79]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.0705, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.58, 95% CI 2-sided [0.92 to 7.22]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0136, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.81, 95% CI 2-sided [1.38 to 16.77]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0043, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.96, 95% CI 2-sided [2.06 to 48.29]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.0760, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.66, 95% CI 2-sided [0.90 to 7.83]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0059, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.75, 95% CI 2-sided [1.65 to 20.00]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0143, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.22, 95% CI 2-sided [1.33 to 13.35]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.2779, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.62 to 5.35]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.7559, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.41 to 3.41]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.9050, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.35 to 3.23]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.2163, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.05, 95% CI 2-sided [0.66 to 6.38]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.1713, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.24, 95% CI 2-sided [0.70 to 7.14]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.3981, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.52 to 5.09]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.9692, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.35 to 2.96]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.2978, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.60 to 5.22]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.8525, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.38 to 3.18]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.5028, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.21 to 2.13]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.4594, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.50 to 4.73]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.1124, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.56, 95% CI 2-sided [0.80 to 8.17]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.3415, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.55 to 5.58]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.3635, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.56 to 4.83]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.5716, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.24 to 2.20]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.5028, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.23 to 2.05]
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.3982, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.18 to 1.98]
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.93, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.30 to 2.87]
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.2364, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.12, 95% CI 2-sided [0.61 to 7.32]
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.7095, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.39 to 4.04]
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.6011, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.26 to 2.20]

18. Secondary Outcome: Number of Participants With Mean Percent Reduction of 70% in The Mean Frequency of Moderate and Severe Vasomotor Symptoms From Baseline to Each Study Week
Description: as for outcome 1
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 2 | 11 | 14 | 21 | 22 | 6 | 11 | 17
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 9 | 18 | 25 | 27 | 25 | 15 | 20 | 22
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 11 | 22 | 27 | 28 | 28 | 21 | 24 | 25
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 13 | 20 | 29 | 25 | 30 | 25 | 28 | 25
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 16 | 20 | 30 | 25 | 29 | 25 | 28 | 26
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 18 | 21 | 29 | 27 | 28 | 23 | 30 | 26
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 18 | 23 | 32 | 25 | 28 | 25 | 28 | 25
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 19 | 26 | 31 | 26 | 28 | 21 | 26 | 26
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 21 | 26 | 29 | 27 | 29 | 25 | 28 | 26
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 18 | 26 | 28 | 23 | 29 | 23 | 29 | 25
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 21 | 27 | 30 | 24 | 28 | 26 | 30 | 28
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 20 | 24 | 27 | 24 | 27 | 25 | 28 | 26
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 5 | 17 | 9 | 11 | 8 | 15 | 7 | 12
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 9 | 10 | 8 | 7 | 3 | 10 | 7 | 10
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 7 | 9 | 8 | 4 | 1 | 8 | 7 | 8
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0181, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.78, 95% CI 2-sided [1.39 to 33.10]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0039, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.97, 95% CI 2-sided [2.10 to 47.48]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 21.20, 95% CI 2-sided [4.51 to 99.65]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 23.97, 95% CI 2-sided [5.09 to 112.9]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.1766, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.17, 95% CI 2-sided [0.59 to 16.87]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0116, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.68, 95% CI 2-sided [1.58 to 37.43]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0013, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 12.74, 95% CI 2-sided [2.71 to 59.81]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0359, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.82, 95% CI 2-sided [1.07 to 7.43]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0004, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.80, 95% CI 2-sided [2.20 to 15.33]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.13, 95% CI 2-sided [2.68 to 18.98]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.84, 95% CI 2-sided [2.53 to 18.46]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.1540, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.04, 95% CI 2-sided [0.76 to 5.47]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0065, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.84, 95% CI 2-sided [1.46 to 10.12]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0052, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.90, 95% CI 2-sided [1.50 to 10.14]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0064, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.68, 95% CI 2-sided [1.44 to 9.39]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.86, 95% CI 2-sided [2.26 to 15.21]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.42, 95% CI 2-sided [2.47 to 16.69]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.21, 95% CI 2-sided [3.01 to 22.42]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0171, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.12, 95% CI 2-sided [1.22 to 7.97]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0020, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.38, 95% CI 2-sided [1.71 to 11.18]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0034, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.97, 95% CI 2-sided [1.58 to 9.99]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0399, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.63, 95% CI 2-sided [1.05 to 6.59]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.76, 95% CI 2-sided [2.23 to 14.84]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0031, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.05, 95% CI 2-sided [1.60 to 10.23]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.82, 95% CI 2-sided [3.41 to 28.28]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0036, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.96, 95% CI 2-sided [1.57 to 10.01]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0009, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.79, 95% CI 2-sided [1.89 to 12.11]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0091, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.33, 95% CI 2-sided [1.35 to 8.21]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.2043, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.73 to 4.34]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0012, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.70, 95% CI 2-sided [1.84 to 12.01]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0058, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.77, 95% CI 2-sided [1.47 to 9.70]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.07, 95% CI 2-sided [2.73 to 23.83]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0221, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.88, 95% CI 2-sided [1.16 to 7.12]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0034, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.00, 95% CI 2-sided [1.58 to 10.13]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0123, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.22, 95% CI 2-sided [1.29 to 8.04]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.3291, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.64 to 3.78]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0118, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.27, 95% CI 2-sided [1.30 to 8.21]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0058, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.93, 95% CI 2-sided [1.49 to 10.40]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0012, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.98, 95% CI 2-sided [2.03 to 17.65]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.1043, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.85 to 5.32]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0015, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.01, 95% CI 2-sided [1.85 to 13.54]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0658, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.33, 95% CI 2-sided [0.95 to 5.73]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.1253, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.82 to 4.98]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0013, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.01, 95% CI 2-sided [1.88 to 13.34]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0096, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.66, 95% CI 2-sided [1.37 to 9.75]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0012, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.06, 95% CI 2-sided [2.04 to 17.96]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0344, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.75, 95% CI 2-sided [1.08 to 7.02]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0045, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.07, 95% CI 2-sided [1.55 to 10.72]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0810, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.24, 95% CI 2-sided [0.91 to 5.55]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.0761, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.92 to 5.70]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0078, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.66, 95% CI 2-sided [1.41 to 9.51]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0253, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.99, 95% CI 2-sided [1.15 to 7.82]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0017, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.23, 95% CI 2-sided [1.99 to 19.55]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.3512, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.62 to 3.87]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0352, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.07 to 7.13]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0704, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.36, 95% CI 2-sided [0.93 to 5.97]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.1651, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.94, 95% CI 2-sided [0.76 to 4.93]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.0964, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.21, 95% CI 2-sided [0.87 to 5.62]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0276, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.12, 95% CI 2-sided [1.13 to 8.59]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0060, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.99, 95% CI 2-sided [1.58 to 15.70]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.1556, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.76 to 5.39]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0202, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.33, 95% CI 2-sided [1.21 to 9.18]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.2063, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.72 to 4.67]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.0383, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.70, 95% CI 2-sided [1.06 to 6.92]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.0118, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.46, 95% CI 2-sided [1.32 to 9.10]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0314, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.96, 95% CI 2-sided [1.10 to 7.97]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0010, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.80, 95% CI 2-sided [2.17 to 21.34]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.0956, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.24, 95% CI 2-sided [0.87 to 5.80]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0027, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.80, 95% CI 2-sided [1.72 to 13.40]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0660, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.94 to 6.14]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.0853, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.32, 95% CI 2-sided [0.89 to 6.05]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0159, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.49, 95% CI 2-sided [1.26 to 9.62]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.0303, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.27, 95% CI 2-sided [1.12 to 9.53]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0071, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.84, 95% CI 2-sided [1.54 to 15.28]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0621, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.60, 95% CI 2-sided [0.95 to 7.09]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0081, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.20, 95% CI 2-sided [1.45 to 12.15]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0533, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.64, 95% CI 2-sided [0.99 to 7.09]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.2666, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.66 to 4.42]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.0754, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.44, 95% CI 2-sided [0.91 to 6.52]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0313, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.27, 95% CI 2-sided [1.11 to 9.64]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0056, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.76, 95% CI 2-sided [1.67 to 19.88]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.0736, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.58, 95% CI 2-sided [0.91 to 7.28]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0184, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.51, 95% CI 2-sided [1.24 to 10.00]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.1187, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.18, 95% CI 2-sided [0.82 to 5.81]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.0299, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.80, 95% CI 2-sided [1.14 to 12.69]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.5989, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.40 to 4.89]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.1337, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.61, 95% CI 2-sided [0.74 to 9.14]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.4605, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.45 to 5.89]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.0188, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.48, 95% CI 2-sided [1.28 to 15.65]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.5854, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.39 to 5.42]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.1768, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.32, 95% CI 2-sided [0.68 to 7.86]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.8426, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.29 to 2.78]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.3017, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.17 to 1.73]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.5958, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.21 to 2.43]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.0515, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.05 to 1.01]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.9734, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.31 to 3.11]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.7969, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.25 to 2.93]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.6637, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.25 to 2.40]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.4921, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.53, 95% CI 2-sided [0.45 to 5.15]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.8910, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.33 to 3.64]
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.5881, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.16 to 2.78]
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.0523, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.11, 95% CI 2-sided [0.01 to 1.02]
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.4646, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.46 to 5.61]
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.5806, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.40 to 5.14]
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.9220, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.28 to 3.12]

19. Secondary Outcome: Number of Participants With Mean Percent Reduction of 90% in The Mean Frequency of Moderate and Severe Vasomotor Symptoms From Baseline to Each Study Week
Description: as for outcome 1
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 1 | 4 | 5 | 10 | 12 | 2 | 4 | 6
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 3 | 8 | 13 | 18 | 21 | 7 | 7 | 14
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 5 | 12 | 15 | 23 | 23 | 9 | 14 | 18
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 8 | 12 | 18 | 23 | 22 | 12 | 14 | 18
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 8 | 12 | 18 | 20 | 24 | 13 | 13 | 19
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 10 | 13 | 21 | 22 | 25 | 12 | 14 | 21
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 9 | 12 | 22 | 21 | 26 | 12 | 17 | 21
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 14 | 17 | 22 | 22 | 27 | 12 | 19 | 22
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 16 | 17 | 22 | 24 | 27 | 12 | 20 | 21
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 14 | 18 | 19 | 20 | 28 | 16 | 18 | 22
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 15 | 18 | 20 | 20 | 26 | 16 | 21 | 21
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 14 | 18 | 19 | 18 | 24 | 16 | 19 | 22
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 1 | 5 | 3 | 9 | 2 | 8 | 3 | 2
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 1 | 4 | 3 | 4 | 1 | 5 | 3 | 1
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 0 | 2 | 3 | 3 | 0 | 1 | 4 | 1
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.1933, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.45, 95% CI 2-sided [0.47 to 42.25]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.1240, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.61, 95% CI 2-sided [0.62 to 50.44]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p = 0.0140, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 14.16, 95% CI 2-sided [1.71 to 117.2]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p = 0.0075, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 17.50, 95% CI 2-sided [2.15 to 142.7]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.5853, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.98, 95% CI 2-sided [0.17 to 22.96]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.1596, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.00, 95% CI 2-sided [0.53 to 47.05]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0908, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.48, 95% CI 2-sided [0.74 to 56.51]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.1318, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.97, 95% CI 2-sided [0.72 to 12.19]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0093, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.99, 95% CI 2-sided [1.56 to 23.04]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0006, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.13, 95% CI 2-sided [2.69 to 38.22]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 15.63, 95% CI 2-sided [4.11 to 59.40]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.2054, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.53, 95% CI 2-sided [0.60 to 10.64]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.1592, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.80, 95% CI 2-sided [0.67 to 11.72]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0070, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.31, 95% CI 2-sided [1.66 to 24.07]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0392, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.39, 95% CI 2-sided [1.06 to 10.85]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0096, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.49, 95% CI 2-sided [1.44 to 13.96]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.11, 95% CI 2-sided [3.28 to 31.16]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.76, 95% CI 2-sided [3.75 to 36.90]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.2217, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.11, 95% CI 2-sided [0.64 to 7.03]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0131, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.26, 95% CI 2-sided [1.36 to 13.38]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0031, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.39, 95% CI 2-sided [1.76 to 16.46]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.1485, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.15, 95% CI 2-sided [0.76 to 6.10]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0128, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.54, 95% CI 2-sided [1.31 to 9.56]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.50, 95% CI 2-sided [2.37 to 17.81]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.42, 95% CI 2-sided [2.32 to 17.77]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.2354, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.87, 95% CI 2-sided [0.67 to 5.26]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0894, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.87 to 6.65]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0201, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.23, 95% CI 2-sided [1.20 to 8.67]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.1614, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.10, 95% CI 2-sided [0.74 to 5.94]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0123, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.57, 95% CI 2-sided [1.32 to 9.66]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0006, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.08, 95% CI 2-sided [2.17 to 17.03]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.82, 95% CI 2-sided [3.40 to 28.36]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.1609, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.75 to 5.81]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0930, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.42, 95% CI 2-sided [0.86 to 6.79]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0063, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.02, 95% CI 2-sided [1.48 to 10.91]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.2621, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.65 to 4.74]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0092, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.55, 95% CI 2-sided [1.37 to 9.21]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0007, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.69, 95% CI 2-sided [2.09 to 15.48]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.85, 95% CI 2-sided [3.08 to 25.43]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.4259, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.55 to 4.08]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.1334, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.79 to 5.74]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0120, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.39, 95% CI 2-sided [1.31 to 8.77]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.2443, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.66 to 5.10]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0022, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.60, 95% CI 2-sided [1.73 to 12.25]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0004, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.60, 95% CI 2-sided [2.35 to 18.58]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 12.17, 95% CI 2-sided [4.05 to 36.63]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.3101, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.70, 95% CI 2-sided [0.61 to 4.71]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0116, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.65, 95% CI 2-sided [1.34 to 10.00]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0045, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.15, 95% CI 2-sided [1.56 to 11.05]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.3505, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.62 to 3.88]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0739, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.28, 95% CI 2-sided [0.92 to 5.62]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0163, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.19, 95% CI 2-sided [1.24 to 8.20]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.49, 95% CI 2-sided [2.81 to 25.64]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.8358, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.35 to 2.35]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.1006, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.18, 95% CI 2-sided [0.86 to 5.52]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0484, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.01 to 6.34]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.6492, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.50 to 3.08]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.2230, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.71 to 4.27]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0126, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.43, 95% CI 2-sided [1.30 to 9.02]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0014, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.56, 95% CI 2-sided [1.94 to 15.98]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.4713, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.27 to 1.83]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.1397, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.79 to 5.12]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.2272, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.71 to 4.34]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.2024, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.72 to 4.64]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.1716, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.76 to 4.79]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0199, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.20, 95% CI 2-sided [1.20 to 8.51]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.45, 95% CI 2-sided [2.80 to 25.54]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.4243, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.57 to 3.77]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.1507, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.78 to 5.09]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0449, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.60, 95% CI 2-sided [1.02 to 6.60]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.2759, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.66 to 4.24]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.1700, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.76 to 4.78]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.0153, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.47, 95% CI 2-sided [1.27 to 9.51]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0009, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.04, 95% CI 2-sided [2.08 to 17.53]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.6228, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.50 to 3.23]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0460, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.02 to 6.76]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.1215, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.82 to 5.23]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.2470, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.68 to 4.48]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.2072, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.72 to 4.66]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0621, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.57, 95% CI 2-sided [0.95 to 6.94]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0016, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.67, 95% CI 2-sided [1.93 to 16.69]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.4372, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.56 to 3.84]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.1100, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.18, 95% CI 2-sided [0.84 to 5.66]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0533, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.55, 95% CI 2-sided [0.99 to 6.59]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.1769, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.68, 95% CI 2-sided [0.50 to 44.00]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.4942, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.22 to 23.53]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.0214, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 12.82, 95% CI 2-sided [1.46 to 112.7]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.6013, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.16 to 22.99]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.0537, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.60, 95% CI 2-sided [0.97 to 76.58]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.2662, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.80, 95% CI 2-sided [0.36 to 39.91]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.7431, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.13 to 17.84]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.2829, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.53, 95% CI 2-sided [0.35 to 35.22]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.5311, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.12, 95% CI 2-sided [0.20 to 22.29]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.1857, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.71, 95% CI 2-sided [0.47 to 46.83]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.9879, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.06 to 17.50]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.1853, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.57, 95% CI 2-sided [0.48 to 43.19]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.2170, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.43, 95% CI 2-sided [0.42 to 46.93]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.8354, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.04 to 12.62]

20. Secondary Outcome: Number of Participants With Mean Percent Reduction of 100% in The Mean Frequency of Moderate and Severe Vasomotor Symptoms From Baseline to Each Study Week
Description: as for outcome 1
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 1 | 1 | 0 | 3 | 3 | 0 | 1 | 0
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 1 | 2 | 3 | 7 | 10 | 0 | 4 | 6
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 1 | 5 | 6 | 9 | 12 | 4 | 6 | 12
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 1 | 3 | 8 | 10 | 14 | 4 | 8 | 9
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 4 | 5 | 8 | 10 | 15 | 6 | 7 | 8
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 1 | 8 | 10 | 12 | 16 | 5 | 6 | 15
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 1 | 7 | 10 | 14 | 16 | 9 | 10 | 15
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 4 | 9 | 12 | 16 | 16 | 6 | 9 | 15
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 5 | 9 | 12 | 15 | 18 | 5 | 12 | 15
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 7 | 9 | 11 | 16 | 19 | 6 | 9 | 17
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 5 | 9 | 11 | 15 | 19 | 10 | 9 | 15
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 9 | 8 | 12 | 14 | 16 | 9 | 14 | 13
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 0 | 1 | 2 | 6 | 1 | 3 | 1 | 1
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 1 | 1 | 2 | 2 | 0 | 2 | 1 | 0
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 0 | 1 | 2 | 3 | 0 | 1 | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.9671, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.06 to 16.04]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p = 0.3289, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.16, 95% CI 2-sided [0.31 to 31.87]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p = 0.3157, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.26, 95% CI 2-sided [0.32 to 32.71]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.991, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.06 to 16.83]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.5139, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.20 to 26.12]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.3079, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.32, 95% CI 2-sided [0.33 to 33.45]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0469, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.83, 95% CI 2-sided [1.03 to 75.68]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0134, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 14.39, 95% CI 2-sided [1.74 to 119.1]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.1606, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.98, 95% CI 2-sided [0.53 to 46.90]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0854, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.69, 95% CI 2-sided [0.77 to 58.35]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.1082, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.07, 95% CI 2-sided [0.67 to 54.72]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0737, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.22, 95% CI 2-sided [0.83 to 63.04]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0217, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.98, 95% CI 2-sided [1.44 to 99.74]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0058, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 19.24, 95% CI 2-sided [2.36 to 157.1]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.1924, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.44, 95% CI 2-sided [0.47 to 41.87]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0680, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.54, 95% CI 2-sided [0.86 to 66.00]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0095, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 15.95, 95% CI 2-sided [1.97 to 129.4]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.2690, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.68, 95% CI 2-sided [0.36 to 37.21]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0321, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.28, 95% CI 2-sided [1.22 to 86.53]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0131, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 14.48, 95% CI 2-sided [1.75 to 119.7]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0025, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 25.22, 95% CI 2-sided [3.11 to 204.6]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.1788, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.65, 95% CI 2-sided [0.49 to 43.72]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0320, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.33, 95% CI 2-sided [1.22 to 87.31]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0251, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.24, 95% CI 2-sided [1.35 to 93.33]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.6154, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.35 to 5.83]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.1906, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.65 to 8.63]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0450, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.67, 95% CI 2-sided [1.03 to 13.07]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p = 0.0017, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.19, 95% CI 2-sided [2.10 to 24.66]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.3939, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.47 to 6.97]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.2869, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.55 to 7.74]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.1817, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.66 to 8.80]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.0256, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.41, 95% CI 2-sided [1.35 to 96.77]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.0153, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 13.65, 95% CI 2-sided [1.65 to 112.8]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0042, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 21.76, 95% CI 2-sided [2.64 to 179.2]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0008, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 35.75, 95% CI 2-sided [4.39 to 291.5]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.0967, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.45, 95% CI 2-sided [0.71 to 58.21]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0564, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.30, 95% CI 2-sided [0.94 to 72.95]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0030, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 23.63, 95% CI 2-sided [2.93 to 190.5]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.0384, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.72, 95% CI 2-sided [1.13 to 83.68]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0153, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 13.65, 95% CI 2-sided [1.65 to 112.9]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0015, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 30.55, 95% CI 2-sided [3.72 to 250.6]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0008, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 35.99, 95% CI 2-sided [4.41 to 293.5]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.0192, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 12.67, 95% CI 2-sided [1.51 to 106.1]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0089, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 16.92, 95% CI 2-sided [2.03 to 141.0]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0025, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 24.96, 95% CI 2-sided [3.09 to 201.6]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.0910, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.03, 95% CI 2-sided [0.84 to 10.94]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0296, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.96, 95% CI 2-sided [1.15 to 13.67]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0009, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.23, 95% CI 2-sided [2.38 to 28.44]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0007, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.54, 95% CI 2-sided [2.46 to 29.63]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.4152, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.45 to 6.86]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0700, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.29, 95% CI 2-sided [0.91 to 11.93]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0048, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.83, 95% CI 2-sided [1.71 to 19.84]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.1497, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.44, 95% CI 2-sided [0.72 to 8.23]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.0608, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.05, 95% CI 2-sided [0.95 to 9.77]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0028, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.99, 95% CI 2-sided [1.85 to 19.34]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0005, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.84, 95% CI 2-sided [2.45 to 25.13]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.8393, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.30 to 4.39]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0215, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.01, 95% CI 2-sided [1.23 to 13.10]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0112, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.42, 95% CI 2-sided [1.40 to 13.94]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.3498, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.55 to 5.29]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.1981, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.05, 95% CI 2-sided [0.69 to 6.08]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0029, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.28, 95% CI 2-sided [1.76 to 15.78]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0011, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.95, 95% CI 2-sided [2.03 to 17.40]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.9511, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.29 to 3.23]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.3241, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.57 to 5.45]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0111, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.90, 95% CI 2-sided [1.36 to 11.16]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.1375, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.51, 95% CI 2-sided [0.74 to 8.48]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.0670, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.02, 95% CI 2-sided [0.93 to 9.83]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.0009, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.57, 95% CI 2-sided [2.29 to 25.04]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.42, 95% CI 2-sided [2.91 to 30.49]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0982, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.75, 95% CI 2-sided [0.83 to 9.14]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.1233, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.60, 95% CI 2-sided [0.77 to 8.80]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0091, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.63, 95% CI 2-sided [1.46 to 14.64]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.9620, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.34 to 3.10]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.3527, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.58 to 4.59]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0394, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.04, 95% CI 2-sided [1.06 to 8.76]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0224, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.36, 95% CI 2-sided [1.19 to 9.53]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.7891, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.39 to 3.44]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0851, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.48, 95% CI 2-sided [0.88 to 6.99]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.2885, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.63 to 4.83]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.8611, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.05 to 13.30]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.7549, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.13 to 17.42]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.5658, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.17 to 24.66]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.6319, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.15 to 21.86]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.9526, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.06 to 18.96]

21. Secondary Outcome: Number of Participants With Absolute Reduction of 2 in Mean Number of Mild, Moderate and Severe VMS Per Day From Baseline to Each Study Week
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 20 | 27 | 32 | 35 | 33 | 23 | 34 | 32
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 28 | 34 | 32 | 38 | 33 | 32 | 36 | 33
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 29 | 33 | 35 | 37 | 35 | 34 | 35 | 39
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 30 | 31 | 34 | 35 | 35 | 33 | 40 | 39
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 33 | 34 | 38 | 33 | 34 | 36 | 38 | 36
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 33 | 36 | 37 | 33 | 33 | 33 | 37 | 39
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 32 | 34 | 36 | 32 | 33 | 32 | 37 | 38
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 34 | 35 | 36 | 34 | 32 | 33 | 37 | 37
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 33 | 34 | 37 | 33 | 33 | 32 | 37 | 37
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 34 | 34 | 32 | 29 | 33 | 33 | 36 | 36
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 34 | 33 | 34 | 27 | 31 | 33 | 36 | 36
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 31 | 34 | 31 | 28 | 31 | 31 | 35 | 35
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 17 | 30 | 26 | 22 | 22 | 21 | 25 | 28
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 17 | 22 | 26 | 16 | 21 | 20 | 21 | 25
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 18 | 18 | 20 | 12 | 20 | 12 | 16 | 22
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.2251, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.71 to 4.26]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0084, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.57, 95% CI 2-sided [1.39 to 9.20]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p = 0.0007, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.71, 95% CI 2-sided [2.09 to 15.62]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p = 0.0015, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.11, 95% CI 2-sided [1.87 to 14.00]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.6976, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.48 to 2.95]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0021, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.57, 95% CI 2-sided [1.73 to 12.05]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0171, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.06, 95% CI 2-sided [1.22 to 7.68]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.2224, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.86, 95% CI 2-sided [0.69 to 5.04]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.2716, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.65 to 4.69]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0112, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.49, 95% CI 2-sided [1.41 to 14.32]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0461, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.08, 95% CI 2-sided [1.02 to 9.31]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.3463, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.59 to 4.47]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0419, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.05, 95% CI 2-sided [1.04 to 8.92]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.2977, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.63 to 4.46]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.2300, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.87, 95% CI 2-sided [0.67 to 5.21]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0655, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.83, 95% CI 2-sided [0.94 to 8.58]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0245, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.79, 95% CI 2-sided [1.19 to 12.11]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0129, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.62, 95% CI 2-sided [1.44 to 21.93]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.1259, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.79 to 7.15]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.1015, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.40, 95% CI 2-sided [0.84 to 6.82]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0167, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.48, 95% CI 2-sided [1.31 to 15.33]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.5232, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.50 to 3.95]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.2055, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.68 to 5.82]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0658, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.00, 95% CI 2-sided [0.93 to 9.64]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0136, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.34, 95% CI 2-sided [1.51 to 35.75]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.3238, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.59 to 5.00]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0118, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.86, 95% CI 2-sided [1.48 to 23.21]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0163, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.29, 95% CI 2-sided [1.36 to 20.62]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.6363, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.42 to 4.18]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0722, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.68, 95% CI 2-sided [0.89 to 15.25]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.2019, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.35, 95% CI 2-sided [0.63 to 8.73]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p = 0.0337, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.15, 95% CI 2-sided [1.20 to 86.09]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.2207, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.61 to 8.24]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0849, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.50, 95% CI 2-sided [0.84 to 14.57]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0844, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.47, 95% CI 2-sided [0.84 to 14.24]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.2383, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.15, 95% CI 2-sided [0.60 to 7.65]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.1653, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.55, 95% CI 2-sided [0.68 to 9.58]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.1836, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.48, 95% CI 2-sided [0.65 to 9.48]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0529, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.30, 95% CI 2-sided [0.97 to 70.80]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.3197, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.52 to 7.27]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0376, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.88, 95% CI 2-sided [1.11 to 31.25]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0343, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.08, 95% CI 2-sided [1.19 to 85.64]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.4435, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.49 to 5.09]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.1805, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.67 to 8.13]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0857, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.54, 95% CI 2-sided [0.84 to 14.95]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0316, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.50, 95% CI 2-sided [1.23 to 89.63]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.3471, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.52 to 6.27]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0313, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.15, 95% CI 2-sided [1.18 to 32.09]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0208, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 12.49, 95% CI 2-sided [1.47 to 106.3]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.8669, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.31 to 3.97]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.6592, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.37 to 4.89]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.2923, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.23, 95% CI 2-sided [0.50 to 9.98]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.1145, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.78, 95% CI 2-sided [0.65 to 51.04]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.4470, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.40 to 7.78]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0753, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.31, 95% CI 2-sided [0.82 to 65.41]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0829, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.85, 95% CI 2-sided [0.78 to 60.24]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.9978, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.28 to 3.59]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.4571, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.43 to 6.65]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.3681, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.44 to 8.94]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.1038, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.12, 95% CI 2-sided [0.69 to 54.38]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.4639, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.39 to 7.72]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0770, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.15, 95% CI 2-sided [0.81 to 63.27]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.9838, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.26 to 4.01]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.6995, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.21 to 2.86]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.8808, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.26 to 4.71]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.1570, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.94, 95% CI 2-sided [0.54 to 45.13]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.3742, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.19, 95% CI 2-sided [0.39 to 12.26]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.1436, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.24, 95% CI 2-sided [0.57 to 48.26]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.1277, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.57, 95% CI 2-sided [0.61 to 50.77]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.6689, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.20 to 2.81]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.8019, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.29 to 4.95]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.9591, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.23 to 4.05]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.3364, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.33, 95% CI 2-sided [0.42 to 13.06]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.3698, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.39 to 12.32]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.1587, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.92, 95% CI 2-sided [0.54 to 45.01]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.1300, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.50, 95% CI 2-sided [0.61 to 50.06]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.4152, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.43 to 7.53]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.9645, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.27 to 3.50]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.3884, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.43 to 8.96]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.2670, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.62, 95% CI 2-sided [0.48 to 14.41]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0861, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.91, 95% CI 2-sided [0.76 to 62.90]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0774, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.21, 95% CI 2-sided [0.80 to 64.66]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.0389, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.73, 95% CI 2-sided [1.08 to 20.65]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.3695, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.50 to 6.57]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.3501, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.48 to 7.89]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.2021, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.49, 95% CI 2-sided [0.61 to 10.14]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.6201, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.36 to 5.62]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.0235, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 13.71, 95% CI 2-sided [1.42 to 132.0]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.0929, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.43, 95% CI 2-sided [0.81 to 14.48]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.9820, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.29 to 3.33]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.4956, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.44 to 5.41]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.5708, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.20 to 2.44]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.1985, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.55, 95% CI 2-sided [0.61 to 10.61]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.8368, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.31 to 4.32]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.1397, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.18, 95% CI 2-sided [0.68 to 14.76]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.0366, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.52 to 6.85]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.7968, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.23 to 3.05]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.9074, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.30 to 3.81]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.1987, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.10 to 1.60]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.2040, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.58, 95% CI 2-sided [0.60 to 11.18]
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.3318, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.13 to 1.99]
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.7437, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.31 to 5.10]
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.6848, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.36 to 4.71]

22. Secondary Outcome: Number of Participants With Absolute Reduction of 3 in Mean Number of Mild, Moderate and Severe VMS Per Day From Baseline to Each Study Week
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 14 | 23 | 29 | 32 | 28 | 18 | 31 | 29
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 19 | 30 | 30 | 36 | 32 | 28 | 33 | 31
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 24 | 31 | 30 | 36 | 34 | 29 | 34 | 32
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 26 | 30 | 32 | 34 | 34 | 29 | 35 | 34
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 29 | 31 | 36 | 33 | 33 | 34 | 35 | 33
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 28 | 29 | 33 | 31 | 32 | 30 | 36 | 38
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 30 | 31 | 34 | 30 | 32 | 31 | 37 | 38
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 31 | 32 | 34 | 32 | 29 | 31 | 37 | 34
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 30 | 32 | 33 | 32 | 32 | 31 | 36 | 34
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 29 | 32 | 29 | 29 | 31 | 31 | 36 | 34
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 30 | 31 | 30 | 27 | 30 | 32 | 36 | 34
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 28 | 31 | 31 | 27 | 28 | 30 | 34 | 33
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 16 | 24 | 20 | 21 | 18 | 20 | 19 | 26
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 15 | 18 | 21 | 15 | 17 | 17 | 18 | 23
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 17 | 15 | 18 | 12 | 13 | 11 | 14 | 17
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.1114, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.12, 95% CI 2-sided [0.84 to 5.32]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0013, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.69, 95% CI 2-sided [1.83 to 12.04]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.01, 95% CI 2-sided [2.65 to 18.54]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p = 0.0010, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.96, 95% CI 2-sided [1.91 to 12.89]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.6384, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.49 to 3.22]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.77, 95% CI 2-sided [2.23 to 14.93]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0025, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.15, 95% CI 2-sided [1.65 to 10.45]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0279, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.82, 95% CI 2-sided [1.12 to 7.12]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0114, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.36, 95% CI 2-sided [1.31 to 8.61]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.55, 95% CI 2-sided [2.66 to 21.45]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0005, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.41, 95% CI 2-sided [2.25 to 18.26]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0695, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.93 to 6.02]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0015, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.83, 95% CI 2-sided [1.83 to 12.77]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0120, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.28, 95% CI 2-sided [1.30 to 8.28]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.662, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.49, 95% CI 2-sided [0.94 to 6.57]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.1019, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.85 to 5.80]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0023, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.44, 95% CI 2-sided [1.83 to 16.18]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0015, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.33, 95% CI 2-sided [2.15 to 25.02]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.2380, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.68 to 4.66]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0120, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.61, 95% CI 2-sided [1.33 to 9.81]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0910, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.88 to 5.77]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.1926, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.72 to 5.18]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.1017, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.85 to 6.15]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0153, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.85, 95% CI 2-sided [1.29 to 11.45]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0034, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.52, 95% CI 2-sided [1.95 to 28.98]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.4539, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.55 to 3.76]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0327, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.03, 95% CI 2-sided [1.10 to 8.40]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0555, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.67, 95% CI 2-sided [0.98 to 7.30]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.3505, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.58 to 4.67]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0265, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.92, 95% CI 2-sided [1.17 to 13.11]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0174, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.77, 95% CI 2-sided [1.32 to 17.32]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p = 0.0075, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.95, 95% CI 2-sided [1.80 to 44.61]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.1228, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.46, 95% CI 2-sided [0.78 to 7.68]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0431, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.28, 95% CI 2-sided [1.04 to 10.38]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0851, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.70, 95% CI 2-sided [0.87 to 8.35]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.4726, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.53 to 3.99]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.1289, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.79 to 6.67]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0400, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.39, 95% CI 2-sided [1.06 to 10.84]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0097, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.22, 95% CI 2-sided [1.67 to 40.55]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.2260, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.66 to 5.94]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0031, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.63, 95% CI 2-sided [2.07 to 35.96]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0043, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.16, 95% CI 2-sided [2.07 to 49.90]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.5571, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.47 to 4.04]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.1911, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.69 to 6.59]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.1101, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.74, 95% CI 2-sided [0.80 to 9.41]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0199, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.86, 95% CI 2-sided [1.36 to 34.74]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.2600, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.96, 95% CI 2-sided [0.61 to 6.33]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0090, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.93, 95% CI 2-sided [1.73 to 46.19]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0089, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 17.22, 95% CI 2-sided [2.04 to 145.2]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.8966, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.36 to 3.19]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.5031, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.48 to 4.51]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.2603, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.59 to 6.92]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.2447, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.16, 95% CI 2-sided [0.59 to 7.88]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.4239, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.49 to 5.55]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0240, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.72, 95% CI 2-sided [1.38 to 99.35]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.1457, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.60, 95% CI 2-sided [0.72 to 9.41]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.9000, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.34 to 3.38]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.7644, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.39 to 3.64]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.2245, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.60 to 8.67]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0475, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.28, 95% CI 2-sided [1.02 to 27.40]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.2569, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.15, 95% CI 2-sided [0.57 to 8.07]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0412, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.32, 95% CI 2-sided [1.09 to 79.44]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.1201, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.84, 95% CI 2-sided [0.76 to 10.61]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.3814, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.53 to 5.23]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.8549, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.38 to 3.23]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.1274, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.77, 95% CI 2-sided [0.75 to 10.24]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0703, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.67, 95% CI 2-sided [0.90 to 15.01]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.1821, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.66 to 8.76]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0187, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 12.96, 95% CI 2-sided [1.53 to 109.5]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0458, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.18, 95% CI 2-sided [1.03 to 17.00]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.6806, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.41 to 3.89]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.8090, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.38 to 3.45]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.2352, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.60 to 8.26]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.1231, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.04, 95% CI 2-sided [0.74 to 12.50]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.1445, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.86, 95% CI 2-sided [0.70 to 11.76]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0230, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 12.03, 95% CI 2-sided [1.41 to 102.7]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0801, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.51, 95% CI 2-sided [0.86 to 14.36]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.4152, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.50 to 5.32]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.3845, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.70, 95% CI 2-sided [0.51 to 5.65]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.1864, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.46, 95% CI 2-sided [0.65 to 9.39]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.01268, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.06, 95% CI 2-sided [0.73 to 12.86]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.1600, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.80, 95% CI 2-sided [0.67 to 11.76]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0317, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.13, 95% CI 2-sided [1.17 to 32.11]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0709, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.73, 95% CI 2-sided [0.89 to 15.53]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.4533, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.47 to 5.41]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.7053, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.24 to 2.60]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.3677, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.49 to 6.99]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.7350, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.35 to 4.40]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.6443, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.36 to 5.15]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.4865, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.43 to 5.76]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.1628, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.52, 95% CI 2-sided [0.69 to 9.27]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.6935, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.24 to 2.57]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.9753, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.32 to 3.28]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.7407, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.23 to 2.81]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.4929, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.44 to 5.49]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.8496, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.25 to 3.15]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.3248, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.92, 95% CI 2-sided [0.52 to 7.05]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.2589, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.59 to 6.92]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.3318, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.16 to 1.87]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.8536, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.26 to 3.01]
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.2817, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.12 to 1.84]
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.4091, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.17 to 2.07]
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.3147, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.13 to 1.93]
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.8547, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.24 to 3.24]
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.5023, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.20 to 2.19]

23. Secondary Outcome: Number of Participants With Absolute Reduction of 4 in Mean Number of Mild, Moderate and Severe VMS Per Day From Baseline to Each Study Week
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 8 | 21 | 21 | 26 | 24 | 16 | 22 | 29
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 16 | 27 | 29 | 33 | 28 | 25 | 27 | 26
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 18 | 28 | 27 | 33 | 31 | 26 | 33 | 31
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 22 | 27 | 28 | 31 | 30 | 26 | 32 | 31
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 24 | 28 | 31 | 30 | 33 | 28 | 34 | 31
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 27 | 28 | 27 | 31 | 30 | 26 | 34 | 33
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 27 | 27 | 32 | 30 | 30 | 26 | 33 | 32
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 28 | 29 | 32 | 31 | 29 | 28 | 34 | 30
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 28 | 30 | 31 | 32 | 31 | 28 | 35 | 32
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 27 | 29 | 27 | 28 | 30 | 30 | 34 | 31
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 27 | 28 | 28 | 26 | 30 | 30 | 35 | 31
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 25 | 26 | 28 | 27 | 27 | 27 | 33 | 32
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 12 | 20 | 16 | 18 | 17 | 18 | 17 | 23
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 14 | 16 | 17 | 12 | 13 | 16 | 15 | 18
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 15 | 14 | 13 | 9 | 12 | 10 | 12 | 13
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0093, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.99, 95% CI 2-sided [1.41 to 11.35]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0035, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.66, 95% CI 2-sided [1.66 to 13.09]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.48, 95% CI 2-sided [3.01 to 23.90]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.57, 95% CI 2-sided [2.65 to 21.59]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.1664, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.73 to 6.22]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0012, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.39, 95% CI 2-sided [1.94 to 14.96]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.85, 95% CI 2-sided [3.49 to 27.86]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0334, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.73, 95% CI 2-sided [1.08 to 6.89]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0034, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.12, 95% CI 2-sided [1.60 to 10.62]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.55, 95% CI 2-sided [2.45 to 17.47]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0014, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.90, 95% CI 2-sided [1.85 to 12.98]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0872, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.89 to 5.74]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0131, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.19, 95% CI 2-sided [1.28 to 7.98]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0386, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.60, 95% CI 2-sided [1.05 to 6.43]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0191, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.11, 95% CI 2-sided [1.20 to 8.05]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0291, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.84, 95% CI 2-sided [1.11 to 7.26]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0004, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.09, 95% CI 2-sided [2.23 to 16.58]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.24, 95% CI 2-sided [2.49 to 21.02]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0992, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.86 to 5.72]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0006, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.66, 95% CI 2-sided [2.11 to 15.16]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0060, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.74, 95% CI 2-sided [1.46 to 9.59]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.1472, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.78 to 5.14]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.1284, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.05, 95% CI 2-sided [0.81 to 5.15]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0117, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.55, 95% CI 2-sided [1.32 to 9.50]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0067, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.24, 95% CI 2-sided [1.49 to 12.03]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.4088, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.59 to 3.71]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0194, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.09, 95% CI 2-sided [1.20 to 7.96]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0423, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.03 to 6.73]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.2151, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.86, 95% CI 2-sided [0.70 to 4.99]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0531, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.71, 95% CI 2-sided [0.99 to 7.42]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0118, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.11, 95% CI 2-sided [1.37 to 12.34]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.0006, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 16.28, 95% CI 2-sided [3.29 to 80.46]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.3698, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.59 to 4.22]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0059, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.58, 95% CI 2-sided [1.55 to 13.53]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0241, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.32, 95% CI 2-sided [1.17 to 9.44]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.5308, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.50 to 3.77]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.8603, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.41 to 2.90]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0264, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.73, 95% CI 2-sided [1.17 to 11.95]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0188, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.60, 95% CI 2-sided [1.29 to 16.42]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.7642, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.42 to 3.27]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0101, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.91, 95% CI 2-sided [1.46 to 16.53]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0572, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.88, 95% CI 2-sided [0.97 to 8.55]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.7348, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.44 to 3.20]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.1397, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.77 to 6.25]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0231, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.07, 95% CI 2-sided [1.21 to 13.64]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0196, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.54, 95% CI 2-sided [1.27 to 16.15]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.7703, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.42 to 3.24]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0222, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.83, 95% CI 2-sided [1.21 to 12.12]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0668, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.77, 95% CI 2-sided [0.93 to 8.21]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.7533, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.43 to 3.22]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.3325, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.59 to 4.73]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0899, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.71, 95% CI 2-sided [0.86 to 8.57]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0642, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.31, 95% CI 2-sided [0.93 to 11.79]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.5964, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.46 to 3.89]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0224, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.43, 95% CI 2-sided [1.23 to 15.91]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.3139, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.60 to 4.96]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.6343, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.45 to 3.76]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.6557, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.45 to 3.61]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0516, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.66, 95% CI 2-sided [0.99 to 13.51]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0400, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.38, 95% CI 2-sided [1.07 to 17.91]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.5825, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.44 to 4.24]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0152, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.46, 95% CI 2-sided [1.47 to 37.83]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.1565, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.30, 95% CI 2-sided [0.73 to 7.30]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.4932, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.50 to 4.25]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.8504, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.39 to 3.12]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0759, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.07, 95% CI 2-sided [0.89 to 10.61]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0477, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.69, 95% CI 2-sided [1.01 to 13.46]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.1448, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.47, 95% CI 2-sided [0.73 to 8.36]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0173, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.54, 95% CI 2-sided [1.35 to 22.71]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.1101, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.57, 95% CI 2-sided [0.81 to 8.17]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.6022, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.46 to 3.78]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.6128, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.46 to 3.73]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.1001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.82, 95% CI 2-sided [0.82 to 9.68]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0255, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.95, 95% CI 2-sided [1.22 to 20.12]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.1521, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.42, 95% CI 2-sided [0.72 to 8.10]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0071, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.37, 95% CI 2-sided [1.84 to 47.69]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.1150, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.52, 95% CI 2-sided [0.80 to 7.93]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.8101, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.40 to 3.22]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.4663, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.51 to 4.33]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0453, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.80, 95% CI 2-sided [1.03 to 14.01]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0659, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.36, 95% CI 2-sided [0.92 to 12.21]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.3117, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.57 to 5.86]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0129, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.02, 95% CI 2-sided [1.46 to 24.73]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0303, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.12, 95% CI 2-sided [1.14 to 14.83]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.2772, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.94, 95% CI 2-sided [0.59 to 6.42]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.9432, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.29 to 3.16]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.2577, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.59 to 7.36]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.1496, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.55, 95% CI 2-sided [0.71 to 9.12]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.2874, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.05, 95% CI 2-sided [0.55 to 7.67]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.1981, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.65 to 7.78]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.0531, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.35, 95% CI 2-sided [0.98 to 11.43]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.5858, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.22 to 2.35]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.5122, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.21 to 2.16]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.3415, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.16 to 1.89]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.8263, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.25 to 2.98]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.8085, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.24 to 3.03]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.6745, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.38 to 4.43]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.9019, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.34 to 3.45]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.4425, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.18 to 2.10]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.3106, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.17 to 1.77]
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.0912, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.08 to 1.20]
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.5681, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.20 to 2.41]
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.4261, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.15 to 2.21]
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.7514, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.24 to 2.82]
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.2712, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.16 to 1.67]

24. Secondary Outcome: Number of Participants With Absolute Reduction of 5 in Mean Number of Mild, Moderate and Severe VMS Per Day From Baseline to Each Study Week
Description: as for outcome 13
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 5 | 17 | 19 | 22 | 21 | 13 | 18 | 20
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 14 | 25 | 24 | 27 | 24 | 21 | 23 | 26
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 16 | 25 | 25 | 29 | 27 | 25 | 29 | 27
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 17 | 24 | 26 | 25 | 28 | 24 | 31 | 27
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 20 | 24 | 26 | 26 | 28 | 26 | 32 | 28
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 22 | 24 | 25 | 30 | 27 | 25 | 30 | 30
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 22 | 27 | 27 | 27 | 28 | 24 | 28 | 30
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 22 | 26 | 26 | 28 | 26 | 23 | 31 | 30
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 26 | 25 | 26 | 28 | 28 | 23 | 32 | 30
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 22 | 26 | 23 | 25 | 29 | 25 | 32 | 30
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 24 | 27 | 25 | 24 | 27 | 27 | 33 | 30
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 23 | 23 | 26 | 22 | 26 | 24 | 31 | 29
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 9 | 18 | 13 | 14 | 14 | 17 | 13 | 17
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 10 | 15 | 12 | 10 | 9 | 16 | 13 | 14
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 11 | 11 | 9 | 8 | 7 | 9 | 11 | 12
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0103, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.89, 95% CI 2-sided [1.46 to 16.40]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0011, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.19, 95% CI 2-sided [2.20 to 23.48]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.06, 95% CI 2-sided [3.41 to 35.86]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.48, 95% CI 2-sided [3.18 to 34.55]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.1571, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.46, 95% CI 2-sided [0.71 to 8.55]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0010, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.14, 95% CI 2-sided [2.21 to 23.04]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0008, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.35, 95% CI 2-sided [2.29 to 23.61]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0342, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.78, 95% CI 2-sided [1.08 to 7.18]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0231, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.98, 95% CI 2-sided [1.16 to 7.66]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0032, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.12, 95% CI 2-sided [1.60 to 10.55]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0059, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.89, 95% CI 2-sided [1.48 to 10.22]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.2471, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.68 to 4.59]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0381, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.66, 95% CI 2-sided [1.05 to 6.70]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0113, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.34, 95% CI 2-sided [1.31 to 8.48]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0486, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.56, 95% CI 2-sided [1.01 to 6.52]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0350, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.71, 95% CI 2-sided [1.07 to 6.87]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0027, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.24, 95% CI 2-sided [1.65 to 10.90]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0020, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.68, 95% CI 2-sided [1.76 to 12.47]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0686, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.94 to 6.19]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0034, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.02, 95% CI 2-sided [1.58 to 10.21]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0222, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.90, 95% CI 2-sided [1.16 to 7.22]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0876, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.28, 95% CI 2-sided [0.89 to 5.84]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0345, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.72, 95% CI 2-sided [1.08 to 6.88]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0319, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.76, 95% CI 2-sided [1.09 to 6.99]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0013, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.27, 95% CI 2-sided [1.92 to 14.47]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.1751, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.75 to 4.87]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0019, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.46, 95% CI 2-sided [1.73 to 11.50]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0284, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.79, 95% CI 2-sided [1.11 to 6.97]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.2650, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.66 to 4.45]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.1238, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.10, 95% CI 2-sided [0.82 to 5.38]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0219, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.22, 95% CI 2-sided [1.18 to 8.74]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p = 0.0022, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.46, 95% CI 2-sided [1.84 to 16.16]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.2230, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.69 to 4.77]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0018, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.05, 95% CI 2-sided [1.83 to 13.97]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0205, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.17, 95% CI 2-sided [1.19 to 8.42]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.4628, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.54 to 3.81]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.4015, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.58 to 3.92]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0031, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.39, 95% CI 2-sided [1.76 to 16.47]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0115, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.15, 95% CI 2-sided [1.38 to 12.50]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.2513, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.66 to 4.98]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0099, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.94, 95% CI 2-sided [1.39 to 11.14]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0242, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.19, 95% CI 2-sided [1.16 to 8.74]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.1518, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.77 to 5.60]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.1811, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.73 to 5.17]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0150, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.88, 95% CI 2-sided [1.30 to 11.55]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0046, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.28, 95% CI 2-sided [1.67 to 16.68]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.3788, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.57 to 4.34]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0424, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.82, 95% CI 2-sided [1.04 to 7.70]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0139, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.69, 95% CI 2-sided [1.30 to 10.43]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.3057, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.63 to 4.42]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.3717, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.59 to 4.02]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0252, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.32, 95% CI 2-sided [1.16 to 9.50]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0235, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.56, 95% CI 2-sided [1.19 to 10.69]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.6580, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.46 to 3.39]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0061, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.58, 95% CI 2-sided [1.54 to 13.62]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0149, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.70, 95% CI 2-sided [1.29 to 10.61]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.9282, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.35 to 2.62]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.7902, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.33 to 2.35]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.1603, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.73 to 6.74]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.1144, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.55, 95% CI 2-sided [0.80 to 8.14]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.5903, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.26 to 2.13]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0290, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.89, 95% CI 2-sided [1.15 to 13.16]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.1721, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.12, 95% CI 2-sided [0.72 to 6.26]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.2439, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.66 to 5.09]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.7402, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.44 to 3.19]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0422, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.17, 95% CI 2-sided [1.04 to 9.63]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0061, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.44, 95% CI 2-sided [1.62 to 18.27]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.3191, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.59 to 4.92]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0037, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.91, 95% CI 2-sided [1.78 to 19.66]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0139, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.02, 95% CI 2-sided [1.33 to 12.20]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.3757, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.57 to 4.42]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.7087, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.45 to 3.28]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.1083, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.53, 95% CI 2-sided [0.81 to 7.88]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0473, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.21, 95% CI 2-sided [1.01 to 10.14]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.2481, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.89, 95% CI 2-sided [0.64 to 5.60]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0066, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.84, 95% CI 2-sided [1.64 to 20.89]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0466, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.06, 95% CI 2-sided [1.02 to 9.18]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.8769, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.34 to 2.53]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.5448, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.49 to 3.82]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.4125, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.53 to 4.64]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0500, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.36, 95% CI 2-sided [1.00 to 11.30]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.6167, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.45 to 3.87]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0233, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.00, 95% CI 2-sided [1.21 to 13.26]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0803, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.68, 95% CI 2-sided [0.89 to 8.09]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.1274, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.64, 95% CI 2-sided [0.76 to 9.18]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.9445, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.29 to 3.71]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.4204, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.69, 95% CI 2-sided [0.47 to 6.03]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.1315, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.78, 95% CI 2-sided [0.74 to 10.49]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.0944, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.24, 95% CI 2-sided [0.82 to 12.87]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.2801, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.57 to 6.89]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.1524, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.44, 95% CI 2-sided [0.72 to 8.30]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.6129, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.40 to 4.75]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.4617, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.18 to 2.18]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.6519, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.20 to 2.70]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.8011, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.22 to 3.18]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.3254, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.51 to 7.41]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.2730, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.58 to 6.94]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.6601, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.39 to 4.41]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.6588, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.20 to 2.76]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.3257, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.14 to 1.92]
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.2229, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.10 to 1.69]
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.2425, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.10 to 1.77]
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.9672, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.23 to 4.11]
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.5838, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.40 to 5.09]
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.9361, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.28 to 3.24]

25. Secondary Outcome: Number of Participants With Absolute Reduction of 2 in Mean Number of Moderate and Severe VMS Per Day From Baseline to Each Study Week
Description: as for outcome 1
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 22 | 33 | 32 | 35 | 36 | 28 | 34 | 32
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 30 | 36 | 33 | 37 | 36 | 36 | 38 | 33
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 31 | 33 | 36 | 36 | 36 | 37 | 37 | 39
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 31 | 34 | 34 | 34 | 36 | 36 | 40 | 39
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 32 | 34 | 39 | 32 | 35 | 37 | 39 | 35
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 33 | 36 | 37 | 32 | 33 | 34 | 37 | 38
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 33 | 35 | 36 | 31 | 34 | 34 | 37 | 38
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 35 | 36 | 36 | 32 | 33 | 35 | 37 | 37
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 33 | 35 | 37 | 31 | 33 | 34 | 37 | 37
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 34 | 35 | 32 | 28 | 33 | 34 | 36 | 35
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 34 | 35 | 34 | 26 | 32 | 34 | 36 | 36
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 31 | 35 | 31 | 27 | 31 | 32 | 35 | 35
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 17 | 29 | 27 | 21 | 24 | 24 | 22 | 27
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 17 | 23 | 26 | 17 | 20 | 23 | 22 | 25
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 18 | 19 | 22 | 14 | 19 | 14 | 17 | 21
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0429, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.60, 95% CI 2-sided [1.03 to 6.55]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0296, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.81, 95% CI 2-sided [1.11 to 7.12]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p = 0.0032, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.48, 95% CI 2-sided [1.65 to 12.13]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p = 0.0006, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.11, 95% CI 2-sided [2.31 to 21.90]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.2073, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.72 to 4.47]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0096, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.54, 95% CI 2-sided [1.36 to 9.20]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0462, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.52, 95% CI 2-sided [1.02 to 6.27]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.1387, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.77 to 6.63]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.3130, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.60 to 4.84]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0392, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.32, 95% CI 2-sided [1.06 to 10.40]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0135, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.70, 95% CI 2-sided [1.43 to 22.71]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0840, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.85, 95% CI 2-sided [0.87 to 9.36]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0163, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.47, 95% CI 2-sided [1.32 to 15.17]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.5056, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.52 to 3.84]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.3358, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.69, 95% CI 2-sided [0.58 to 4.90]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0696, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.05, 95% CI 2-sided [0.91 to 10.18]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0794, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.80, 95% CI 2-sided [0.89 to 8.82]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0149, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.32, 95% CI 2-sided [1.48 to 36.28]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0377, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.37, 95% CI 2-sided [1.09 to 17.59]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0454, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.32, 95% CI 2-sided [1.03 to 10.77]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0390, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.77, 95% CI 2-sided [1.07 to 13.26]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.1947, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.12, 95% CI 2-sided [0.68 to 6.64]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.2913, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.61 to 5.25]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.1665, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.21, 95% CI 2-sided [0.72 to 6.82]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0157, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 13.41, 95% CI 2-sided [1.63 to 110.3]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0846, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.01, 95% CI 2-sided [0.86 to 10.49]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0171, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.42, 95% CI 2-sided [1.35 to 21.75]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0262, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.71, 95% CI 2-sided [1.20 to 18.49]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.2858, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.59 to 5.95]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0155, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.65, 95% CI 2-sided [1.47 to 39.72]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.1249, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.66, 95% CI 2-sided [0.76 to 9.31]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0616, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.85, 95% CI 2-sided [0.94 to 15.82]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0126, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.32, 95% CI 2-sided [1.58 to 43.90]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0853, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.10, 95% CI 2-sided [0.85 to 11.23]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.1562, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.56, 95% CI 2-sided [0.70 to 9.35]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.1297, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.83, 95% CI 2-sided [0.74 to 10.91]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.2001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.64 to 8.55]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0495, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.60, 95% CI 2-sided [1.00 to 73.70]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.1553, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.86, 95% CI 2-sided [0.67 to 12.20]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0199, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.67, 95% CI 2-sided [1.38 to 42.67]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0472, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.28, 95% CI 2-sided [1.02 to 27.34]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.3736, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.51 to 5.98]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.2628, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.58 to 7.26]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.1998, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.43, 95% CI 2-sided [0.63 to 9.39]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.1507, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.89, 95% CI 2-sided [0.68 to 12.28]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0385, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.92, 95% CI 2-sided [1.10 to 31.94]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0299, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.85, 95% CI 2-sided [1.26 to 93.28]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.8034, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.30 to 4.74]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.8532, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.29 to 4.42]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.8823, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.28 to 4.41]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.1651, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.79, 95% CI 2-sided [0.52 to 43.76]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.1048, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.36, 95% CI 2-sided [0.68 to 59.55]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.1168, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.87, 95% CI 2-sided [0.64 to 53.53]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.6936, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.35 to 4.95]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.4315, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.74, 95% CI 2-sided [0.44 to 6.90]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.7936, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.31 to 4.53]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0990, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.30, 95% CI 2-sided [0.71 to 56.03]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.1128, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.86, 95% CI 2-sided [0.66 to 52.21]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.0732, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.36, 95% CI 2-sided [0.83 to 65.38]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.6559, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.33 to 5.91]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.7333, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.21 to 2.96]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.9266, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.24 to 3.74]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.1518, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.04, 95% CI 2-sided [0.55 to 46.13]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.1714, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.69, 95% CI 2-sided [0.51 to 42.91]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.1299, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.60, 95% CI 2-sided [0.60 to 51.95]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.2495, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.75, 95% CI 2-sided [0.49 to 15.44]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.7065, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.31 to 5.60]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.7504, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.30 to 5.24]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.7862, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.21 to 3.29]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.1550, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.98, 95% CI 2-sided [0.54 to 45.59]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.1706, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.70, 95% CI 2-sided [0.51 to 42.96]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.1415, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.31, 95% CI 2-sided [0.57 to 49.11]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.1241, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.67, 95% CI 2-sided [0.62 to 51.74]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.2169, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.64, 95% CI 2-sided [0.57 to 12.29]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.9982, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.28 to 3.60]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.5364, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.38 to 6.54]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.1210, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.68, 95% CI 2-sided [0.63 to 51.07]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0726, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.65, 95% CI 2-sided [0.83 to 70.58]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0749, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.34, 95% CI 2-sided [0.82 to 65.81]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.0530, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.01, 95% CI 2-sided [0.98 to 16.35]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.2134, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.32, 95% CI 2-sided [0.62 to 8.72]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.3688, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.48 to 7.41]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.0563, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.61, 95% CI 2-sided [0.96 to 22.11]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.0935, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.94, 95% CI 2-sided [0.79 to 19.52]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.0901, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.71, 95% CI 2-sided [0.81 to 16.93]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.1366, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.84, 95% CI 2-sided [0.72 to 11.26]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.7876, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.34 to 4.08]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.4658, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.45 to 5.59]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.8707, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.25 to 3.20]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.3584, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.89, 95% CI 2-sided [0.49 to 7.36]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.1455, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.13, 95% CI 2-sided [0.67 to 14.57]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.0661, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.07, 95% CI 2-sided [0.90 to 28.66]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.3034, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.54 to 7.17]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.9901, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.28 to 3.60]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.5070, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.42 to 5.68]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.7927, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.21 to 3.26]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.4426, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.44 to 6.69]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.8925, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.23 to 3.56]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.4285, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.42 to 7.52]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.9000, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.31 to 3.72]

26. Secondary Outcome: Number of Participants With Absolute Reduction of 3 in Mean Number of Moderate and Severe VMS Per Day From Baseline to Each Study Week
Description: as for outcome 1
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 15 | 25 | 30 | 30 | 33 | 23 | 33 | 28
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 22 | 33 | 32 | 35 | 34 | 32 | 35 | 30
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 25 | 32 | 31 | 34 | 35 | 33 | 37 | 33
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 26 | 32 | 32 | 33 | 35 | 33 | 37 | 34
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 31 | 34 | 36 | 31 | 34 | 36 | 37 | 33
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 30 | 33 | 33 | 30 | 33 | 33 | 36 | 37
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 31 | 32 | 33 | 29 | 33 | 32 | 34 | 37
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 32 | 33 | 33 | 31 | 31 | 33 | 35 | 32
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 30 | 32 | 33 | 31 | 33 | 33 | 34 | 34
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 28 | 33 | 30 | 28 | 33 | 34 | 36 | 34
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 30 | 32 | 31 | 26 | 32 | 34 | 36 | 33
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 28 | 32 | 31 | 26 | 31 | 31 | 34 | 33
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 16 | 25 | 22 | 20 | 21 | 22 | 21 | 26
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 15 | 21 | 21 | 14 | 18 | 19 | 19 | 22
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 18 | 17 | 18 | 12 | 15 | 13 | 16 | 17
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0602, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.96 to 6.06]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0010, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.88, 95% CI 2-sided [1.89 to 12.57]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p = 0.0006, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.24, 95% CI 2-sided [2.03 to 13.51]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.07, 95% CI 2-sided [3.23 to 25.45]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.1259, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.82 to 5.22]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.05, 95% CI 2-sided [2.65 to 18.71]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0070, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.51, 95% CI 2-sided [1.41 to 8.76]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0193, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.15, 95% CI 2-sided [1.20 to 8.23]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0148, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.34, 95% CI 2-sided [1.27 to 8.81]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0018, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.05, 95% CI 2-sided [1.83 to 13.94]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0007, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.27, 95% CI 2-sided [2.32 to 22.78]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0246, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.11, 95% CI 2-sided [1.16 to 8.35]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0016, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.22, 95% CI 2-sided [1.87 to 14.60]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0825, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.90 to 5.62]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0542, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.66, 95% CI 2-sided [0.98 to 7.20]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0837, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.38, 95% CI 2-sided [0.89 to 6.33]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0131, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.67, 95% CI 2-sided [1.31 to 10.26]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0012, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.34, 95% CI 2-sided [2.41 to 36.19]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0359, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.10, 95% CI 2-sided [1.08 to 8.93]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0019, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.86, 95% CI 2-sided [1.91 to 17.92]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0715, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.43, 95% CI 2-sided [0.93 to 6.38]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0465, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.89, 95% CI 2-sided [1.02 to 8.20]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0839, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.89 to 6.53]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0191, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.56, 95% CI 2-sided [1.23 to 10.28]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0019, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 12.11, 95% CI 2-sided [2.52 to 58.22]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0593, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.76, 95% CI 2-sided [0.96 to 7.90]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0048, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.95, 95% CI 2-sided [1.63 to 15.04]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0494, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.75, 95% CI 2-sided [1.00 to 7.57]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.1887, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.15, 95% CI 2-sided [0.69 to 6.70]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.0717, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.06, 95% CI 2-sided [0.91 to 10.7]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.1419, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.43, 95% CI 2-sided [0.74 to 7.92]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority — 0.0141; p = 0.0141, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 14.37, 95% CI 2-sided [1.71 to 120.6]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0775, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.19, 95% CI 2-sided [0.88 to 11.54]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0283, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.35, 95% CI 2-sided [1.17 to 16.19]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.1767, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.21, 95% CI 2-sided [0.70 to 6.96]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.1675, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.72 to 6.72]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.2717, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.62 to 5.49]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.1367, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.40, 95% CI 2-sided [0.76 to 7.64]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0162, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 13.53, 95% CI 2-sided [1.62 to 113.0]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.0765, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.23, 95% CI 2-sided [0.88 to 11.78]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0061, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.80, 95% CI 2-sided [1.79 to 33.87]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0181, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.40, 95% CI 2-sided [1.33 to 21.85]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.3925, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.53 to 4.99]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.3740, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.54 to 5.12]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.1753, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.33, 95% CI 2-sided [0.69 to 7.93]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0195, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 12.85, 95% CI 2-sided [1.51 to 109.5]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.1932, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.66 to 8.02]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0537, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.55, 95% CI 2-sided [0.98 to 12.86]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0144, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.72, 95% CI 2-sided [1.50 to 39.66]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.6660, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.41 to 4.09]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.7923, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.37 to 3.62]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.3796, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.51 to 5.90]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0874, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.20, 95% CI 2-sided [0.81 to 21.73]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.1925, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.60, 95% CI 2-sided [0.62 to 10.96]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0651, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.99, 95% CI 2-sided [0.92 to 17.38]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.5361, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.44 to 4.81]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.6258, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.42 to 4.17]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.6275, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.43 to 4.06]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.2212, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.21, 95% CI 2-sided [0.62 to 7.90]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0280, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 11.13, 95% CI 2-sided [1.30 to 95.49]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.0589, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.88, 95% CI 2-sided [0.94 to 25.32]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0799, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.63, 95% CI 2-sided [0.86 to 15.39]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.1112, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.91, 95% CI 2-sided [0.78 to 10.87]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.0959, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.76, 95% CI 2-sided [0.84 to 9.11]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.3886, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.54 to 4.85]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0864, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.00, 95% CI 2-sided [0.85 to 10.52]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0145, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 14.22, 95% CI 2-sided [1.69 to 119.5]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.0180, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 13.08, 95% CI 2-sided [1.56 to 110.0]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0080, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 18.53, 95% CI 2-sided [2.14 to 160.6]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0236, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.07, 95% CI 2-sided [1.24 to 20.65]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.4303, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.59, 0.4303% CI 2-sided [0.50 to 5.07]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.5529, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.45 to 4.39]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.3268, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.87, 95% CI 2-sided [0.53 to 6.55]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0343, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.02, 95% CI 2-sided [1.19 to 84.66]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0391, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.45, 95% CI 2-sided [1.12 to 79.82]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0187, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 13.31, 95% CI 2-sided [1.54 to 115.1]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.1475, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.60, 95% CI 2-sided [0.71 to 9.47]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.2161, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.19, 95% CI 2-sided [0.63 to 7.55]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.3478, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.53 to 6.04]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.2269, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.61 to 8.14]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.0683, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.66, 95% CI 2-sided [0.89 to 24.35]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0228, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.11, 95% CI 2-sided [1.31 to 38.49]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0620, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.95, 95% CI 2-sided [0.93 to 16.72]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.2251, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.18, 95% CI 2-sided [0.62 to 7.67]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.7908, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.35 to 3.99]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.3735, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.48 to 7.06]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.1856, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.49, 95% CI 2-sided [0.64 to 9.64]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.01798, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.67, 95% CI 2-sided [0.64 to 11.20]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.1101, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.19, 95% CI 2-sided [0.77 to 13.22]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.1060, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.99, 95% CI 2-sided [0.79 to 11.31]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.5258, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.45 to 4.86]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.8746, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.34 to 3.50]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.7434, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.24 to 2.77]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.3211, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.90, 95% CI 2-sided [0.53 to 6.80]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.5330, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.41 to 5.48]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.1119, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.00, 95% CI 2-sided [0.77 to 11.64]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.3540, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.53 to 5.85]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.5076, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.19 to 2.29]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.5801, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.21 to 2.41]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.2785, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.13 to 1.82]
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.5656, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.19 to 2.45]
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.6445, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.19 to 2.81]
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.7363, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.32 to 4.99]
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.3455, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.17 to 1.86]

27. Secondary Outcome: Number of Participants With Absolute Reduction of 4 in Mean Number of Moderate and Severe VMS Per Day From Baseline to Each Study Week
Description: as for outcome 1
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 11 | 25 | 23 | 26 | 26 | 19 | 26 | 27
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 16 | 30 | 29 | 32 | 32 | 26 | 29 | 26
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 20 | 31 | 29 | 31 | 33 | 28 | 36 | 31
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 23 | 28 | 29 | 29 | 31 | 31 | 33 | 30
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 27 | 29 | 31 | 28 | 34 | 33 | 35 | 31
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 28 | 31 | 29 | 29 | 31 | 30 | 34 | 32
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 28 | 31 | 32 | 28 | 32 | 30 | 32 | 31
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 29 | 33 | 32 | 30 | 30 | 31 | 34 | 30
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 28 | 31 | 30 | 31 | 33 | 31 | 34 | 32
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 27 | 31 | 27 | 26 | 31 | 32 | 35 | 31
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 27 | 31 | 28 | 24 | 31 | 33 | 35 | 30
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 25 | 29 | 28 | 25 | 29 | 29 | 31 | 31
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 13 | 23 | 18 | 17 | 19 | 20 | 18 | 21
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 14 | 19 | 16 | 11 | 16 | 18 | 15 | 17
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 15 | 15 | 12 | 10 | 14 | 13 | 11 | 13
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0037, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.30, 95% CI 2-sided [1.60 to 11.54]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0057, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.95, 95% CI 2-sided [1.49 to 10.48]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.03, 95% CI 2-sided [2.26 to 16.13]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.42, 95% CI 2-sided [2.37 to 17.39]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.1410, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.11, 95% CI 2-sided [0.78 to 5.73]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0004, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.85, 95% CI 2-sided [2.20 to 15.55]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0006, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.50, 95% CI 2-sided [2.08 to 14.54]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0037, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.09, 95% CI 2-sided [1.58 to 10.57]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0026, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.31, 95% CI 2-sided [1.67 to 11.16]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.26, 95% CI 2-sided [2.63 to 16.60]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.40, 95% CI 2-sided [3.23 to 27.34]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0431, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.03 to 6.76]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0020, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.40, 95% CI 2-sided [1.72 to 11.29]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0291, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.76, 95% CI 2-sided [1.11 to 6.86]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0063, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.96, 95% CI 2-sided [1.48 to 10.61]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0202, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.11, 95% CI 2-sided [1.19 to 8.11]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0044, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.10, 95% CI 2-sided [1.55 to 10.84]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.21, 95% CI 2-sided [2.89 to 29.38]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0706, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.43, 95% CI 2-sided [0.93 to 6.37]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.20, 95% CI 2-sided [2.79 to 24.08]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0146, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.24, 95% CI 2-sided [1.26 to 8.32]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0816, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.90 to 6.24]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0930, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.87 to 5.81]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.365, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.81, 95% CI 2-sided [1.07 to 7.39]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0042, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.93, 95% CI 2-sided [1.65 to 14.73]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.0488, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.73, 95% CI 2-sided [1.01 to 7.41]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0075, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.85, 95% CI 2-sided [1.43 to 10.36]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0984, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.86 to 5.59]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.2226, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.89, 95% CI 2-sided [0.68 to 5.29]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.1467, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.16, 95% CI 2-sided [0.76 to 6.08]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0705, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.74, 95% CI 2-sided [0.92 to 8.19]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p = 0.0025, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 26.62, 95% CI 2-sided [3.16 to 223.9]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.0757, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.75, 95% CI 2-sided [0.90 to 8.40]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0045, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.66, 95% CI 2-sided [1.71 to 18.74]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.0771, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.63, 95% CI 2-sided [0.90 to 7.67]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.1856, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.71 to 5.81]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.5973, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.48 to 3.54]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0935, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.57, 95% CI 2-sided [0.85 to 7.77]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0157, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.52, 95% CI 2-sided [1.38 to 22.10]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.1963, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.68 to 6.32]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0085, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.31, 95% CI 2-sided [1.53 to 18.43]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.1433, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.21, 95% CI 2-sided [0.76 to 6.38]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.1577, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.17, 95% CI 2-sided [0.74 to 6.37]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.1608, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.16, 95% CI 2-sided [0.74 to 6.34]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0693, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.96, 95% CI 2-sided [0.92 to 9.53]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0063, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.57, 95% CI 2-sided [1.89 to 48.39]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.1637, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.72 to 7.05]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0326, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.57, 95% CI 2-sided [1.11 to 11.47]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.1455, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.24, 95% CI 2-sided [0.76 to 6.67]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.1951, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.69 to 6.32]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.4097, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.54 to 4.53]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.1554, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.73 to 7.22]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0440, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.22, 95% CI 2-sided [1.04 to 17.14]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.1928, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.23, 95% CI 2-sided [0.67 to 7.47]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0222, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.67, 95% CI 2-sided [1.25 to 17.47]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.4075, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.54 to 4.65]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.3659, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.56 to 4.93]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.7878, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.41 to 3.24]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.0635, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.26, 95% CI 2-sided [0.94 to 11.38]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0137, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 14.62, 95% CI 2-sided [1.73 to 123.3]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.1069, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.91, 95% CI 2-sided [0.79 to 10.62]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0186, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.60, 95% CI 2-sided [1.33 to 23.47]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.1434, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.75 to 7.56]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.1670, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.20, 95% CI 2-sided [0.72 to 6.75]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.7810, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.41 to 3.28]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.1682, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.27, 95% CI 2-sided [0.71 to 7.26]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0215, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.22, 95% CI 2-sided [1.28 to 21.39]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.0306, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.75, 95% CI 2-sided [1.16 to 19.52]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0059, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.10, 95% CI 2-sided [1.92 to 52.29]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.1004, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.64, 95% CI 2-sided [0.83 to 8.43]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.1837, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.11, 95% CI 2-sided [0.70 to 6.36]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.5929, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.47 to 3.75]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.2588, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.62 to 6.07]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0129, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.69, 95% CI 2-sided [1.54 to 38.41]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0168, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.12, 95% CI 2-sided [1.42 to 35.61]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0058, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 9.95, 95% CI 2-sided [1.94 to 50.97]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.1934, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.08, 95% CI 2-sided [0.69 to 6.26]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.2181, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.66 to 6.12]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.4116, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.53 to 4.71]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0938, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.84, 95% CI 2-sided [0.84 to 9.66]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0125, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.02, 95% CI 2-sided [1.57 to 41.08]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.0761, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.29, 95% CI 2-sided [0.88 to 12.23]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0305, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.02, 95% CI 2-sided [1.14 to 14.16]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0501, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.42, 95% CI 2-sided [1.00 to 11.68]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.1212, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.61, 95% CI 2-sided [0.78 to 8.77]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.8332, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.35 to 3.68]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.4285, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.66, 95% CI 2-sided [0.48 to 5.76]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.0954, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.98, 95% CI 2-sided [0.83 to 10.74]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.1110, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.98, 95% CI 2-sided [0.78 to 11.38]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.1642, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.44, 95% CI 2-sided [0.69 to 8.55]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.1976, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.19, 95% CI 2-sided [0.66 to 7.24]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.5761, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.43 to 4.58]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.4540, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.20 to 2.04]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.3732, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.17 to 1.96]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.4665, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.46 to 5.50]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.5634, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.41 to 5.25]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.4297, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.48 to 5.70]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.9789, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.31 to 3.14]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.7357, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.24 to 2.70]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.1977, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.14 to 1.50]
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.3203, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.14 to 1.88]
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.9739, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.30 to 3.44]
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.6714, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.36 to 4.97]
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.6375, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.22 to 2.52]
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.2980, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.17 to 1.71]

28. Secondary Outcome: Number of Participants With Absolute Reduction of 5 in Mean Number of Moderate and Severe VMS Per Day From Baseline to Each Study Week
Description: as for outcome 1
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14 and 15
Population: FAS population with available data at specified time point.
Measure: Number; unit: participants
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 45 | 43 | 43 | 41 | 41 | 44 | 44
participants
  Week 1 | 6 | 19 | 22 | 23 | 22 | 14 | 17 | 22
  Week 2: number analyzed (Participants) | 42 | 44 | 42 | 43 | 39 | 41 | 43 | 43
  Week 2 | 14 | 25 | 27 | 27 | 25 | 24 | 27 | 24
  Week 3: number analyzed (Participants) | 42 | 42 | 41 | 42 | 38 | 40 | 43 | 43
  Week 3 | 16 | 25 | 27 | 28 | 28 | 25 | 31 | 25
  Week 4: number analyzed (Participants) | 42 | 40 | 41 | 40 | 37 | 40 | 43 | 42
  Week 4 | 19 | 24 | 28 | 26 | 29 | 25 | 31 | 26
  Week 5: number analyzed (Participants) | 42 | 41 | 41 | 37 | 35 | 40 | 41 | 39
  Week 5 | 23 | 25 | 28 | 26 | 28 | 29 | 33 | 27
  Week 6: number analyzed (Participants) | 41 | 41 | 41 | 37 | 34 | 37 | 39 | 40
  Week 6 | 23 | 26 | 28 | 27 | 28 | 27 | 31 | 29
  Week 7: number analyzed (Participants) | 41 | 41 | 41 | 35 | 34 | 37 | 39 | 39
  Week 7 | 23 | 29 | 29 | 25 | 29 | 27 | 31 | 29
  Week 8: number analyzed (Participants) | 40 | 41 | 41 | 37 | 33 | 36 | 38 | 38
  Week 8 | 25 | 26 | 28 | 26 | 26 | 27 | 31 | 29
  Week 9: number analyzed (Participants) | 39 | 40 | 41 | 36 | 34 | 35 | 37 | 38
  Week 9 | 24 | 27 | 29 | 26 | 29 | 27 | 32 | 29
  Week 10: number analyzed (Participants) | 39 | 39 | 38 | 33 | 34 | 35 | 37 | 37
  Week 10 | 22 | 27 | 26 | 24 | 29 | 29 | 32 | 29
  Week 11: number analyzed (Participants) | 39 | 39 | 38 | 31 | 33 | 35 | 37 | 37
  Week 11 | 24 | 29 | 27 | 23 | 27 | 30 | 31 | 30
  Week 12: number analyzed (Participants) | 37 | 38 | 37 | 31 | 31 | 33 | 36 | 36
  Week 12 | 23 | 25 | 27 | 21 | 26 | 27 | 31 | 28
  Week 13: number analyzed (Participants) | 24 | 34 | 33 | 27 | 27 | 27 | 26 | 32
  Week 13 | 9 | 20 | 15 | 13 | 14 | 20 | 13 | 16
  Week 14: number analyzed (Participants) | 24 | 32 | 33 | 25 | 25 | 26 | 24 | 31
  Week 14 | 10 | 17 | 13 | 9 | 10 | 17 | 12 | 13
  Week 15: number analyzed (Participants) | 25 | 27 | 28 | 20 | 24 | 20 | 21 | 29
  Week 15 | 9 | 12 | 10 | 8 | 7 | 11 | 10 | 12
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 1; Test type: Superiority; p = 0.0044, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.35, 95% CI 2-sided [1.69 to 16.96]
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 1; Test type: Superiority; p = 0.0002, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 8.65, 95% CI 2-sided [2.79 to 26.83]
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.82, 95% CI 2-sided [3.49 to 33.54]
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 1; Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 10.01, 95% CI 2-sided [3.20 to 31.29]
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 1; Test type: Superiority; p = 0.1266, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.51, 95% CI 2-sided [0.77 to 8.15]
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 1; Test type: Superiority; p = 0.0024, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.72, 95% CI 2-sided [1.85 to 17.66]
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 1; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.93, 95% CI 2-sided [2.59 to 24.26]
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 2; Test type: Superiority; p = 0.0217, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.11, 95% CI 2-sided [1.18 to 8.17]
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 2; Test type: Superiority; p = 0.0021, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.63, 95% CI 2-sided [1.75 to 12.25]
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 2; Test type: Superiority; p = 0.0016, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.72, 95% CI 2-sided [1.80 to 12.37]
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 2; Test type: Superiority; p = 0.0018, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.80, 95% CI 2-sided [1.79 to 12.86]
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 2; Test type: Superiority; p = 0.0467, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.69, 95% CI 2-sided [1.01 to 7.14]
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 2; Test type: Superiority; p = 0.0016, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.70, 95% CI 2-sided [1.80 to 12.28]
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 2; Test type: Superiority; p = 0.0234, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.98, 95% CI 2-sided [1.16 to 7.65]
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 3; Test type: Superiority; p = 0.0294, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.88, 95% CI 2-sided [1.11 to 7.46]
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 3; Test type: Superiority; p = 0.0068, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.74, 95% CI 2-sided [1.44 to 9.73]
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 3; Test type: Superiority; p = 0.0025, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.35, 95% CI 2-sided [1.68 to 11.29]
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 3; Test type: Superiority; p = 0.0006, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.82, 95% CI 2-sided [2.13 to 15.92]
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 3; Test type: Superiority; p = 0.0572, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.53, 95% CI 2-sided [0.97 to 6.61]
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 3; Test type: Superiority; p = 0.0003, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.03, 95% CI 2-sided [2.28 to 15.97]
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 3; Test type: Superiority; p = 0.0460, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.55, 95% CI 2-sided [1.02 to 6.38]
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.1406, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.79 to 5.23]
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0234, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.97, 95% CI 2-sided [1.16 to 7.63]
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0302, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.82, 95% CI 2-sided [1.10 to 7.22]
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0016, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.23, 95% CI 2-sided [1.87 to 14.63]
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.2105, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.71 to 4.64]
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0033, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.17, 95% CI 2-sided [1.61 to 10.81]
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.1087, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.10, 95% CI 2-sided [0.85 to 5.21]
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 5; Test type: Superiority; p = 0.3600, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.60 to 4.03]
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 5; Test type: Superiority; p = 0.1394, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.05, 95% CI 2-sided [0.79 to 5.32]
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 5; Test type: Superiority; p = 0.0522, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.70, 95% CI 2-sided [0.99 to 7.36]
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 5; Test type: Superiority; p = 0.0119, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.97, 95% CI 2-sided [1.63 to 11.61]
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 5; Test type: Superiority; p = 0.1474, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.77 to 5.53]
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 5; Test type: Superiority; p = 0.0026, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.08, 95% CI 2-sided [1.76 to 14.67]
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 5; Test type: Superiority; p = 0.1263, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.11, 95% CI 2-sided [0.81 to 5.51]
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 6; Test type: Superiority; p = 0.2327, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.68 to 4.95]
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 6; Test type: Superiority; p = 0.1359, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.12, 95% CI 2-sided [0.79 to 5.70]
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 6; Test type: Superiority; p = 0.0258, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.35, 95% CI 2-sided [1.16 to 9.69]
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 6; Test type: Superiority; p = 0.0076, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.77, 95% CI 2-sided [1.51 to 15.04]
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 6; Test type: Superiority; p = 0.1088, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.36, 95% CI 2-sided [0.83 to 6.75]
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 6; Test type: Superiority; p = 0.0045, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.89, 95% CI 2-sided [1.64 to 14.62]
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 6; Test type: Superiority; p = 0.0493, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.74, 95% CI 2-sided [1.00 to 7.50]
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 7; Test type: Superiority; p = 0.0376, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.99, 95% CI 2-sided [1.06 to 8.41]
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 7; Test type: Superiority; p = 0.0723, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.53, 95% CI 2-sided [0.92 to 6.94]
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 7; Test type: Superiority; p = 0.0396, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.11, 95% CI 2-sided [1.06 to 9.17]
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 7; Test type: Superiority; p = 0.0031, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 6.18, 95% CI 2-sided [1.85 to 20.67]
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 7; Test type: Superiority; p = 0.1044, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.41, 95% CI 2-sided [0.83 to 6.96]
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 7; Test type: Superiority; p = 0.0029, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.47, 95% CI 2-sided [1.78 to 16.75]
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 7; Test type: Superiority; p = 0.0364, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.01, 95% CI 2-sided [1.07 to 8.45]
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.6396, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.47 to 3.37]
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.4378, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.55 to 3.91]
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.2045, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.70 to 5.44]
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0958, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.54, 95% CI 2-sided [0.85 to 7.62]
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.3210, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.70, 95% CI 2-sided [0.60 to 4.85]
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.0199, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.75, 95% CI 2-sided [1.23 to 11.39]
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.1219, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.26, 95% CI 2-sided [0.80 to 6.36]
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 9; Test type: Superiority; p = 0.2975, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.62 to 4.76]
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 9; Test type: Superiority; p = 0.2763, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.64 to 4.80]
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 9; Test type: Superiority; p = 0.1235, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.33, 95% CI 2-sided [0.79 to 6.82]
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 9; Test type: Superiority; p = 0.0190, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.24, 95% CI 2-sided [1.27 to 14.19]
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 9; Test type: Superiority; p = 0.2213, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.98, 95% CI 2-sided [0.66 to 5.93]
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 9; Test type: Superiority; p = 0.0050, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.88, 95% CI 2-sided [1.71 to 20.25]
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 9; Test type: Superiority; p = 0.1053, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.39, 95% CI 2-sided [0.83 to 6.85]
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 10; Test type: Superiority; p = 0.0991, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.39, 95% CI 2-sided [0.85 to 6.72]
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 10; Test type: Superiority; p = 0.2056, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.70 to 5.32]
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 10; Test type: Superiority; p = 0.0407, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.17, 95% CI 2-sided [1.05 to 9.57]
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 10; Test type: Superiority; p = 0.0059, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.47, 95% CI 2-sided [1.63 to 18.30]
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 10; Test type: Superiority; p = 0.0230, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.85, 95% CI 2-sided [1.20 to 12.30]
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 10; Test type: Superiority; p = 0.0015, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.36, 95% CI 2-sided [2.14 to 25.29]
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 10; Test type: Superiority; p = 0.0248, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.45, 95% CI 2-sided [1.17 to 10.16]
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 11; Test type: Superiority; p = 0.1091, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.82 to 6.83]
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 11; Test type: Superiority; p = 0.3054, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.61 to 4.75]
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 11; Test type: Superiority; p = 0.1129, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.48, 95% CI 2-sided [0.81 to 7.61]
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 11; Test type: Superiority; p = 0.0432, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.28, 95% CI 2-sided [1.04 to 10.37]
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 11; Test type: Superiority; p = 0.0315, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.77, 95% CI 2-sided [1.13 to 12.60]
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 11; Test type: Superiority; p = 0.0147, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 4.26, 95% CI 2-sided [1.33 to 13.64]
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 11; Test type: Superiority; p = 0.0405, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.18, 95% CI 2-sided [1.05 to 9.59]
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.5238, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.50 to 3.93]
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.3060, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.60 to 4.97]
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.3747, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.55 to 4.86]
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0443, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.49, 95% CI 2-sided [1.03 to 11.80]
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.1269, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.49, 95% CI 2-sided [0.77 to 8.06]
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.0095, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 5.15, 95% CI 2-sided [1.49 to 17.13]
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.1254, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.79 to 6.94]
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 13; Test type: Superiority; p = 0.0402, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 3.66, 95% CI 2-sided [1.06 to 12.63]
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 13; Test type: Superiority; p = 0.4547, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.47 to 5.42]
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 13; Test type: Superiority; p = 0.4008, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.49 to 5.99]
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 13; Test type: Superiority; p = 0.1535, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.55, 95% CI 2-sided [0.71 to 9.22]
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 13; Test type: Superiority; p = 0.0055, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 7.19, 95% CI 2-sided [1.79 to 28.95]
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 13; Test type: Superiority; p = 0.2116, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.19, 95% CI 2-sided [0.64 to 7.50]
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 13; Test type: Superiority; p = 0.1668, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.70 to 7.83]
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 14; Test type: Superiority; p = 0.1824, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.32, 95% CI 2-sided [0.67 to 7.98]
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 14; Test type: Superiority; p = 0.7970, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.25 to 2.90]
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 14; Test type: Superiority; p = 0.7065, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.21 to 2.85]
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 14; Test type: Superiority; p = 0.9126, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.29 to 3.93]
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 14; Test type: Superiority; p = 0.1282, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.82, 95% CI 2-sided [0.74 to 10.70]
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 14; Test type: Superiority; p = 0.2661, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.58 to 7.04]
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 14; Test type: Superiority; p = 0.7457, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.36 to 4.09]
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.4095, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.47 to 6.41]
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.9571, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.28 to 3.77]
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.8827, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.23 to 3.59]
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.5944, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.17 to 2.74]
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.1647, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.74, 95% CI 2-sided [0.66 to 11.39]
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.2684, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.57 to 7.48]
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.5338, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.43 to 5.07]

29. Secondary Outcome: Change From Baseline in Hot Flash-Related Daily Interference Scale (HFRDIS) at Weeks 4, 8, 12, and 15
Description: The HFRDIS is a 10-item scale that measures a woman's perceptions of the degree to which VMS interfere with 9 daily life activities (work, social activities, leisure, sleep, mood, concentration, relations with others, sexuality, and enjoying life); the tenth item measures interference with overall quality of life. This scale was modeled after items on the Brief Pain Inventory and Brief Fatigue Inventory, which assess the extent to which pain or fatigue interfere with daily life. Participants were asked to rate the extent to which VMS had interfered with each item during the previous 2-week time interval using a 0 (do not interfere) to 10 (completely interfere) scale. Overall mean score is the average of individual item scores (sum of items/10).
Time Frame: Baseline and weeks 4, 8, 12, and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 42 | 41 | 41 | 38 | 39 | 43 | 40
Score on a scale
  Week 4 | -2.2 (0.34) | -3.3 (0.32) | -3.6 (0.33) | -3.8 (0.33) | -3.7 (0.35) | -2.5 (0.35) | -3.4 (0.32) | -3.5 (0.34)
  Week 8: number analyzed (Participants) | 41 | 40 | 41 | 36 | 36 | 37 | 39 | 40
  Week 8 | -2.7 (0.34) | -3.3 (0.33) | -3.6 (0.34) | -4.1 (0.35) | -4.2 (0.36) | -3.0 (0.36) | -3.3 (0.33) | -3.6 (0.35)
  Week 12: number analyzed (Participants) | 36 | 40 | 33 | 30 | 29 | 28 | 35 | 36
  Week 12 | -2.9 (0.33) | -3.6 (0.31) | -3.8 (0.33) | -4.3 (0.34) | -4.2 (0.35) | -3.3 (0.35) | -3.5 (0.32) | -3.9 (0.33)
  Week 15: number analyzed (Participants) | 37 | 40 | 38 | 35 | 34 | 33 | 37 | 37
  Week 15 | -2.4 (0.39) | -2.6 (0.37) | -2.2 (0.39) | -2.3 (0.40) | -1.9 (0.41) | -2.9 (0.42) | -2.4 (0.38) | -2.5 (0.40)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4; Test type: Superiority; p = 0.0179, Mixed model repeated measures (MMRM) — LSM, SE, CI, & p-values come from an MMRM model with CFB as dependent variable & TG, visit & smoking status as factors and baseline measurement as a covariate, as well as interaction of treatment by week & interaction of baseline measurement by week; LSMean difference = -1.1, 95% CI 2-sided [-1.95 to -0.18], Standard Error of Mean 0.45
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4; Test type: Superiority; p = 0.0027, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-2.25 to -0.47], Standard Error of Mean 0.45
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-2.50 to -0.73], Standard Error of Mean 0.45
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4; Test type: Superiority; p = 0.0009, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-2.43 to -0.64], Standard Error of Mean 0.46
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4; Test type: Superiority; p = 0.5806, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-1.14 to 0.64], Standard Error of Mean 0.45
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4; Test type: Superiority; p = 0.0105, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -1.2, 95% CI 2-sided [-2.03 to -0.27], Standard Error of Mean 0.45
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4; Test type: Superiority; p = 0.0048, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -1.3, 95% CI 2-sided [-2.16 to -0.39], Standard Error of Mean 0.45
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8; Test type: Superiority; p = 0.1801, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.52 to 0.29], Standard Error of Mean 0.46
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8; Test type: Superiority; p = 0.0609, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.76 to 0.04], Standard Error of Mean 0.46
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8; Test type: Superiority; p = 0.0028, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-2.33 to -0.49], Standard Error of Mean 0.47
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8; Test type: Superiority; p = 0.0018, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-2.40 to -0.55], Standard Error of Mean 0.47
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8; Test type: Superiority; p = 0.5519, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-1.19 to 0.64], Standard Error of Mean 0.46
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8; Test type: Superiority; p = 0.1922, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.51 to 0.31], Standard Error of Mean 0.46
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8; Test type: Superiority; p = 0.0463, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.82 to -0.02], Standard Error of Mean 0.46
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12; Test type: Superiority; p = 0.1288, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.53 to 0.19], Standard Error of Mean 0.44
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12; Test type: Superiority; p = 0.0577, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.72 to 0.03], Standard Error of Mean 0.44
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12; Test type: Superiority; p = 0.0027, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-2.26 to -0.48], Standard Error of Mean 0.45
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12; Test type: Superiority; p = 0.0043, MMRM — [p-value comment as in outcome 29, analysis 1]; -1.3 = -1.3, 95% CI 2-sided [-2.20 to -0.41], Standard Error of Mean 0.45
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12; Test type: Superiority; p = 0.4089, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-1.27 to 0.52], Standard Error of Mean 0.45
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12; Test type: Superiority; p = 0.2050, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.44 to 0.31], Standard Error of Mean 0.44
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12; Test type: Superiority; p = 0.0265, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.84 to -0.11], Standard Error of Mean 0.44
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15; Test type: Superiority; p = 0.7617, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-1.20 to 0.88], Standard Error of Mean 0.53
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15; Test type: Superiority; p = 0.6061, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = 0.3, 95% CI 2-sided [-0.77 to 1.32], Standard Error of Mean 0.53
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15; Test type: Superiority; p = 0.7997, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = 0.1, 95% CI 2-sided [-0.93 to 1.21], Standard Error of Mean 0.54
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15; Test type: Superiority; p = 0.3391, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = 0.5, 95% CI 2-sided [-0.55 to 1.60], Standard Error of Mean 0.55
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15; Test type: Superiority; p = 0.3934, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-1.55 to 0.61], Standard Error of Mean 0.55
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15; Test type: Superiority; p = 0.9750, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.00, 95% CI 2-sided [-1.08 to 1.04], Standard Error of Mean 0.54
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15; Test type: Superiority; p = 0.8830, MMRM — [p-value comment as in outcome 29, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-1.13 to 0.97], Standard Error of Mean 0.53

30. Secondary Outcome: Leeds Sleep Evaluation Questionnaire (LSEQ) Domain Scores at Weeks 4, 8, 12 and 15
Description: The LSEQ is a 10-item self-rated questionnaire that assesses a participants aspects of sleep and early morning behavior. The questions are grouped into 4 chronological areas: ease of getting to sleep, perceived quality of sleep, ease of awaking from sleep, and integrity of early morning behavior following wakefulness. The LSEQ is a visual analog scale that requires respondents to place marks on a group of 10 cm lines. Lines extend between extremes like "more difficult than usual" and "easier than usual." Responses are measured using a 100 mm scale and are averaged to a score for each domain. Higher scores indicates better sleep and better early morning behavior.
Time Frame: Weeks 4, 8, 12, and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 40 | 41 | 38 | 38 | 38 | 43 | 40
Score on a scale
  Week 4: Ease of Getting to Sleep: number analyzed (Participants) | 42 | 40 | 40 | 38 | 38 | 38 | 43 | 39
  Week 4: Ease of Getting to Sleep | 40.7 (3.18) | 43.1 (3.06) | 44.6 (3.25) | 36.7 (3.25) | 41.7 (3.38) | 43.1 (3.35) | 40.3 (2.98) | 44.7 (3.32)
  Week 4: Quality of Sleep: number analyzed (Participants) | 42 | 40 | 40 | 38 | 38 | 38 | 43 | 39
  Week 4: Quality of Sleep | 38.7 (3.75) | 40.4 (3.64) | 36.1 (3.81) | 32.8 (3.84) | 42.0 (4.00) | 36.7 (3.98) | 38.6 (3.53) | 42.4 (3.95)
  Week 4: Ease of Awaking From Sleep: number analyzed (Participants) | 42 | 40 | 40 | 38 | 38 | 38 | 43 | 39
  Week 4: Ease of Awaking From Sleep | 43.6 (3.31) | 47.1 (3.18) | 43.9 (3.36) | 37.8 (3.38) | 41.7 (3.53) | 41.8 (3.51) | 37.5 (3.10) | 43.3 (3.48)
  Week 4: Integrity of Behavior Following Awaking: number analyzed (Participants) | 42 | 40 | 40 | 38 | 38 | 38 | 43 | 39
  Week 4: Integrity of Behavior Following Awaking | 41.2 (3.40) | 42.0 (3.23) | 41.5 (3.44) | 32.4 (3.44) | 38.0 (3.61) | 43.3 (3.58) | 41.8 (3.16) | 41.3 (3.56)
  Week 8:Ease of Getting to Sleep: number analyzed (Participants) | 41 | 39 | 41 | 35 | 35 | 36 | 39 | 40
  Week 8:Ease of Getting to Sleep | 40.3 (3.09) | 39.2 (2.96) | 41.5 (3.10) | 35.6 (3.18) | 38.3 (3.28) | 41.7 (3.24) | 43.6 (2.98) | 43.7 (3.15)
  Week 8: Quality of Sleep: number analyzed (Participants) | 41 | 39 | 41 | 35 | 35 | 36 | 39 | 40
  Week 8: Quality of Sleep | 41.1 (3.63) | 36.3 (3.52) | 39.5 (3.62) | 33.6 (3.75) | 38.6 (3.86) | 36.9 (3.83) | 37.7 (3.54) | 38.2 (3.71)
  Week 8:Ease of Awaking From Sleep: number analyzed (Participants) | 41 | 39 | 41 | 35 | 35 | 36 | 39 | 40
  Week 8:Ease of Awaking From Sleep | 40.3 (3.35) | 38.8 (3.22) | 37.5 (3.34) | 36.4 (3.46) | 41.2 (3.56) | 37.7 (3.53) | 44.3 (3.27) | 41.2 (3.43)
  Week 8: Integrity of Behavior Following Awake: number analyzed (Participants) | 41 | 39 | 41 | 35 | 35 | 36 | 39 | 40
  Week 8: Integrity of Behavior Following Awake | 40.9 (3.49) | 40.6 (3.33) | 38.8 (3.47) | 35.2 (3.56) | 41.4 (3.69) | 35.9 (3.66) | 41.3 (3.36) | 40.5 (3.55)
  Wek 12: Ease of Getting Sleep: number analyzed (Participants) | 36 | 40 | 33 | 30 | 28 | 27 | 35 | 35
  Wek 12: Ease of Getting Sleep | 32.0 (3.30) | 37.2 (3.04) | 38.9 (3.41) | 37.7 (3.44) | 39.6 (3.69) | 39.4 (3.78) | 41.6 (3.19) | 38.4 (3.39)
  Week 12: Quality of Sleep: number analyzed (Participants) | 36 | 40 | 33 | 30 | 28 | 27 | 35 | 35
  Week 12: Quality of Sleep | 36.3 (3.76) | 37.2 (3.46) | 38.4 (3.89) | 36.0 (3.92) | 34.5 (4.22) | 37.1 (4.35) | 37.6 (3.64) | 36.6 (3.88)
  Week 12: Ease of Awaking From Sleep: number analyzed (Participants) | 36 | 40 | 33 | 30 | 28 | 27 | 35 | 35
  Week 12: Ease of Awaking From Sleep | 37.3 (3.68) | 37.1 (3.41) | 35.9 (3.77) | 37.4 (3.82) | 37.8 (4.06) | 37.1 (4.15) | 41.9 (3.57) | 40.9 (3.78)
  Week 12: Integrity of Behavior Following Awaking: number analyzed (Participants) | 36 | 40 | 33 | 30 | 28 | 27 | 35 | 35
  Week 12: Integrity of Behavior Following Awaking | 35.5 (3.82) | 38.3 (3.54) | 36.6 (3.90) | 37.3 (3.93) | 41.2 (4.18) | 35.2 (4.27) | 44.2 (3.67) | 39.0 (3.92)
  Wek 15:Ease of Getting Sleep: number analyzed (Participants) | 37 | 40 | 37 | 34 | 31 | 32 | 37 | 37
  Wek 15:Ease of Getting Sleep | 39.8 (3.62) | 39.2 (3.29) | 42.8 (3.51) | 41.5 (3.59) | 49.4 (3.91) | 38.8 (3.85) | 44.8 (3.45) | 44.0 (3.64)
  Week 15: Quality of Sleep: number analyzed (Participants) | 37 | 40 | 37 | 34 | 31 | 32 | 37 | 37
  Week 15: Quality of Sleep | 39.3 (4.54) | 34.7 (4.19) | 37.1 (4.39) | 36.2 (4.52) | 45.9 (4.95) | 33.0 (4.88) | 42.4 (4.39) | 41.4 (4.60)
  Week 15: Ease of Awaking From Sleep: number analyzed (Participants) | 37 | 40 | 37 | 34 | 31 | 32 | 37 | 37
  Week 15: Ease of Awaking From Sleep | 33.9 (4.20) | 34.9 (3.88) | 37.1 (4.08) | 36.1 (4.21) | 45.4 (4.57) | 35.6 (4.51) | 49.4 (4.08) | 45.0 (4.26)
  Week 15: Integrity of Behavior Following Awaking: number analyzed (Participants) | 37 | 40 | 37 | 34 | 31 | 32 | 37 | 37
  Week 15: Integrity of Behavior Following Awaking | 40.9 (4.15) | 35.1 (3.81) | 46.7 (4.01) | 42.8 (4.11) | 50.9 (4.48) | 35.9 (4.43) | 47.1 (3.98) | 43.8 (4.19)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Ease of Getting to Sleep; Test type: Superiority; p = 0.5872, MMRM — LSM, SE, CI, & p-values come from an MMRM model with domain score as dependent variable & TG, visit & smoking status as factors & baseline measurement (BM) as a covariate, as well as interaction of treatment by week & an interaction of BM by week; LSMean difference = 2.3, 95% CI 2-sided [-6.09 to 10.73], Standard Error of Mean 4.27
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Ease of Getting to Sleep; Test type: Superiority; p = 0.3779, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 3.8, 95% CI 2-sided [-4.70 to 12.35], Standard Error of Mean 4.33
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Ease of Getting to Sleep; Test type: Superiority; p = 0.3506, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -4.1, 95% CI 2-sided [-12.61 to 4.49], Standard Error of Mean 4.34
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Ease of Getting to Sleep; Test type: Superiority; p = 0.8236, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 1.0, 95% CI 2-sided [-7.66 to 9.62], Standard Error of Mean 4.39
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Ease of Getting to Sleep; Test type: Superiority; p = 0.5949, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 2.3, 95% CI 2-sided [-6.24 to 10.87], Standard Error of Mean 4.35
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Ease of Getting to Sleep; Test type: Superiority; p = 0.9237, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-8.65 to 7.85], Standard Error of Mean 4.19
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Ease of Getting to Sleep; Test type: Superiority; p = 0.3599, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 4.0, 95% CI 2-sided [-4.54 to 12.46], Standard Error of Mean 4.32
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Quality of Sleep; Test type: Superiority; p = 0.7422, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 1.7, 95% CI 2-sided [-8.33 to 11.68], Standard Error of Mean 5.08
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Quality of Sleep; Test type: Superiority; p = 0.6030, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-12.67 to 7.37], Standard Error of Mean 5.09
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Quality of Sleep; Test type: Superiority; p = 0.2478, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -6.0, 95% CI 2-sided [-16.07 to 4.17], Standard Error of Mean 5.14
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Quality of Sleep; Test type: Superiority; p = 0.5295, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 3.3, 95% CI 2-sided [-6.94 to 13.47], Standard Error of Mean 5.18
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Quality of Sleep; Test type: Superiority; p = 0.6938, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-12.20 to 8.13], Standard Error of Mean 5.16
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Quality of Sleep; Test type: Superiority; p = 0.9765, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-9.93 to 9.63], Standard Error of Mean 4.97
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Quality of Sleep; Test type: Superiority; p = 0.4771, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 3.7, 95% CI 2-sided [-6.45 to 13.76], Standard Error of Mean 5.13
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Ease of Awaking From Sleep; Test type: Superiority; p = 0.4256, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 3.5, 95% CI 2-sided [-5.19 to 12.27], Standard Error of Mean 4.44
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Ease of Awaking From Sleep; Test type: Superiority; p = 0.9559, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-8.52 to 9.01], Standard Error of Mean 4.45
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Ease of Awaking From Sleep; Test type: Superiority; p = 0.2003, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -5.8, 95% CI 2-sided [-14.60 to 3.07], Standard Error of Mean 4.49
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Ease of Awaking From Sleep; Test type: Superiority; p = 0.6692, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -1.9, 95% CI 2-sided [-10.86 to 6.98], Standard Error of Mean 4.53
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Ease of Awaking From Sleep; Test type: Superiority; p = 0.6894, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-10.68 to 7.08], Standard Error of Mean 4.51
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Ease of Awaking From Sleep; Test type: Superiority; p = 0.1627, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -6.1, 95% CI 2-sided [-14.66 to 2.48], Standard Error of Mean 4.35
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Ease of Awaking From Sleep; Test type: Superiority; p = 0.9371, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-9.18 to 8.47], Standard Error of Mean 4.48
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Integrity of Behavior following Awaking; Test type: Superiority; p = 0.8521, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.8, 95% CI 2-sided [-8.07 to 9.77], Standard Error of Mean 4.53
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Integrity of Behavior following Awaking; Test type: Superiority; p = 0.9367, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.4, 95% CI 2-sided [-8.62 to 9.35], Standard Error of Mean 4.56
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Integrity of Behavior following Awaking; Test type: Superiority; p = 0.0551, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -8.8, 95% CI 2-sided [-17.82 to 0.19], Standard Error of Mean 4.57
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Integrity of Behavior following Awaking; Test type: Superiority; p = 0.4936, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean differencce = -3.2, 95% CI 2-sided [-12.32 to 5.96], Standard Error of Mean 4.64
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Integrity of Behavior following Awaking; Test type: Superiority; p = 0.6404, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 2.1, 95% CI 2-sided [-6.89 to 11.17], Standard Error of Mean 4.59
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Integrity of Behavior following Awaking; Test type: Superiority; p = 0.8955, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.6, 95% CI 2-sided [-8.17 to 9.34], Standard Error of Mean 4.45
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Integrity of Behavior following Awaking; Test type: Superiority; p = 0.9776, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.1, 95% CI 2-sided [-8.91 to 9.17], Standard Error of Mean 4.59
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Ease of Getting to Sleep; Test type: Superiority; p = 0.7852, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-9.27 to 7.01], Standard Error of Mean 4.14
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Ease of Getting to Sleep; Test type: Superiority; p = 0.7812, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 1.2, 95% CI 2-sided [-7.02 to 9.33], Standard Error of Mean 4.15
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Ease of Getting to Sleep; Test type: Superiority; p = 0.2648, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -4.7, 95% CI 2-sided [-13.07 to 3.61], Standard Error of Mean 4.23
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Ease of Getting to Sleep; Test type: Superiority; p = 0.6312, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-10.41 to 6.32], Standard Error of Mean 4.25
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Ease of Getting to Sleep; Test type: Superiority; p = 0.7416, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 1.4, 95% CI 2-sided [-6.89 to 9.67], Standard Error of Mean 4.20
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Ease of Getting to Sleep; Test type: Superiority; p = 0.4254, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 3.3, 95% CI 2-sided [-4.83 to 11.41], Standard Error of Mean 4.12
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Ease of Getting to Sleep; Test type: Superiority; p = 0.4038, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 3.4, 95% CI 2-sided [-4.66 to 11.54], Standard Error of Mean 4.11
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Quality of Sleep; Test type: Superiority; p = 0.3270, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -4.8, 95% CI 2-sided [-14.49 to 4.85], Standard Error of Mean 4.91
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Quality of Sleep; Test type: Superiority; p = 0.7333, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -1.7, 95% CI 2-sided [-11.21 to 7.90], Standard Error of Mean 4.85
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Quality of Sleep; Test type: Superiority; p = 0.1319, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -7.5, 95% CI 2-sided [-17.36 to 2.28], Standard Error of Mean 4.99
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Quality of Sleep; Test type: Superiority; p = 0.6132, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -2.5, 95% CI 2-sided [-12.38 to 7.32], Standard Error of Mean 5.00
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Quality of Sleep; Test type: Superiority; p = 0.4024, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -4.2, 95% CI 2-sided [-13.98 to 5.63], Standard Error of Mean 4.98
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Quality of Sleep; Test type: Superiority; p = 0.4904, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -3.4, 95% CI 2-sided [-12.97 to 6.23], Standard Error of Mean 4.88
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Quality of Sleep; Test type: Superiority; p = 0.5521, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -2.9, 95% CI 2-sided [-12.48 to 6.69], Standard Error of Mean 4.87
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Ease of Awaking From Sleep; Test type: Superiority; p = 0.7370, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-10.38 to 7.35], Standard Error of Mean 4.50
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Ease of Awaking From Sleep; Test type: Superiority; p = 0.5269, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -2.8, 95% CI 2-sided [-11.62 to 5.96], Standard Error of Mean 4.46
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Ease of Awaking From Sleep; Test type: Superiority; p = 0.3937, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -3.9, 95% CI 2-sided [-12.93 to 5.11], Standard Error of Mean 4.58
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Ease of Awaking From Sleep; Test type: Superiority; p = 0.8460, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.9, 95% CI 2-sided [-8.15 to 9.94], Standard Error of Mean 4.59
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Ease of Awaking From Sleep; Test type: Superiority; p = 0.5673, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-11.62 to 6.38], Standard Error of Mean 4.57
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Ease of Awaking From Sleep; Test type: Superiority; p = 0.3791, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 4.0, 95% CI 2-sided [-4.88 to 12.79], Standard Error of Mean 4.49
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Ease of Awaking From Sleep; Test type: Superiority; p = 0.8340, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.9, 95% CI 2-sided [-7.86 to 9.73], Standard Error of Mean 4.47
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.9457, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-9.51 to 8.88], Standard Error of Mean 4.67
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.6570, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -2.1, 95% CI 2-sided [-11.22 to 7.09], Standard Error of Mean 4.65
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.2310, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -5.7, 95% CI 2-sided [-15.00 to 3.64], Standard Error of Mean 4.73
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.9066, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.6, 95% CI 2-sided [-8.84 to 9.96], Standard Error of Mean 4.77
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.2914, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean differnce = -5.0, 95% CI 2-sided [-14.26 to 4.30], Standard Error of Mean 4.71
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.9277, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.4, 95% CI 2-sided [-8.73 to 9.57], Standard Error of Mean 4.64
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.9367, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-9.51 to 8.77], Standard Error of Mean 4.64
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Ease of Getting to Sleep; Test type: Superiority; p = 0.2407, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 5.1, 95% CI 2-sided [-3.46 to 13.69], Standard Error of Mean 4.35
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Ease of Getting to Sleep; Test type: Superiority; p = 0.1305, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 6.9, 95% CI 2-sided [-2.06 to 15.89], Standard Error of Mean 4.55
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Ease of Getting to Sleep; Test type: Superiority; p = 0.2152, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 5.7, 95% CI 2-sided [-3.34 to 14.75], Standard Error of Mean 4.59
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Ease of Getting to Sleep; Test type: Superiority; p = 0.1099, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 7.6, 95% CI 2-sided [-1.73 to 16.89], Standard Error of Mean 4.72
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Ease of Getting to Sleep; Test type: Superiority; p = 0.1219, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 7.4, 95% CI 2-sided [-1.99 to 16.75], Standard Error of Mean 4.75
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Ease of Getting to Sleep; Test type: Superiority; p = 0.0316, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 9.6, 95% CI 2-sided [0.85 to 18.36], Standard Error of Mean 4.44
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Ease of Getting to Sleep; Test type: Superiority; p = 0.1557, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 6.4, 95% CI 2-sided [-2.44 to 15.16], Standard Error of Mean 4.47
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Quality of Sleep; Test type: Superiority; p = 0.8592, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.9, 95% CI 2-sided [-8.91 to 10.67], Standard Error of Mean 4.97
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Quality of Sleep; Test type: Superiority; p = 0.6891, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 2.1, 95% CI 2-sided [-8.08 to 12.20], Standard Error of Mean 5.15
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Quality of Sleep; Test type: Superiority; p = 0.9481, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-10.59 to 9.92], Standard Error of Mean 5.20
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Quality of Sleep; Test type: Superiority; p = 0.7246, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -1.9, 95% CI 2-sided [-12.46 to 8.68], Standard Error of Mean 5.36
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Quality of Sleep; Test type: Superiority; p = 0.8842, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.8, 95% CI 2-sided [-9.94 to 11.53], Standard Error of Mean 5.45
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Quality of Sleep; Test type: Superiority; p = 0.8103, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 1.2, 95% CI 2-sided [-8.74 to 11.17], Standard Error of Mean 5.05
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Quality of Sleep; Test type: Superiority; p = 0.9631, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-9.81 to 10.28], Standard Error of Mean 5.10
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Ease of Awaking From Sleep; Test type: Superiority; p = 0.9788, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-9.73 to 9.47], Standard Error of Mean 4.87
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Ease of Awaking From Sleep; Test type: Superiority; p = 0.7875, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-11.26 to 8.54], Standard Error of Mean 5.02
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Ease of Awaking From Sleep; Test type: Superiority; p = 0.9746, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-9.85 to 10.17], Standard Error of Mean 5.08
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Ease of Awaking From Sleep; Test type: Superiority; p = 0.9092, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.6, 95% CI 2-sided [-9.67 to 10.86], Standard Error of Mean 5.21
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Ease of Awaking From Sleep; Test type: Superiority; p = 0.9745, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-10.55 to 10.21], Standard Error of Mean 5.27
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Ease of Awaking From Sleep; Test type: Superiority; p = 0.3458, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 4.7, 95% CI 2-sided [-5.08 to 14.44], Standard Error of Mean 4.95
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Ease of Awaking From Sleep; Test type: Superiority; p = 0.4657, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean differnce = 3.6, 95% CI 2-sided [-6.17 to 13.45], Standard Error of Mean 4.98
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.5838, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 2.8, 95% CI 2-sided [-7.20 to 12.76], Standard Error of Mean 5.07
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.8322, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 1.1, 95% CI 2-sided [-9.18 to 11.39], Standard Error of Mean 5.22
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.7366, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 1.8, 95% CI 2-sided [-8.59 to 12.13], Standard Error of Mean 5.26
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.2971, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 5.6, 95% CI 2-sided [-4.99 to 16.28], Standard Error of Mean 5.40
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.9562, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-10.96 to 10.37], Standard Error of Mean 5.41
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.0926, MMRM — [p-value comment as in outcome 30, analysis 1]; 0.28 = 8.7, 95% CI 2-sided [-1.44 to 18.76], Standard Error of Mean 5.13
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.4996, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 3.5, 95% CI 2-sided [-6.70 to 13.70], Standard Error of Mean 5.18
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Ease of Getting to Sleep; Test type: Superiority; p = 0.8960, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-9.99 to 8.75], Standard Error of Mean 4.76
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Ease of Getting to Sleep; Test type: Superiority; p = 0.5471, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 2.9, 95% CI 2-sided [-6.68 to 12.58], Standard Error of Mean 4.89
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Ease of Getting to Sleep; Test type: Superiority; p = 0.7380, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 1.7, 95% CI 2-sided [-8.06 to 11.36], Standard Error of Mean 4.93
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Ease of Getting to Sleep; Test type: Superiority; p = 0.0644, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 9.6, 95% CI 2-sided [-0.58 to 19.69], Standard Error of Mean 5.14
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Ease of Getting to Sleep; Test type: Superiority; p = 0.8475, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-10.90 to 8.96], Standard Error of Mean 5.04
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Ease of Getting to Sleep; Test type: Superiority; p = 0.3044, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 5.0, 95% CI 2-sided [-4.57 to 14.59], Standard Error of Mean 4.86
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Ease of Getting to Sleep; Test type: Superiority; p = 0.3895, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 4.2, 95% CI 2-sided [-5.42 to 13.86], Standard Error of Mean 4.89
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Quality of Sleep; Test type: Superiority; p = 0.4551, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -4.5, 95% CI 2-sided [-16.50 to 7.42], Standard Error of Mean 6.07
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Quality of Sleep; Test type: Superiority; p = 0.7182, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean differencce = -2.2, 95% CI 2-sided [-14.21 to 9.81], Standard Error of Mean 6.10
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Quality of Sleep; Test type: Superiority; p = 0.6259, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -3.0, 95% CI 2-sided [-15.26 to 9.20], Standard Error of Mean 6.21
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Quality of Sleep; Test type: Superiority; p = 0.3120, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 6.6, 95% CI 2-sided [-6.22 to 19.40], Standard Error of Mean 6.50
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Quality of Sleep; Test type: Superiority; p = 0.3297, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -6.3, 95% CI 2-sided [-18.89 to 6.37], Standard Error of Mean 6.41
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Quality of Sleep; Test type: Superiority; p = 0.6130, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 3.1, 95% CI 2-sided [-9.02 to 15.26], Standard Error of Mean 6.16
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Quality of Sleep; Test type: Superiority; p = 0.7292, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 2.2, 95% CI 2-sided [-10.09 to 14.40], Standard Error of Mean 6.22
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Ease of Awaking From Sleep; Test type: Superiority; p = 0.8695, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 0.9, 95% CI 2-sided [-1.11 to 11.96], Standard Error of Mean 5.60
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Ease of Awaking From Sleep; Test type: Superiority; p = 0.5800, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 3.1, 95% CI 2-sided [-7.99 to 14.25], Standard Error of Mean 5.64
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Ease of Awaking From Sleep; Test type: Superiority; p = 0.7024, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 2.2, 95% CI 2-sided [-9.11 to 13.50], Standard Error of Mean 5.74
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Ease of Awaking From Sleep; Test type: Superiority; p = 0.0572, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 11.4, 95% CI 2-sided [-0.35 to 23.23], Standard Error of Mean 5.99
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Ease of Awaking From Sleep; Test type: Superiority; p = 0.7830, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 1.6, 95% CI 2-sided [-10.04 to 13.31], Standard Error of Mean 5.93
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Ease of Awaking From Sleep; Test type: Superiority; p = 0.0074, MMRM — [p-value comment as in outcome 30, analysis 1]; 0.1 = 15.4, 95% CI 2-sided [4.19 to 26.67], Standard Error of Mean 5.71
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Ease of Awaking From Sleep; Test type: Superiority; p = 0.0551, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 11.0, 95% CI 2-sided [-0.24 to 22.32], Standard Error of Mean 5.73
Statistical Analysis 106: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.2959, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -5.8, 95% CI 2-sided [-16.63 to 5.08], Standard Error of Mean 5.51
Statistical Analysis 107: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.2976, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 5.8, 95% CI 2-sided [-5.14 to 16.74], Standard Error of Mean 5.55
Statistical Analysis 108: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.7236, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 2.0, 95% CI 2-sided [-9.07 to 13.05], Standard Error of Mean 5.62
Statistical Analysis 109: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.0884, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 10.1, 95% CI 2-sided [-1.52 to 21.63], Standard Error of Mean 5.88
Statistical Analysis 110: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.3887, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = -5.0, 95% CI 2-sided [-16.35 to 6.38], Standard Error of Mean 5.77
Statistical Analysis 111: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.2671, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 6.2, 95% CI 2-sided [-4.80 to 17.24], Standard Error of Mean 5.59
Statistical Analysis 112: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Integrity of Behavior Following Awaking; Test type: Superiority; p = 0.6076, MMRM — [p-value comment as in outcome 30, analysis 1]; LSMean difference = 2.9, 95% CI 2-sided [-8.20 to 13.99], Standard Error of Mean 5.63

31. Secondary Outcome: Change From Baseline in Greene Climacteric Scale (GCS) at Weeks 4, 8, 12, and 15
Description: The GCS is a 21-item scale that provides a brief but comprehensive and valid measure of climacteric symptomatology. Each item is rated by the participant according to its severity using a 4-point rating scale from 0 (none) to 3 (severe). The first 20 items of the scale combine into 3 main independent symptom measures by summing up the individual item scores: psychological symptoms (items 1 to 11; score 0 to 33), physical symptoms (items 12 to 18; score 0 to 21), and VMS (items 19 to 20; score 0 to 6). Item 21 is a probe for sexual dysfunction. The total score can range from 0 to 63. Higher scores indicate worse symptoms.
Time Frame: Baseline and weeks 4, 8, 12, and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 42 | 41 | 41 | 39 | 40 | 43 | 40
Score on a scale
  Week 4: Psychological Symptoms: number analyzed (Participants) | 41 | 42 | 41 | 40 | 39 | 40 | 42 | 40
  Week 4: Psychological Symptoms | -2.6 (0.70) | -3.8 (0.66) | -4.5 (0.69) | -5.0 (0.68) | -4.4 (0.71) | -3.7 (0.70) | -2.1 (0.65) | -4.9 (0.71)
  Week 4: Physical Symptoms: number analyzed (Participants) | 42 | 42 | 41 | 41 | 39 | 40 | 42 | 40
  Week 4: Physical Symptoms | -1.1 (0.38) | -1.1 (0.37) | -1.6 (0.38) | -1.1 (0.37) | -1.2 (0.39) | -1.4 (0.39) | -0.8 (0.36) | -1.9 (0.39)
  Week 4: VasomotorSymptoms Score | -1.7 (0.27) | -2.1 (0.25) | -2.7 (0.26) | -3.3 (0.26) | -3.2 (0.27) | -2.2 (0.27) | -2.6 (0.25) | -2.9 (0.27)
  Week 4: Sexual Dysfunction Score: number analyzed (Participants) | 42 | 42 | 41 | 41 | 39 | 39 | 43 | 40
  Week 4: Sexual Dysfunction Score | -0.4 (0.13) | -0.7 (0.12) | -0.7 (0.13) | -0.9 (0.13) | -0.7 (0.13) | -0.3 (0.13) | -0.4 (0.12) | -0.6 (0.13)
  Week 4: Total Score: number analyzed (Participants) | 41 | 42 | 41 | 40 | 39 | 39 | 41 | 40
  Week 4: Total Score | -6.1 (1.17) | -7.8 (1.10) | -9.6 (1.16) | -10.4 (1.15) | -9.5 (1.19) | -7.6 (1.19) | -5.8 (1.10) | -10.3 (1.19)
  Week 8: Psychological Symptoms: number analyzed (Participants) | 41 | 40 | 41 | 35 | 36 | 38 | 39 | 40
  Week 8: Psychological Symptoms | -3.3 (0.71) | -5.0 (0.69) | -4.7 (0.71) | -4.9 (0.73) | -4.5 (0.74) | -3.3 (0.73) | -2.8 (0.69) | -4.6 (0.73)
  Week 8: Physical Symptoms: number analyzed (Participants) | 41 | 40 | 41 | 36 | 36 | 38 | 39 | 40
  Week 8: Physical Symptoms | -1.1 (0.40) | -1.5 (0.39) | -1.3 (0.40) | -0.8 (0.40) | -1.6 (0.41) | -1.4 (0.41) | -0.9 (0.39) | -1.9 (0.40)
  Week 8: VasomotorSymptoms Score: number analyzed (Participants) | 41 | 40 | 41 | 36 | 36 | 38 | 39 | 40
  Week 8: VasomotorSymptoms Score | -1.9 (0.27) | -2.5 (0.26) | -3.0 (0.27) | -3.4 (0.28) | -3.5 (0.28) | -2.2 (0.28) | -2.9 (0.26) | -3.0 (0.28)
  Week 8: Sexual Dysfunction Score: number analyzed (Participants) | 41 | 40 | 41 | 36 | 36 | 37 | 39 | 40
  Week 8: Sexual Dysfunction Score | -0.4 (0.14) | -0.5 (0.13) | -0.8 (0.14) | -0.7 (0.14) | -0.6 (0.14) | -0.6 (0.14) | -0.3 (0.13) | -0.8 (0.14)
  Week 8: Total Score: number analyzed (Participants) | 41 | 40 | 41 | 35 | 36 | 37 | 39 | 40
  Week 8: Total Score | -6.9 (1.23) | -9.4 (1.18) | -9.9 (1.21) | -9.9 (1.25) | -10.1 (1.27) | -7.6 (1.26) | -7.0 (1.18) | -10.2 (1.24)
  Week 12: Psychological Symptoms: number analyzed (Participants) | 36 | 40 | 33 | 30 | 29 | 29 | 34 | 36
  Week 12: Psychological Symptoms | -3.3 (0.73) | -5.0 (0.68) | -4.9 (0.73) | -4.8 (0.75) | -4.3 (0.77) | -4.4 (0.77) | -3.6 (0.70) | -4.9 (0.74)
  Week 12: Physical Symptoms Score: number analyzed (Participants) | 36 | 40 | 33 | 30 | 29 | 29 | 35 | 36
  Week 12: Physical Symptoms Score | -1.5 (0.38) | -2.1 (0.36) | -1.0 (0.39) | -1.3 (0.40) | -1.6 (0.41) | -1.7 (0.41) | -0.9 (0.37) | -1.9 (0.39)
  Week 12: Vasomotor Symptoms Score: number analyzed (Participants) | 36 | 40 | 33 | 30 | 29 | 29 | 35 | 36
  Week 12: Vasomotor Symptoms Score | -2.1 (0.26) | -2.7 (0.24) | -3.1 (0.26) | -3.6 (0.26) | -3.6 (0.27) | -2.9 (0.27) | -2.8 (0.25) | -2.9 (0.26)
  Week 12: Sexual Dysfunction Score: number analyzed (Participants) | 36 | 40 | 33 | 30 | 29 | 29 | 35 | 36
  Week 12: Sexual Dysfunction Score | -0.5 (0.14) | -0.7 (0.13) | -1.1 (0.14) | -0.9 (0.15) | -0.8 (0.15) | -0.5 (0.15) | -0.5 (0.14) | -0.6 (0.14)
  Week 12: Total Score: number analyzed (Participants) | 36 | 40 | 33 | 30 | 29 | 29 | 34 | 36
  Week 12: Total Score | -7.6 (1.23) | -10.4 (1.15) | -10.1 (1.23) | -10.7 (1.25) | -10.3 (1.29) | -9.6 (1.29) | -7.8 (1.18) | -10.3 (1.24)
  Week 15: Psychological Symptoms Score ;: number analyzed (Participants) | 36 | 40 | 38 | 34 | 34 | 34 | 36 | 37
  Week 15: Psychological Symptoms Score ; | -2.7 (0.82) | -4.6 (0.76) | -4.3 (0.79) | -2.7 (0.82) | -2.3 (0.83) | -4.4 (0.84) | -2.6 (0.79) | -4.1 (0.82)
  Week 15: Physical Symptoms Score: number analyzed (Participants) | 36 | 40 | 38 | 35 | 34 | 34 | 37 | 37
  Week 15: Physical Symptoms Score | -1.4 (0.43) | -1.7 (0.40) | -1.8 (0.42) | -1.0 (0.42) | -1.4 (0.43) | -1.4 (0.44) | -1.2 (0.41) | -2.1 (0.43)
  Week 15: Vasomotor Symptoms Score: number analyzed (Participants) | 36 | 40 | 38 | 35 | 34 | 34 | 37 | 37
  Week 15: Vasomotor Symptoms Score | -1.4 (0.34) | -2.1 (0.32) | -1.6 (0.33) | -1.7 (0.34) | -1.9 (0.35) | -1.9 (0.35) | -1.8 (0.33) | -1.5 (0.34)
  Week 15: Sexual Dysfunction Score: number analyzed (Participants) | 36 | 40 | 38 | 35 | 34 | 34 | 37 | 37
  Week 15: Sexual Dysfunction Score | -0.5 (0.15) | -0.7 (0.14) | -0.6 (0.15) | -0.7 (0.15) | -0.5 (0.15) | -0.7 (0.16) | -0.6 (0.15) | -0.7 (0.15)
  Week 15: Total Score: number analyzed (Participants) | 36 | 40 | 38 | 34 | 34 | 34 | 36 | 37
  Week 15: Total Score | -6.3 (1.41) | -9.1 (1.31) | -8.3 (1.37) | -6.3 (1.41) | -6.0 (1.43) | -8.6 (1.44) | -6.3 (1.36) | -8.3 (1.41)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Psychological Symptoms Score; Test type: Superiority; p = 0.2159, MMRM — LSM, SE, CI, & p-values come from an MMRM model with CFB as dependent variable &TG, visit & smoking status as factors & baseline measurement as a covariate, as well as interaction of treatment by week & an interaction of baseline measurement by week; LSMean difference = -1.1, 95% CI 2-sided [-2.93 to 0.67], Standard Error of Mean 0.91
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Psychological Symptoms Score; Test type: Superiority; p = 0.0405, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.9, 95% CI 2-sided [-3.70 to -0.08], Standard Error of Mean 0.92
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Psychological Symptoms Score; Test type: Superiority; p = 0.0115, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -2.4, 95% CI 2-sided [-4.18 to -0.53], Standard Error of Mean 0.93
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Psychological Symptoms Score; Test type: Superiority; p = 0.0553, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-3.62 to 0.04], Standard Error of Mean 0.93
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Psychological Symptoms Score; Test type: Superiority; p = 0.2753, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-2.82 to 0.80], Standard Error of Mean 0.92
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Psychological Symptoms Score; Test type: Superiority; p = 0.5140, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.6, 95% CI 2-sided [-1.20 to 2.40], Standard Error of Mean 0.91
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Psychological Symptoms Score; Test type: Superiority; p = 0.0178, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -2.2, 95% CI 2-sided [-4.03 to -0.38], Standard Error of Mean 0.93
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Physical Symptoms Score; Test type: Superiority; p = 0.9675, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-1.02 to 0.98], Standard Error of Mean 0.51
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Physical Symptoms Score; Test type: Superiority; p = 0.3122, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-1.52 to 0.49], Standard Error of Mean 0.51
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Physical Symptoms Score; Test type: Superiority; p = 0.9977, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-1.00 to 1.00], Standard Error of Mean 0.51
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Physical Symptoms Score; Test type: Superiority; p = 0.9312, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean Difference = -0.0, 95% CI 2-sided [-1.05 to 0.97], Standard Error of Mean 0.51
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Physical Symptoms Score; Test type: Superiority; p = 0.6005, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-1.27 to 0.74], Standard Error of Mean 0.51
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Physical Symptoms Score; Test type: Superiority; p = 0.5284, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.3, 95% CI 2-sided [-0.68 to 1.32], Standard Error of Mean 0.51
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Physical Symptoms Score; Test type: Superiority; p = 0.1111, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.82 to 0.19], Standard Error of Mean 0.51
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Vasomotor Symptoms Score; Test type: Superiority; p = 0.1764, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-1.16 to 0.21], Standard Error of Mean 0.35
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Vasomotor Symptoms; Test type: Superiority; p = 0.0037, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.73 to -0.34], Standard Error of Mean 0.35
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Vasomotor Symptoms Score; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-2.30 to -0.92], Standard Error of Mean 0.35
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Vasomotor Symptoms Score; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-2.21 to -0.81], Standard Error of Mean 0.36
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Vasomotor Symptoms Score; Test type: Superiority; p = 0.1444, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-1.21 to 0.18], Standard Error of Mean 0.35
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Vasomotor Symptoms Score; Test type: Superiority; p = 0.0088, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.60 to -0.23], Standard Error of Mean 0.35
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Vasomotor Symptoms Score; Test type: Superiority; p = 0.0005, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.2, 95% CI 2-sided [-1.93 to -0.54], Standard Error of Mean 0.35
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Sexual Dysfunction Score; Test type: Superiority; p = 0.0416, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.69 to -0.01], Standard Error of Mean 0.17
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Sexual Dysfunction Score; Test type: Superiority; p = 0.0353, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.71 to -0.03], Standard Error of Mean 0.17
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Sexual Dysfunction Score; Test type: Superiority; p = 0.0040, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.84 to -0.16], Standard Error of Mean 0.17
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Sexual Dysfunction Score; Test type: Superiority; p = 0.0495, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.69 to -0.00], Standard Error of Mean 0.17
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Sexual Dysfunction Score; Test type: Superiority; p = 0.8665, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-0.31 to 0.37], Standard Error of Mean 0.17
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Sexual Dysfunction Score; Test type: Superiority; p = 0.9303, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.35 to 0.32], Standard Error of Mean 0.17
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Sexual Dysfunction Score; Test type: Superiority; p = 0.1039, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.62 to 0.06], Standard Error of Mean 0.17
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Total Score; Test type: Superiority; p = 0.2547, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-4.78 to 1.27], Standard Error of Mean 1.54
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Total Score; Test type: Superiority; p = 0.0225, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -3.6, 95% CI 2-sided [-6.60 to -0.50], Standard Error of Mean 1.55
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Total Score; Test type: Superiority; p = 0.0058, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean differencce = -4.3, 95% CI 2-sided [-7.38 to -1.26], Standard Error of Mean 1.55
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Total Score; Test type: Superiority; p = 0.0301, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -3.4, 95% CI 2-sided [-6.48 to -0.33], Standard Error of Mean 1.56
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Total Score; Test type: Superiority; p = 0.3220, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-4.59 to 1.51], Standard Error of Mean 1.55
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Total Score; Test type: Superiority; p = 0.8782, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-2.80 to 3.27], Standard Error of Mean 1.54
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Total Score; Test type: Superiority; p = 0.0069, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -4.2, 95% CI 2-sided [-7.27 to -1.17], Standard Error of Mean 1.55
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Psychological Symptoms Score; Test type: Superiority; p = 0.0890, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-3.49 to 0.25], Standard Error of Mean 0.95
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Psychological Symptoms Score; Test type: Superiority; p = 0.1444, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-3.25 to 0.48], Standard Error of Mean 0.95
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Psychological Symptoms Score; Test type: Superiority; p = 0.1022, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-3.51 to 0.32], Standard Error of Mean 0.97
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Psychological Symptoms Score; Test type: Superiority; p = 0.2342, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.2, 95% CI 2-sided [-3.07 to 0.75], Standard Error of Mean 0.97
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Psychological Symptoms Score; Test type: Superiority; p = 0.9906, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-1.89 to 1.87], Standard Error of Mean 0.96
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Psychological Symptoms Score; Test type: Superiority; p = 0.5770, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.5, 95% CI 2-sided [-1.34 to 2.40], Standard Error of Mean 0.95
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Psychological Symptoms Score; Test type: Superiority; p = 0.1865, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.3, 95% CI 2-sided [-3.14 to 0.61], Standard Error of Mean 0.95
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Physical Symptoms Score; Test type: Superiority; p = 0.4575, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-1.45 to 0.65], Standard Error of Mean 0.53
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Physical Symptoms Score; Test type: Superiority; p = 0.6016, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-1.33 to 0.77], Standard Error of Mean 0.53
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Physical Symptoms Score; Test type: Superiority; p = 0.7026, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-0.86 to 1.28], Standard Error of Mean 0.54
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Physical Symptoms Score; Test type: Superiority; p = 0.2971, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.64 to 0.50], Standard Error of Mean 0.54
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Physical Symptoms Score; Test type: Superiority; p = 0.5491, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-1.38 to 0.74], Standard Error of Mean 0.54
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Physical Symptoms Score; Test type: Superiority; p = 0.7142, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-0.86 to 1.25], Standard Error of Mean 0.54
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Physical Symptoms Score; Test type: Superiority; p = 0.1157, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.89 to 0.21], Standard Error of Mean 0.53
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Vasomotor Symptoms Score; Test type: Superiority; p = 0.1114, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.30 to 0.14], Standard Error of Mean 0.36
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Vasomotor Symptoms Score; Test type: Superiority; p = 0.0025, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.83 to -0.40], Standard Error of Mean 0.36
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Vasomotor Symptoms Scre; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-2.20 to -0.74], Standard Error of Mean 0.37
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Vasomotor Symptoms Score; Test type: Superiority; p = 0.5093, MMRM; LSMean difference = -0.2, 95% CI 2-sided [-0.96 to 0.48], Standard Error of Mean 0.37
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Vasomotor Symptoms Score; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-2.33 to -0.86], Standard Error of Mean 0.37
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Vasomotor Symptoms Score; Test type: Superiority; p = 0.0090, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.67 to -0.24], Standard Error of Mean 0.36
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Vasomotor Symptoms Score; Test type: Superiority; p = 0.0024, LSMean difference — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.84 to -0.40], Standard Error of Mean 0.37
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Sexual Dysfunction Score; Test type: Superiority; p = 0.5497, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.47 to 0.25], Standard Error of Mean 0.18
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Sexual Dysfunction Score; Test type: Superiority; p = 0.0276, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.76 to -0.04], Standard Error of Mean 0.18
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Sexual Dysfunction Score; Test type: Superiority; p = 0.1274, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.65 to 0.08], Standard Error of Mean 0.19
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Sexual Dysfunction Score; Test type: Superiority; p = 0.1865, LSMean difference — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.61 to 0.12], Standard Error of Mean 0.19
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Sexual Dysfunction Score; Test type: Superiority; p = 0.1857, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.61 to 0.12], Standard Error of Mean 0.18
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Sexual Dysfunction Score; Test type: Superiority; p = 0.8631, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-0.33 to 0.39], Standard Error of Mean 0.18
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Sexual Dysfunction Score; Test type: Superiority; p = 0.0304, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.75 to -0.04], Standard Error of Mean 0.18
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Total Score; Test type: Superiority; p = 0.1246, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -2.5, 95% CI 2-sided [-5.71 to 0.70], Standard Error of Mean 1.63
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Total Score; Test type: Superiority; p = 0.0680, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -3.0, 95% CI 2-sided [-6.19 to 0.22], Standard Error of Mean 1.63
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Total Score; Test type: Superiority; p = 0.0729, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -3.0, 95% CI 2-sided [-6.28 to 0.28], Standard Error of Mean 1.67
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Total Score; Test type: Superiority; p = 0.0541, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -3.2, 95% CI 2-sided [-6.49 to 0.06], Standard Error of Mean 1.66
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Total Score; Test type: Superiority; p = 0.6960, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-3.87 to 2.59], Standard Error of Mean 1.64
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Total Score; Test type: Superiority; p = 0.9725, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-3.27 to 3.15], Standard Error of Mean 1.63
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Total Score; Test type: Superiority; p = 0.0419, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -3.3, 95% CI 2-sided [-6.53 to -0.12], Standard Error of Mean 1.63
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Psychological Symptoms Score; Test type: Superiority; p = 0.0794, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.7, 95% CI 2-sided [-3.57 to 0.20], Standard Error of Mean 0.96
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Psychological Symptoms Score; Test type: Superiority; p = 0.1153, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-3.47 to 0.38], Standard Error of Mean 0.98
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Psychological Symptoms Score; Test type: Superiority; p = 0.1334, MMRM — [p-value comment as in outcome 31, analysis 1]; -1.5 = -1.5, 95% CI 2-sided [-3.47 to 0.46], Standard Error of Mean 1.00
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Psychological Symptoms Score; Test type: Superiority; p = 0.3457, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-2.93 to 1.03], Standard Error of Mean 1.00
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Psychological Symptoms Score; Test type: Superiority; p = 0.2607, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-3.07 to 0.83], Standard Error of Mean 0.99
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Psychological Symptoms Score; Test type: Superiority; p = 0.7816, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-2.18 to 1.64], Standard Error of Mean 0.97
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Psychological Symptoms Score; Test type: Superiority; p = 0.0955, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-3.54 to 0.29], Standard Error of Mean 0.97
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Physical Symptoms Score; Test type: Superiority; p = 0.2582, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.57 to 0.42], Standard Error of Mean 0.50
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Physical Symptoms Score; Test type: Superiority; p = 0.3448, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.5, 95% CI 2-sided [-0.53 to 1.52], Standard Error of Mean 0.52
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Physical Symptoms Score; Test type: Superiority; p = 0.6587, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-0.81 to 1.28], Standard Error of Mean 0.53
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Physical Symptoms Score; Test type: Superiority; p = 0.8299, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-1.16 to 0.93], Standard Error of Mean 0.53
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Physical Symptoms Score; Test type: Superiority; p = 0.8129, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-1.17 to 0.92], Standard Error of Mean 0.53
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Physical Symptoms Score; Test type: Superiority; p = 0.2130, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean Difference = 0.6, 95% CI 2-sided [-0.37 to 1.66], Standard Error of Mean 0.52
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Physical Symptoms Score; Test type: Superiority; p = 0.4131, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-1.42 to 0.59], Standard Error of Mean 0.51
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Vasomotor Symptoms Score; Test type: Superiority; p = 0.1273, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-1.20 to 0.15], Standard Error of Mean 0.34
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Vasomotor Symptoms Score; Test type: Superiority; p = 0.0046, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.69 to -0.31], Standard Error of Mean 0.35
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Vasomotor Symptoms Score; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-2.19 to -0.80], Standard Error of Mean 0.35
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Vasomotor Symptoms Score; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-2.19 to -0.78], Standard Error of Mean 0.36
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Vasomotor Symptoms Score; Test type: Superiority; p = 0.0333, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.45 to -0.06], Standard Error of Mean 0.35
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Vasomotor Symptoms Score; Test type: Superiority; p = 0.0423, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.39 to -0.02], Standard Error of Mean 0.35
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Vasomotor Symptoms Score; Test type: Superiority; p = 0.0208, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.49 to -0.12], Standard Error of Mean 0.35
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Sexual Dysfunction Score; Test type: Superiority; p = 0.3435, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.55 to 0.19], Standard Error of Mean 0.19
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Sexual Dysfunction Score; Test type: Superiority; p = 0.0021, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-0.98 to -0.22], Standard Error of Mean 0.19
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Sexual Dysfunction Score; Test type: Superiority; p = 0.0408, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.79 to -0.02], Standard Error of Mean 0.20
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Sexual Dysfunction Score; Test type: Superiority; p = 0.0911, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean differencce = -0.3, 95% CI 2-sided [-0.73 to 0.05], Standard Error of Mean 0.20
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Sexual Dysfunction Score; Test type: Superiority; p = 0.7891, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.44 to 0.33], Standard Error of Mean 0.20
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Sexual Dysfunction Score; Test type: Superiority; p = 0.9973, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-0.38 to 0.38], Standard Error of Mean 0.19
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Sexual Dysfunction Score; Test type: Superiority; p = 0.6377, MMRM — [p-value comment as in outcome 31, analysis 1]; -0.1 = -0.1, 95% CI 2-sided [-0.47 to 0.29], Standard Error of Mean 0.19
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Total Score; Test type: Superiority; p = 0.0862, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -2.8, 95% CI 2-sided [-5.95 to 0.40], Standard Error of Mean 1.61
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Total Score; Test type: Superiority; p = 0.1305, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -2.5, 95% CI 2-sided [-5.74 to 0.74], Standard Error of Mean 1.65
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Total Score; Test type: Superiority; p = 0.0707, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -3.0, 95% CI 2-sided [-6.34 to 0.26], Standard Error of Mean 1.68
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Total Score; Test type: Superiority; p = 0.1232, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-5.92 to 0.71], Standard Error of Mean 1.68
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Total Score; Test type: Superiority; p = 0.2530, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.9, 95% CI 2-sided [-5.18 to 1.37], Standard Error of Mean 1.66
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Total Score; Test type: Superiority; p = 0.9133, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-3.40 to 3.04], Standard Error of Mean 1.64
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Total Score; Test type: Superiority; p = 0.1078, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -2.6, 95% CI 2-sided [-5.85 to 0.58], Standard Error of Mean 1.63
Statistical Analysis 106: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Psychological Symptoms Score; Test type: Superiority; p = 0.0719, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean differencce = -1.9, 95% CI 2-sided [-4.07 to 0.18], Standard Error of Mean 1.08
Statistical Analysis 107: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Psychological Symptoms Score; Test type: Superiority; p = 0.1298, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.7, 95% CI 2-sided [-3.80 to 0.49], Standard Error of Mean 1.09
Statistical Analysis 108: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Psychological Symptoms Score; Test type: Superiority; p = 0.9532, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-2.26 to 2.13], Standard Error of Mean 1.11
Statistical Analysis 109: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Psychological Symptoms Score; Test type: Superiority; p = 0.7510, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.4, 95% CI 2-sided [-1.84 to 2.55], Standard Error of Mean 1.12
Statistical Analysis 110: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Psychological Symptoms Score; Test type: Superiority; p = 0.1120, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.8, 95% CI 2-sided [-3.95 to 0.42], Standard Error of Mean 1.11
Statistical Analysis 111: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Psychological Symptoms Score; Test type: Superiority; p = 0.9781, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-2.13 to 2.19], Standard Error of Mean 1.10
Statistical Analysis 112: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Psychological Symptoms Score; Test type: Superiority; p = 0.2060, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -1.4, 95% CI 2-sided [-3.57 to 0.77], Standard Error of Mean 1.10
Statistical Analysis 113: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Physical Symptoms Score; Test type: Superiority; p = 0.5332, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-1.46 to 0.76], Standard Error of Mean 0.56
Statistical Analysis 114: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Physical Symptoms Score; Test type: Superiority; p = 0.4599, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-1.54 to 0.70], Standard Error of Mean 0.57
Statistical Analysis 115: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Physical Symptoms Score; Test type: Superiority; p = 0.4752, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.4, 95% CI 2-sided [-0.72 to 1.55], Standard Error of Mean 0.58
Statistical Analysis 116: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Physical Symptoms Score; Test type: Superiority; p = 0.9051, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-1.21 to 1.07], Standard Error of Mean 0.58
Statistical Analysis 117: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Physical Symptoms Score; Test type: Superiority; p = 0.9937, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-1.14 to 1.15], Standard Error of Mean 0.58
Statistical Analysis 118: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Physical Symptoms Score; Test type: Superiority; p = 0.6956, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-0.91 to 1.35], Standard Error of Mean 0.57
Statistical Analysis 119: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Physical Symptoms Score; Test type: Superiority; p = 0.2302, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.81 to 0.44], Standard Error of Mean 0.57
Statistical Analysis 120: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Vasomotor Symptoms Score; Test type: Superiority; p = 0.1544, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.55 to 0.25], Standard Error of Mean 0.46
Statistical Analysis 121: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Vasomotor Symptoms Score; Test type: Superiority; p = 0.6847, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-1.10 to 0.72], Standard Error of Mean 0.46
Statistical Analysis 122: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Vasomotor Symptoms Score; Test type: Superiority; p = 0.5520, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-1.20 to 0.64], Standard Error of Mean 0.47
Statistical Analysis 123: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Vasomotor Symptoms Score; Test type: Superiority; p = 0.3632, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-1.36 to 0.50], Standard Error of Mean 0.47
Statistical Analysis 124: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Vasomotor Symptoms Score; Test type: Superiority; p = 0.2828, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-1.43 to 0.42], Standard Error of Mean 0.47
Statistical Analysis 125: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Vasomotor Symptoms Score; Test type: Superiority; p = 0.4702, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-1.24 to 0.58], Standard Error of Mean 0.47
Statistical Analysis 126: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Vasomotor Symptoms Score; Test type: Superiority; p = 0.8262, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-1.02 to 0.81], Standard Error of Mean 0.47
Statistical Analysis 127: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Sexual Dysfunction Score; Test type: Superiority; p = 0.3152, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.60 to 0.19], Standard Error of Mean 0.20
Statistical Analysis 128: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Sexual Dysfunction Score; Test type: Superiority; p = 0.4399, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.56 to 0.24], Standard Error of Mean 0.20
Statistical Analysis 129: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Sexual Dysfunction Score; Test type: Superiority; p = 0.1898, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.67 to 0.13], Standard Error of Mean 0.21
Statistical Analysis 130: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Sexual Dysfunction Score; Test type: Superiority; p = 0.9791, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-0.40 to 0.41], Standard Error of Mean 0.21
Statistical Analysis 131: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Sexual Dysfunction Score; Test type: Superiority; p = 0.3178, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.61 to 0.20], Standard Error of Mean 0.21
Statistical Analysis 132: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Sexual Dysfunction Score; Test type: Superiority; p = 0.4174, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.57 to 0.24], Standard Error of Mean 0.20
Statistical Analysis 133: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Sexual Dysfunction Score; Test type: Superiority; p = 0.2490, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.63 to 0.16], Standard Error of Mean 0.20
Statistical Analysis 134: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Total Score; Test type: Superiority; p = 0.1233, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -2.9, 95% CI 2-sided [-6.57 to 0.79], Standard Error of Mean 1.87
Statistical Analysis 135: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Total Score; Test type: Superiority; p = 0.2858, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-5.76 to 1.70], Standard Error of Mean 1.90
Statistical Analysis 136: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Total Score; Test type: Superiority; p = 0.9716, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-3.87 to 3.73], Standard Error of Mean 1.93
Statistical Analysis 137: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Total Score; Test type: Superiority; p = 0.9072, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-3.58 to 4.03], Standard Error of Mean 1.93
Statistical Analysis 138: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Total Score; Test type: Superiority; p = 0.2334, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -2.3, 95% CI 2-sided [-6.07 to 1.49], Standard Error of Mean 1.92
Statistical Analysis 139: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Total Score; Test type: Superiority; p = 0.9859, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-3.79 to 3.72], Standard Error of Mean 1.91
Statistical Analysis 140: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Total Score; Test type: Superiority; p = 0.2870, MMRM — [p-value comment as in outcome 31, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-5.77 to 1.72], Standard Error of Mean 1.90

32. Secondary Outcome: Change From Baseline in Menopause-Specific Quality of Life (MENQoL) at Weeks 4, 8, 12, and 15
Description: The MENQoL is self-administered and consists of a total of 29 items in a Likert-scale format. Each item assesses the impact of 1 of 4 domains of menopausal symptoms, as experienced over the last month: vasomotor (items 1 to 3), psychosocial (items 4 to 10), physical (items 11 to 26), and sexual (items 27 to 29). Items pertaining to a specific symptom are rated as present or not present, and if present, how bothersome on a 0 (not bothersome) to 6 (extremely bothersome) scale. Means are computed for each subscale by dividing the sum of the domain's items by the number of items within that domain. Non-endorsement of an item is scored a "1" and endorsement a "2," plus the number of the particular rating, so that the possible score on any item ranges from 1 to 8. Higher scores indicate that menopause symptoms are more bothersome.
Time Frame: Baseline and weeks 4, 8, 12, and 15
Population: FAS population with available data at specified time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 42 | 42 | 41 | 41 | 39 | 40 | 43 | 40
Score on a scale
  Week 4: Vasomotor Mean Score | -1.8 (0.32) | -2.4 (0.30) | -3.0 (0.32) | -3.4 (0.31) | -3.6 (0.32) | -1.9 (0.32) | -2.4 (0.30) | -2.8 (0.32)
  Week 4:Psychological Mean Score | -1.0 (0.21) | -1.2 (0.20) | -1.3 (0.21) | -1.3 (0.20) | -1.2 (0.21) | -0.8 (0.21) | -0.6 (0.20) | -1.0 (0.21)
  Week 4: Physical Mean Score | -0.8 (0.18) | -1.2 (0.17) | -1.4 (0.18) | -1.1 (0.18) | -1.3 (0.19) | -1.1 (0.19) | -0.8 (0.17) | -1.3 (0.19)
  Week 4: Sexual Mean Score: number analyzed (Participants) | 42 | 42 | 41 | 41 | 39 | 39 | 43 | 40
  Week 4: Sexual Mean Score | -0.7 (0.27) | -1.5 (0.25) | -1.8 (0.27) | -1.4 (0.26) | -1.2 (0.27) | -0.8 (0.28) | -0.7 (0.25) | -1.2 (0.27)
  Week 4: Overall Mean Score: number analyzed (Participants) | 42 | 42 | 41 | 41 | 39 | 39 | 43 | 40
  Week 4: Overall Mean Score | -0.9 (0.18) | -1.3 (0.17) | -1.6 (0.18) | -1.4 (0.17) | -1.5 (0.18) | -1.1 (0.18) | -0.9 (0.17) | -1.3 (0.18)
  Week 8: Vasomotor Mean Score: number analyzed (Participants) | 41 | 40 | 41 | 36 | 36 | 38 | 39 | 40
  Week 8: Vasomotor Mean Score | -2.1 (0.31) | -2.6 (0.30) | -3.4 (0.31) | -3.8 (0.31) | -4.1 (0.32) | -2.5 (0.32) | -3.1 (0.30) | -3.4 (0.32)
  Week 8: Psychological Mean Score: number analyzed (Participants) | 41 | 40 | 41 | 36 | 36 | 38 | 39 | 40
  Week 8: Psychological Mean Score | -1.2 (0.20) | -1.2 (0.19) | -1.3 (0.20) | -1.4 (0.20) | -1.3 (0.21) | -1.0 (0.20) | -1.0 (0.19) | -1.1 (0.20)
  Week 8: Physical Mean Score: number analyzed (Participants) | 41 | 40 | 41 | 36 | 36 | 38 | 39 | 40
  Week 8: Physical Mean Score | -1.0 (0.19) | -1.2 (0.18) | -1.5 (0.19) | -1.4 (0.19) | -1.5 (0.19) | -1.3 (0.19) | -1.0 (0.18) | -1.3 (0.19)
  Week 8: Sexual Mean Score: number analyzed (Participants) | 41 | 40 | 41 | 36 | 36 | 37 | 39 | 40
  Week 8: Sexual Mean Score | -0.9 (0.26) | -1.0 (0.25) | -1.7 (0.26) | -1.2 (0.27) | -1.2 (0.27) | -1.3 (0.27) | -0.8 (0.25) | -1.2 (0.27)
  Week 8: Overall Mean Score: number analyzed (Participants) | 41 | 40 | 41 | 36 | 36 | 37 | 39 | 40
  Week 8: Overall Mean Score | -1.2 (0.18) | -1.3 (0.17) | -1.7 (0.18) | -1.6 (0.18) | -1.7 (0.18) | -1.4 (0.18) | -1.2 (0.17) | -1.5 (0.18)
  Week 12: Vasomotor Mean Score: number analyzed (Participants) | 36 | 40 | 33 | 30 | 29 | 29 | 35 | 36
  Week 12: Vasomotor Mean Score | -2.3 (0.31) | -3.2 (0.29) | -3.5 (0.31) | -3.8 (0.31) | -4.4 (0.32) | -2.9 (0.32) | -3.3 (0.30) | -3.6 (0.31)
  Week 12: Psychological Mean Score: number analyzed (Participants) | 36 | 40 | 33 | 30 | 29 | 29 | 35 | 36
  Week 12: Psychological Mean Score | -1.3 (0.20) | -1.3 (0.19) | -1.7 (0.20) | -1.5 (0.21) | -1.4 (0.22) | -1.0 (0.22) | -1.1 (0.20) | -1.2 (0.21)
  Week 12: Physical Mean Score: number analyzed (Participants) | 36 | 40 | 33 | 30 | 29 | 29 | 35 | 35
  Week 12: Physical Mean Score | -1.3 (0.19) | -1.4 (0.18) | -1.6 (0.19) | -1.4 (0.19) | -1.5 (0.20) | -1.4 (0.20) | -1.0 (0.18) | -1.4 (0.19)
  Week 12: Sexual Score: number analyzed (Participants) | 36 | 40 | 33 | 30 | 29 | 28 | 35 | 36
  Week 12: Sexual Score | -0.8 (0.29) | -0.9 (0.27) | -1.8 (0.29) | -1.4 (0.29) | -0.9 (0.30) | -1.4 (0.31) | -0.8 (0.28) | -1.3 (0.29)
  Week 12: Overall Mean Score: number analyzed (Participants) | 36 | 40 | 33 | 30 | 29 | 28 | 35 | 35
  Week 12: Overall Mean Score | -1.3 (0.18) | -1.5 (0.17) | -1.8 (0.18) | -1.7 (0.18) | -1.7 (0.19) | -1.5 (0.19) | -1.3 (0.17) | -1.6 (0.18)
  Week 15: Vasomotor Mean Score: number analyzed (Participants) | 37 | 40 | 38 | 35 | 34 | 34 | 37 | 37
  Week 15: Vasomotor Mean Score | -1.8 (0.36) | -2.1 (0.34) | -1.7 (0.36) | -1.4 (0.37) | -1.7 (0.37) | -2.1 (0.38) | -2.2 (0.35) | -1.3 (0.37)
  Week 15: Psychological Mean Score: number analyzed (Participants) | 37 | 40 | 38 | 35 | 34 | 34 | 37 | 37
  Week 15: Psychological Mean Score | -1.0 (0.23) | -1.0 (0.22) | -1.3 (0.23) | -1.1 (0.23) | -0.9 (0.24) | -1.2 (0.24) | -0.9 (0.22) | -1.0 (0.23)
  Week 15: Physical Mean Score: number analyzed (Participants) | 37 | 40 | 38 | 35 | 34 | 34 | 37 | 37
  Week 15: Physical Mean Score | -1.2 (0.20) | -1.3 (0.18) | -1.5 (0.19) | -0.9 (0.20) | -1.2 (0.20) | -1.4 (0.20) | -1.0 (0.19) | -1.2 (0.20)
  Week 15: Sexual Mean Score: number analyzed (Participants) | 37 | 40 | 38 | 35 | 34 | 33 | 37 | 37
  Week 15: Sexual Mean Score | -0.6 (0.30) | -0.9 (0.28) | -1.5 (0.30) | -1.4 (0.30) | -0.6 (0.31) | -1.3 (0.32) | -0.6 (0.29) | -1.2 (0.30)
  Week 15: Overall Mean Score: number analyzed (Participants) | 37 | 40 | 38 | 35 | 34 | 33 | 37 | 37
  Week 15: Overall Mean Score | -1.1 (0.19) | -1.3 (0.18) | -1.5 (0.19) | -1.1 (0.19) | -1.2 (0.20) | -1.4 (0.21) | -1.0 (0.19) | -1.2 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Vasomotor Mean Score; Test type: Superiority; p = 0.1632, MMRM — LSM, SE, CI, & p-values come from an MMRM model with CFB as dependent variable & TG, visit & smoking status as factors & baseline measurement as a covariate, as well as interaction of treatment by week & interaction of baseline measurement by week; LSMean difference = -0.6, 95% CI 2-sided [-1.41 to 0.24], Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Vasomotor Mean Score; Test type: Superiority; p = 0.0045, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.2, 95% CI 2-sided [-2.03 to -0.38], Standard Error of Mean 0.42
Statistical Analysis 3: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Vasomotor Mean Score; Test type: Superiority; p = 0.0002, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.6, 95% CI 2-sided [-2.43 to -0.77], Standard Error of Mean 0.42
Statistical Analysis 4: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Vasomotor Mean Score; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.9, 95% CI 2-sided [-2.70 to -1.02], Standard Error of Mean 0.42
Statistical Analysis 5: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Vasomotor Mean Score; Test type: Superiority; p = 0.8569, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.91 to 0.76], Standard Error of Mean 0.42
Statistical Analysis 6: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Vasomotor Mean Score; Test type: Superiority; p = 0.1110, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.49 to 0.15], Standard Error of Mean 0.42
Statistical Analysis 7: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Vasomotor Mean Score; Test type: Superiority; p = 0.0187, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.83 to -0.17], Standard Error of Mean 0.42
Statistical Analysis 8: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Psychological Mean Score; Test type: Superiority; p = 0.4972, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.73 to 0.36], Standard Error of Mean 0.28
Statistical Analysis 9: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Psychological Mean Score; Test type: Superiority; p = 0.2568, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.86 to 0.23], Standard Error of Mean 0.28
Statistical Analysis 10: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Psychological Mean Score; Test type: Superiority; p = 0.2609, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.86 to 0.23], Standard Error of Mean 0.28
Statistical Analysis 11: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Psychological Mean Score; Test type: Superiority; p = 0.4148, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.78 to 0.32], Standard Error of Mean 0.28
Statistical Analysis 12: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Psychological Mean Score; Test type: Superiority; p = 0.5575, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-0.38 to 0.71], Standard Error of Mean 0.28
Statistical Analysis 13: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Psychological Mean Score; Test type: Superiority; p = 0.1671, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.4, 95% CI 2-sided [-0.16 to 0.92], Standard Error of Mean 0.28
Statistical Analysis 14: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Psychological Mean Score; Test type: Superiority; p = 0.9462, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.57 to 0.53], Standard Error of Mean 0.28
Statistical Analysis 15: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Physical Mean Score; Test type: Superiority; p = 0.0699, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.91 to 0.04], Standard Error of Mean 0.24
Statistical Analysis 16: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Physical Mean Score; Test type: Superiority; p = 0.0056, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.15 to -0.20], Standard Error of Mean 0.24
Statistical Analysis 17: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Physical Mean Score; Test type: Superiority; p = 0.1117, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.86 to 0.09], Standard Error of Mean 0.24
Statistical Analysis 18: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Physical Mean Score; Test type: Superiority; p = 0.0265, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-1.02 to -0.06], Standard Error of Mean 0.24
Statistical Analysis 19: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Physical Mean Score; Test type: Superiority; p = 0.1119, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.86 to 0.09], Standard Error of Mean 0.24
Statistical Analysis 20: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Physical Mean Score; Test type: Superiority; p = 0.7607, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.54 to 0.40], Standard Error of Mean 0.24
Statistical Analysis 21: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Physical Mean Score; Test type: Superiority; p = 0.0437, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.97 to -0.01], Standard Error of Mean 0.24
Statistical Analysis 22: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Sexual Mean Score; Test type: Superiority; p = 0.0211, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.51 to -0.12], Standard Error of Mean 0.35
Statistical Analysis 23: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Sexual Mean Score; Test type: Superiority; p = 0.0017, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.1, 95% CI 2-sided [-1.82 to -0.42], Standard Error of Mean 0.35
Statistical Analysis 24: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Sexual Mean Score; Test type: Superiority; p = 0.0598, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.37 to 0.03], Standard Error of Mean 0.35
Statistical Analysis 25: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Sexual Mean Score; Test type: Superiority; p = 0.1573, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean differencce = -0.5, 95% CI 2-sided [-1.21 to 0.20], Standard Error of Mean 0.36
Statistical Analysis 26: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Sexual Mean Score; Test type: Superiority; p = 0.7257, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.83 to 0.58], Standard Error of Mean 0.36
Statistical Analysis 27: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Sexual Mean Score; Test type: Superiority; p = 0.9324, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.72 to 0.66], Standard Error of Mean 0.35
Statistical Analysis 28: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Sexual Mean Score; Test type: Superiority; p = 0.2172, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-1.14 to 0.26], Standard Error of Mean 0.35
Statistical Analysis 29: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 4: Overall Mean Score; Test type: Superiority; p = 0.0742, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.88 to 0.04], Standard Error of Mean 0.23
Statistical Analysis 30: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 4: Overall Score; Test type: Superiority; p = 0.0035, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.16 to -0.23], Standard Error of Mean 0.24
Statistical Analysis 31: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 4: Overall Mean Score; Test type: Superiority; p = 0.0266, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.99 to -0.06], Standard Error of Mean 0.24
Statistical Analysis 32: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 4: Overall Mean Score; Test type: Superiority; p = 0.0124, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.06 to -0.13], Standard Error of Mean 0.24
Statistical Analysis 33: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 4: Overall Mean Score; Test type: Superiority; p = 0.4367, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.65 to 0.28], Standard Error of Mean 0.24
Statistical Analysis 34: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 4: Overall Mean Score; Test type: Superiority; p = 0.9318, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.48 to 0.44], Standard Error of Mean 0.23
Statistical Analysis 35: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 4: Overall Mean Score; Test type: Superiority; p = 0.0714, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.89 to 0.04], Standard Error of Mean 0.24
Statistical Analysis 36: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Vasomotor Mean Score; Test type: Superiority; p = 0.2027, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-1.35 to 0.29], Standard Error of Mean 0.42
Statistical Analysis 37: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Vasomotor Mean Score; Test type: Superiority; p = 0.0013, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.3, 95% CI 2-sided [-2.16 to -0.53], Standard Error of Mean 0.41
Statistical Analysis 38: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Vasomotor Mean Score; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.7, 95% CI 2-sided [-2.53 to -0.87], Standard Error of Mean 0.42
Statistical Analysis 39: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Vasomotor Mean Score; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-2.83 to -1.16], Standard Error of Mean 0.42
Statistical Analysis 40: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Vasomotor Mean Score; Test type: Superiority; p = 0.3791, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-1.19 to 0.45], Standard Error of Mean 0.42
Statistical Analysis 41: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Vasomotor Mean Score; Test type: Superiority; p = 0.0211, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.78 to -0.15], Standard Error of Mean 0.42
Statistical Analysis 42: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Vasomotor Mean Score; Test type: Superiority; p = 0.0021, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.3, 95% CI 2-sided [-2.10 to -0.47], Standard Error of Mean 0.42
Statistical Analysis 43: Comparison: Placebo vs Fezolinetant 15 mg BID; Wek 8: Psychological Mean Score; Test type: Superiority; p = 0.8890, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.55 to 0.48], Standard Error of Mean 0.26
Statistical Analysis 44: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Psychological Mean Score; Test type: Superiority; p = 0.5568, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.67 to 0.36], Standard Error of Mean 0.26
Statistical Analysis 45: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Psychological Mean Score; Test type: Superiority; p = 0.3989, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.75 to 0.30], Standard Error of Mean 0.27
Statistical Analysis 46: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Psychological Mean Score; Test type: Superiority; p = 0.6094, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.66 to 0.39], Standard Error of Mean 0.27
Statistical Analysis 47: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Psychological Mean Score; Test type: Superiority; p = 0.5229, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-0.35 to 0.69], Standard Error of Mean 0.26
Statistical Analysis 48: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Psychological Mean Score; Test type: Superiority; p = 0.4409, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-0.31 to 0.72], Standard Error of Mean 0.26
Statistical Analysis 49: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Psychological Mean Score; Test type: Superiority; p = 0.8062, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.1, 95% CI 2-sided [-0.45 to 0.58], Standard Error of Mean 0.26
Statistical Analysis 50: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Physical Mean Score; Test type: Superiority; p = 0.3663, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.71 to 0.26], Standard Error of Mean 0.25
Statistical Analysis 51: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Physical Mean Score; Test type: Superiority; p = 0.0424, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.99 to -0.02], Standard Error of Mean 0.25
Statistical Analysis 52: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Physical Mean Score; Test type: Superiority; p = 0.1597, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.85 to 0.14], Standard Error of Mean 0.25
Statistical Analysis 53: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Physical Mean Score; Test type: Superiority; p = 0.0595, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.97 to 0.02], Standard Error of Mean 0.25
Statistical Analysis 54: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Physical Symptoms Score; Test type: Superiority; p = 0.2162, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean differnce = -0.3, 95% CI 2-sided [-0.80 to 0.18], Standard Error of Mean 0.25
Statistical Analysis 55: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Physical Mean Score; Test type: Superiority; p = 0.9833, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.49 to 0.48], Standard Error of Mean 0.25
Statistical Analysis 56: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Physical Mean Score; Test type: Superiority; p = 0.2034, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.81 to 0.17], Standard Error of Mean 0.25
Statistical Analysis 57: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Sexual Mean Score; Test type: Superiority; p = 0.9576, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.70 to 0.67], Standard Error of Mean 0.35
Statistical Analysis 58: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Sexual Mean Score; Test type: Superiority; p = 0.0410, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.7, 95% CI 2-sided [-1.40 to -0.03], Standard Error of Mean 0.35
Statistical Analysis 59: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Sexual Mean Score; Test type: Superiority; p = 0.3961, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-1.00 to 0.40], Standard Error of Mean 0.35
Statistical Analysis 60: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 8: Sexual Mean Score; Test type: Superiority; p = 0.5012, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.94 to 0.46], Standard Error of Mean 0.36
Statistical Analysis 61: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Sexual Mean Score; Test type: Superiority; p = 0.2592, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-1.10 to 0.30], Standard Error of Mean 0.35
Statistical Analysis 62: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Sexual Mean Score; Test type: Superiority; p = 0.6141, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-0.51 to 0.86], Standard Error of Mean 0.35
Statistical Analysis 63: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Sexual Mean Score; Test type: Superiority; p = 0.4390, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.95 to 0.41], Standard Error of Mean 0.35
Statistical Analysis 64: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 8: Overall Mean Score; Test type: Superiority; p = 0.4521, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.64 to 0.29], Standard Error of Mean 0.23
Statistical Analysis 65: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 8: Overall Mean Score; Test type: Superiority; p = 0.0257, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.99 to -0.06], Standard Error of Mean 0.23
Statistical Analysis 66: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 8: Overall Mean Score; Test type: Superiority; p = 0.0564, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.93 to 0.01], Standard Error of Mean 0.24
Statistical Analysis 67: Comparison: Placebo vs Fezolinetant 90 mg BID; Wek 8: Overall Mean Score; Test type: Superiority; p = 0.0293, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.99 to -0.05], Standard Error of Mean 0.24
Statistical Analysis 68: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 8: Overall Mean Score; Test type: Superiority; p = 0.3742, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.68 to 0.26], Standard Error of Mean 0.24
Statistical Analysis 69: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 8: Overall Mean Score; Test type: Superiority; p = 0.9106, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.49 to 0.44], Standard Error of Mean 0.23
Statistical Analysis 70: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 8: Overall Mean SCore; Test type: Superiority; p = 0.1844, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.78 to 0.15], Standard Error of Mean 0.23
Statistical Analysis 71: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Vasomotor Mean Score; Test type: Superiority; p = 0.0287, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.69 to -0.09], Standard Error of Mean 0.41
Statistical Analysis 72: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Vasomotor Mean Score; Test type: Superiority; p = 0.0028, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.2, 95% CI 2-sided [-2.05 to -0.43], Standard Error of Mean 0.41
Statistical Analysis 73: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Vasomotor Mean Score; Test type: Superiority; p = 0.0004, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.5, 95% CI 2-sided [-2.32 to -0.67], Standard Error of Mean 0.42
Statistical Analysis 74: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Vasomotor Mean Score; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -2.0, 95% CI 2-sided [-2.87 to -1.22], Standard Error of Mean 0.42
Statistical Analysis 75: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Vasomotor Mean Score; Test type: Superiority; p = 0.1826, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.38 to 0.26], Standard Error of Mean 0.42
Statistical Analysis 76: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Vasomotor Mean Score; Test type: Superiority; p = 0.0178, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -1.0, 95% CI 2-sided [-1.79 to -0.17], Standard Error of Mean 0.41
Statistical Analysis 77: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Vasomotor Mean Score; Test type: Superiority; p = 0.0025, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean differnce = -1.2, 95% CI 2-sided [-2.06 to -0.44], Standard Error of Mean 0.41
Statistical Analysis 78: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Psychological Mean Score; Test type: Superiority; p = 0.9163, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.55 to 0.50], Standard Error of Mean 0.27
Statistical Analysis 79: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Psychological Mean Score; Test type: Superiority; p = 0.1597, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.92 to 0.15], Standard Error of Mean 0.27
Statistical Analysis 80: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Psychological Mean Score; Test type: Superiority; p = 0.4871, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.74 to 0.35], Standard Error of Mean 0.28
Statistical Analysis 81: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Psychological Mean Score; Test type: Superiority; p = 0.5401, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.72 to 0.38], Standard Error of Mean 0.28
Statistical Analysis 82: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Psychological Mean Score; Test type: Superiority; p = 0.3788, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-0.30 to 0.79], Standard Error of Mean 0.28
Statistical Analysis 83: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Psychological Mean Score; Test type: Superiority; p = 0.4541, MMRM — [p-value comment as in outcome 32, analysis 1]; 0.28 = 0.2, 95% CI 2-sided [-0.33 to 0.74], Standard Error of Mean 0.27
Statistical Analysis 84: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Psychological Mean Score; Test type: Superiority; p = 0.9233, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-0.51 to 0.56], Standard Error of Mean 0.27
Statistical Analysis 85: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Physical Mean Score; Test type: Superiority; p = 0.6043, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.61 to 0.35], Standard Error of Mean 0.24
Statistical Analysis 86: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Physical Mean Score; Test type: Superiority; p = 0.1781, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.82 to 0.15], Standard Error of Mean 0.25
Statistical Analysis 87: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Physical Mean Score; Test type: Superiority; p = 0.5221, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.66 to 0.34], Standard Error of Mean 0.25
Statistical Analysis 88: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Physical Mean Score; Test type: Superiority; p = 0.4744, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.68 to 0.32], Standard Error of Mean 0.25
Statistical Analysis 89: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Physical Mean Score; Test type: Superiority; p = 0.5167, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.66 to 0.33], Standard Error of Mean 0.25
Statistical Analysis 90: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Physical Mean Score; Test type: Superiority; p = 0.3441, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-0.25 to 0.72], Standard Error of Mean 0.25
Statistical Analysis 91: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Physical Mean Score; Test type: Superiority; p = 0.5362, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.64 to 0.33], Standard Error of Mean 0.25
Statistical Analysis 92: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Sexual Mean Score; Test type: Superiority; p = 0.9349, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.78 to 0.71], Standard Error of Mean 0.38
Statistical Analysis 93: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Sexual Mean Score; Test type: Superiority; p = 0.0084, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean differencce = -1.0, 95% CI 2-sided [-1.78 to -0.26], Standard Error of Mean 0.39
Statistical Analysis 94: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Sexual Mean Score; Test type: Superiority; p = 0.1212, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.38 to 0.16], Standard Error of Mean 0.39
Statistical Analysis 95: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Sexual Mean Score; Test type: Superiority; p = 0.7709, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.89 to 0.66], Standard Error of Mean 0.39
Statistical Analysis 96: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Sexual Mean Score; Test type: Superiority; p = 0.1667, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-1.33 to 0.23], Standard Error of Mean 0.40
Statistical Analysis 97: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Sexual Mean Score; Test type: Superiority; p = 0.9213, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-0.72 to 0.79], Standard Error of Mean 0.38
Statistical Analysis 98: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Sexual Mean Score; Test type: Superiority; p = 0.2315, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-1.21 to 0.29], Standard Error of Mean 0.38
Statistical Analysis 99: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 12: Overall Mean Score; Test type: Superiority; p = 0.4731, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.63 to 0.29], Standard Error of Mean 0.23
Statistical Analysis 100: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 12: Overall Mean Score; Test type: Superiority; p = 0.0310, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-0.98 to -0.05], Standard Error of Mean 0.24
Statistical Analysis 101: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 12: Overall Mean Score; Test type: Superiority; p = 0.1320, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.84 to 0.11], Standard Error of Mean 0.24
Statistical Analysis 102: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 12: Overall Mean Score; Test type: Superiority; p = 0.1212, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.85 to 0.10], Standard Error of Mean 0.24
Statistical Analysis 103: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Overall Mean Score; Test type: Superiority; p = 0.5689, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.62 to 0.34], Standard Error of Mean 0.24
Statistical Analysis 104: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 12: Overall Mean Score; Test type: Superiority; p = 0.7340, MMRM — [p-value comment as in outcome 32, analysis 1]; 0.1 = 0.1, 95% CI 2-sided [-0.39 to 0.55], Standard Error of Mean 0.24
Statistical Analysis 105: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 12: Overall Mean Score; Test type: Superiority; p = 0.2704, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.73 to 0.20], Standard Error of Mean 0.24
Statistical Analysis 106: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Vasomotor Mean Score; Test type: Superiority; p = 0.5610, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-1.24 to 0.67], Standard Error of Mean 0.48
Statistical Analysis 107: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Vasomotor Mean Score; Test type: Superiority; p = 0.7966, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.1, 95% CI 2-sided [-0.83 to 1.09], Standard Error of Mean 0.49
Statistical Analysis 108: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Vasomotor Mean Score; Test type: Superiority; p = 0.3965, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.4, 95% CI 2-sided [-0.56 to 1.40], Standard Error of Mean 0.50
Statistical Analysis 109: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Vasomotor Mean Score; Test type: Superiority; p = 0.8189, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.1, 95% CI 2-sided [-0.87 to 1.10], Standard Error of Mean 0.50
Statistical Analysis 110: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 12: Vasomotor Mean Score; Test type: Superiority; p = 0.5693, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-1.27 to 0.70], Standard Error of Mean 0.50
Statistical Analysis 111: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Vasomotor Mean Score; Test type: Superiority; p = 0.5217, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-1.29 to 0.65], Standard Error of Mean 0.49
Statistical Analysis 112: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Vasomotor Mean Score; Test type: Superiority; p = 0.2988, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.5, 95% CI 2-sided [-0.46 to 1.48], Standard Error of Mean 0.49
Statistical Analysis 113: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Psychological Mean Score; Test type: Superiority; p = 0.7957, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.69 to 0.53], Standard Error of Mean 0.31
Statistical Analysis 114: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Psychological Mean Score; Test type: Superiority; p = 0.2540, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.4, 95% CI 2-sided [-0.97 to 0.26], Standard Error of Mean 0.31
Statistical Analysis 115: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Psychological Mean Score; Test type: Superiority; p = 0.6956, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.75 to 0.50], Standard Error of Mean 0.32
Statistical Analysis 116: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Psychological Mean Score; Test type: Superiority; p = 0.8694, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.1, 95% CI 2-sided [-0.57 to 0.68], Standard Error of Mean 0.32
Statistical Analysis 117: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Psychological Mean Score; Test type: Superiority; p = 0.5047, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.84 to 0.41], Standard Error of Mean 0.32
Statistical Analysis 118: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Psychological Mean Score; Test type: Superiority; p = 0.7515, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.1, 95% CI 2-sided [-0.52 to 0.71], Standard Error of Mean 0.31
Statistical Analysis 119: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Psychological Mean Score; Test type: Superiority; p = 0.7818, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.70 to 0.53], Standard Error of Mean 0.31
Statistical Analysis 120: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Physical Mean Score; Test type: Superiority; p = 0.5770, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.65 to 0.36], Standard Error of Mean 0.26
Statistical Analysis 121: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Physical Mean Score; Test type: Superiority; p = 0.1893, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.85 to 0.17], Standard Error of Mean 0.26
Statistical Analysis 122: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Physical Mean Score; Test type: Superiority; p = 0.2997, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.3, 95% CI 2-sided [-0.25 to 0.79], Standard Error of Mean 0.26
Statistical Analysis 123: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Physical Mean Score; Test type: Superiority; p = 0.7529, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.60 to 0.44], Standard Error of Mean 0.26
Statistical Analysis 124: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Physical Mean Score; Test type: Superiority; p = 0.4173, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.2, 95% CI 2-sided [-0.73 to 0.31], Standard Error of Mean 0.26
Statistical Analysis 125: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Physical Mean Score; Test type: Superiority; p = 0.4944, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.2, 95% CI 2-sided [-0.34 to 0.69], Standard Error of Mean 0.26
Statistical Analysis 126: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Physical Mean Score; Test type: Superiority; p = 0.9231, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean differencce = -0.0, 95% CI 2-sided [-0.54 to 0.49], Standard Error of Mean 0.26
Statistical Analysis 127: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Sexual Mean Score; Test type: Superiority; p = 0.5112, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean differencce = -0.3, 95% CI 2-sided [-1.04 to 0.52], Standard Error of Mean 0.40
Statistical Analysis 128: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Sexual Mean Score; Test type: Superiority; p = 0.0300, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.9, 95% CI 2-sided [-1.66 to -0.09], Standard Error of Mean 0.40
Statistical Analysis 129: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Sexual Mean Score; Test type: Superiority; p = 0.0634, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.8, 95% CI 2-sided [-1.57 to 0.04], Standard Error of Mean 0.41
Statistical Analysis 130: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Sexual Mean Score; Test type: Superiority; p = 0.9406, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-0.78 to 0.84], Standard Error of Mean 0.41
Statistical Analysis 131: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Sexual Mean Score; Test type: Superiority; p = 0.1168, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.6, 95% CI 2-sided [-1.46 to 0.16], Standard Error of Mean 0.41
Statistical Analysis 132: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Sexual Mean Score; Test type: Superiority; p = 0.9937, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.0, 95% CI 2-sided [-0.79 to 0.80], Standard Error of Mean 0.40
Statistical Analysis 133: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Sexual Mean Score; Test type: Superiority; p = 0.1858, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.5, 95% CI 2-sided [-1.32 to 0.26], Standard Error of Mean 0.40
Statistical Analysis 134: Comparison: Placebo vs Fezolinetant 15 mg BID; Week 15: Overall Mean Score; Test type: Superiority; p = 0.5765, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.1, 95% CI 2-sided [-0.65 to 0.36], Standard Error of Mean 0.26
Statistical Analysis 135: Comparison: Placebo vs Fezolinetant 30 mg BID; Week 15: Overall Mean Score; Test type: Superiority; p = 0.1848, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.86 to 0.17], Standard Error of Mean 0.26
Statistical Analysis 136: Comparison: Placebo vs Fezolinetant 60 mg BID; Week 15: Overall Mean Score; Test type: Superiority; p = 0.7299, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.1, 95% CI 2-sided [-0.43 to 0.61], Standard Error of Mean 0.26
Statistical Analysis 137: Comparison: Placebo vs Fezolinetant 90 mg BID; Week 15: Overall Mean Score; Test type: Superiority; p = 0.9415, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.54 to 0.50], Standard Error of Mean 0.26
Statistical Analysis 138: Comparison: Placebo vs Fezolinetant 30 mg QD; Week 15: Overall Mean Score; Test type: Superiority; p = 0.2742, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.3, 95% CI 2-sided [-0.82 to 0.23], Standard Error of Mean 0.27
Statistical Analysis 139: Comparison: Placebo vs Fezolinetant 60 mg QD; Week 15: Overall Mean Score; Test type: Superiority; p = 0.6946, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = 0.1, 95% CI 2-sided [-0.41 to 0.62], Standard Error of Mean 0.26
Statistical Analysis 140: Comparison: Placebo vs Fezolinetant 120 mg QD; Week 15: Overall Mean Score; Test type: Superiority; p = 0.9442, MMRM — [p-value comment as in outcome 32, analysis 1]; LSMean difference = -0.0, 95% CI 2-sided [-0.53 to 0.50], Standard Error of Mean 0.26

33. Secondary Outcome: Change Over Time From Baseline in Plasma Concentrations of Luteinizing Hormone (LH) at Week 12
Description: Change was calculated as the post-baseline measurement minus the baseline measurement. Baseline was the last measurement taken prior to initial study drug administration.
Time Frame: Baseline and week 12
Population: FAS population with available data at baseline and specified time point.
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 37 | 40 | 33 | 30 | 28 | 28 | 35 | 36
International unit per liter (IU/L) | -1.14 (8.00) | -1.28 (8.53) | -3.28 (8.93) | -7.30 (15.49) | -10.86 (12.64) | -3.69 (11.21) | -3.97 (9.55) | -8.62 (11.95)

34. Secondary Outcome: Change Over Time From Baseline in Plasma Concentrations of Follicle-Stimulating Hormone (FSH) at Week 12
Description: as for outcome 33
Time Frame: Baseline and week 12
Population: FAS population with available data at baseline and specified time point.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 37 | 40 | 33 | 30 | 28 | 28 | 35 | 36
IU/L | -0.91 (9.79) | -1.52 (12.88) | -1.00 (13.51) | -6.49 (25.58) | -9.43 (17.40) | -0.98 (26.90) | -0.07 (8.97) | -9.94 (16.96)

35. Secondary Outcome: Change Over Time From Baseline in Plasma Concentrations of Estradiol (E2) at Week 12
Description: Change was calculated as the post-baseline measurement minus the baseline measurement. Baseline was the last measurement taken prior to initial study drug administration. The analysis value for Estradiol was imputed as 73.4/2 = 36.7 when result was < 73.4.
Time Frame: Baseline and week 12
Population: FAS population with available data at baseline and specified time point.
Measure: Mean (Standard Deviation); unit: picomole per milliliter (pmol/L)
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 37 | 40 | 33 | 30 | 28 | 28 | 35 | 36
picomole per milliliter (pmol/L) | 1.49 (7.41) | -1.29 (53.58) | 20.47 (93.37) | 10.15 (96.52) | -4.85 (56.56) | -15.99 (213.04) | -32.08 (198.54) | 1.32 (5.68)

36. Secondary Outcome: Change Over Time From Baseline in Plasma Concentrations of Sex Hormone-Binding Globulin (SHBG) at Week 12
Description: as for outcome 33
Time Frame: Baseline and week 12
Population: FAS population with available data at baseline and specified time point.
Measure: Mean (Standard Deviation); unit: Nanomole per liter (nmol/L)
Arm/Group | Placebo | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
Number analyzed (Participants) | 37 | 40 | 33 | 30 | 28 | 28 | 35 | 36
Nanomole per liter (nmol/L) | 1.877 (12.270) | 0.720 (14.220) | 4.867 (10.492) | 1.621 (16.329) | 6.643 (11.107) | 2.350 (17.852) | 0.143 (8.741) | 0.583 (14.283)

ADVERSE EVENTS:
Time Frame: From date of informed consent until end of the study (up to 15 weeks)
Arm/Group | Placebo BID | Fezolinetant 15 mg BID | Fezolinetant 30 mg BID | Fezolinetant 60 mg BID | Fezolinetant 90 mg BID | Fezolinetant 30 mg QD | Fezolinetant 60 mg QD | Fezolinetant 120 mg QD
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/45 | 0/43 | 0/45 | 0/44 | 0/43 | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/45 | 0/43 | 0/45 | 0/44 | 0/43 | 1/45 | 0/44
Other Adverse Events (participants affected / at risk) | 5/43 | 9/45 | 7/43 | 11/45 | 11/44 | 12/43 | 14/45 | 11/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo BID (N=43) | Fezolinetant 15 mg BID (N=45) | Fezolinetant 30 mg BID (N=43) | Fezolinetant 60 mg BID (N=45) | Fezolinetant 90 mg BID (N=44) | Fezolinetant 30 mg QD (N=43) | Fezolinetant 60 mg QD (N=45) | Fezolinetant 120 mg QD (N=44)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo BID (N=43) | Fezolinetant 15 mg BID (N=45) | Fezolinetant 30 mg BID (N=43) | Fezolinetant 60 mg BID (N=45) | Fezolinetant 90 mg BID (N=44) | Fezolinetant 30 mg QD (N=43) | Fezolinetant 60 mg QD (N=45) | Fezolinetant 120 mg QD (N=44)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 3 (4)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 6 (6) | 3 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT03192176/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT03192176/SAP_001.pdf